# I1F-MC-RHCD Statistical Analysis Plan Version 3

Multicenter, Double-Blind, Randomized, Placebo-Controlled Study to Evaluate Safety, Tolerability, and Efficacy of Ixekizumab in Patients from 6 to Less than 18 Years of Age with Moderate-to-Severe Plaque Psoriasis.

NCT03073200

Approval Date: 26-Jun-2019

# 1. Statistical Analysis Plan:

I1F-MC-RHCD: A Multicenter, Double-Blind, Randomized, Placebo-Controlled Study to Evaluate Safety, Tolerability, and Efficacy of Ixekizumab in Patients from 6 to Less than 18 Years of Age with Moderate-to-Severe Plaque Psoriasis

#### **Confidential Information**

The information contained in this document is confidential and the information contained within it may not be reproduced or otherwise disseminated without the approval of Eli Lilly and Company or its subsidiaries.

Note to Regulatory Authorities: This document may contain protected personal data and/or commercially confidential information exempt from public disclosure. Eli Lilly and Company requests consultation regarding release/redaction prior to any public release. In the United States, this document is subject to Freedom of Information Act (FOIA) Exemption 4 and may not be reproduced or otherwise disseminated without the written approval of Eli Lilly and Company or its subsidiaries.

#### Ixekizumab (LY2439821) Pediatric Psoriasis

Study I1F-MC-RHCD is a Phase 3, multicenter, randomized, double-blind, placebo-controlled study, examining the effects of ixekizumab versus placebo on PASI 75 and sPGA in subjects from 6 to <18 years of age with moderate to severe plaque psoriasis (PASI  $\geq$ 12, sPGA  $\geq$ 3, BSA  $\geq$ 10%) at screening and baseline.

Eli Lilly and Company Indianapolis, Indiana USA 46285 Protocol I1F-MC-RHCD (Phase 3)

Statistical Analysis Plan Version 1 electronically signed and approved by Lilly: 06-June-2017

Statistical Analysis Plan Version 2 electronically signed and approved by Lilly: 18-March-2019

Statistical Analysis Plan Version 3 electronically signed and approved by Lilly on date provided below.

Approval Date: 26-Jun-2019 GMT

# 2. Table of Contents

| Section | Page |
|---|---|
| 1. Statistical Analysis Plan: I1F-MC-RHCD: A Blind, Randomized, Placebo-Controlled Study Tolerability, and Efficacy of Ixekizumab in Pa than 18 Years of Age with Moderate-to-Severe | to Evaluate Safety,<br>tients from 6 to Less |
| | • |
| 2. Table of Contents | |
| 3. Revision History | |
| 4. Study Objectives | |
| 5. Study Design | |
| , , , | |
| <u>e</u> | |
| 6. A Priori Statistical Methods | |
| • | 23 |
| 6.1.3.1. Double-Blind Treatment Period (P | |
| 6.1.3.2. Double-Blind Treatment Period (P Addendum(2) | eriod 2): Protocol25 |
| 6.1.3.3. Combined Treatment Periods | 25 |
| 6.1.3.4. Double-Blind Randomized Withdr | rawal Period (Period 4)25 |
| 6.2. Adjustments for Covariates | 26 |
| | 26 |
| | 26 |
| | OCF)26 |
| | 27 |
| | 27 |
| - | |
| - | 27 |
| 6.8. Patient Characteristics | 28 |

| 6.8.1. | Demographics and Baseline Characteristics | 28 |
|---|---|---|
| 6.8.2. | Historical Illnesses and Preexisting Conditions | 30 |
| 6.9. Tı | reatment Compliance | 31 |
| 6.10. Pr | revious and Concomitant Therapy | 32 |
| 6.10.1. | Previous Therapy | 32 |
| 6.10.2. | Concomitant Therapy | 32 |
| 6.11. Et | fficacy Analyses | 34 |
| 6.11.1. | Co-Primary Outcome and Primary Analysis Methodology | 45 |
| 6.11.2. | Gated Secondary Efficacy Analyses | 45 |
| 6.11.3. | Additional Analyses of the Co-Primary Outcome | 45 |
| 6.11.4. | Other Secondary Efficacy Analyses | 45 |
| 6.12. H | ealth-Outcome/Quality-of-Life Analyses | 47 |
| 6.13. Ph | narmacokinetic/Pharmacodynamic Methods | 53 |
| 6.14. Sa | ıfety Analyses | 53 |
| 6.14.1. | Extent of Exposure | 54 |
| 6.14.2. | Adverse Events | 55 |
| 6.14.3. | | |
| | Adverse Events | 57 |
| 6.14. | J $J$ $I$ | <b>5</b> 0 |
| C 1 4 4 | Special Interest | |
| 6.14.4. | | |
| | 4.1. Leukocytes (White Blood Cells [WBCs]) and Platelets | |
| | 4.2. Neutrophil Follow-Up | |
| 6.14.5. | $\varepsilon$ | |
| 6.14.6. | | |
| 6.14.7. | F ( ) | |
| 6.14.8. | | |
| 6.14.9. | | |
| | 0. Immunization | |
| | 1. Immunogenicity | |
| | 11.1. Definitions and Terms | |
| | 4.11.1.1. Sample Category Definitions | |
| | 4.11.1.2. Patient Category Definitions | 76 |
| 6.1 | 4.11.1.3. Definitions for Clinical Interpretation of Assay Results | 77 |
| 6.14 | 11.2. Immunogenicity Analyses | |
| | 4.11.2.1. Analyses of Characteristics of ADA Immune | 19 |
| 0.1 | Response | 81 |
| | * | |

| 6.14.11.2.2. Analyses of Treatment-Emergent ADA Effects on Efficacy | 81 |
|---|---|
| 6.14.11.2.3. Analyses of Treatment-Emergent ADA on Specific Adverse Events | 82 |
| 6.15. Subgroup Analyses | 82 |
| 6.15.1. Efficacy Subgroup Analyses | 82 |
| 6.15.2. Safety Subgroup Analyses | 83 |
| 6.16. Protocol Deviations | 84 |
| 6.17. Interim Analyses and Data Monitoring | 94 |
| 6.18. Planned Exploratory Analyses | 95 |
| 6.18.1. Psychometric Analyses of the Itch NRS | 95 |
| 6.18.1.1. Descriptive Statistics | 95 |
| 6.18.1.2. Test-Retest Reliability | 95 |
| 6.18.1.3. Construct Validity | 96 |
| 6.18.1.3.1. Convergent and Discriminant Validity | 96 |
| 6.18.1.3.2. Known-Groups Validity | 96 |
| 6.18.1.4. Responsiveness | 96 |
| 6.18.1.5. Clinical Significance (Minimal Within-Patient Change) | 97 |
| 6.18.1.5.1. Anchor-Based Method | |
| 6.18.1.5.2. Distribution-Based Methods | 98 |
| 6.18.1.5.2.1. Standard Error of Measurement | 98 |
| 6.18.1.5.2.2. Empirical Cumulative Distribution Functions | 98 |
| 6.18.1.5.2.3. Probability Density Functions | 98 |
| 6.19. Clinical Trial Registry Analyses | 99 |
| 7. Unblinding Plan | 100 |
| 8. References | 101 |
| 9. Appendices | 104 |

# **Table of Contents**

| Table | | Page |
|---|---|---|
| Table RHCD.4.1. | Study Objectives | 10 |
| Table RHCD.4.2. | Protocol Addendum I1F-MC-RHCD(2) Study Objectives | 11 |
| Table RHCD.6.1. | Analysis Populations | 21 |
| Table RHCD.6.2. | Treatment Groups and Comparisons for Each Study Period and Analysis Population | 23 |
| Table RHCD.6.3. | Description and Derivation of Primary and Secondary Efficacy Outcomes | 35 |
| Table RHCD.6.4. | Description of Primary and Secondary Efficacy Analyses | 40 |
| Table RHCD.6.5. | Description and Derivation of Health-Outcome and Quality-of-Life Measures | 48 |
| Table RHCD.6.6. | Description of Health-Outcomes and Quality-of-Life Analyses | 52 |
| Table RHCD.6.7. | Definitions and Analyses of Special Safety Topics including<br>Adverse Events of Special Interest | 59 |
| Table RHCD.6.8. | Blood Pressure Levels for Children by Age and Gender (Median Height) | 71 |
| Table RHCD.6.9. | Categorical Criteria for Abnormal Treatment-Emergent Pulse Rate in Children and Adolescents Requiring Evaluation and Potential Intervention by a Health Care Professional | 72 |
| Table RHCD.6.10. | Baseline Definition for Immunogenicity Analyses for Overall Ixekizumab Treatment Period | 77 |
| Table RHCD.6.11. | TE-ADA Status Dichotomous Variables for AE Analysis | 80 |
| Table RHCD.6.12. | Identification and Action of Important Protocol Deviations | 85 |

# **Table of Contents**

| Figure | | Page |
|---|---|---|
| Figure RHCD.5.1. | Illustration of study design for Clinical Protocol I1F-MC-RHCD | 14 |
| Figure RHCD.5.2. | Illustration of study design for Protocol Addendum I1F-MC-RHCD(2) | 16 |
| Figure RHCD.6.1. | Sample definitions. | 75 |
| Figure RHCD.6.2. | Patient categories (evaluable/unevaluable) based on sample status at baseline and postbaseline. | 76 |
| Figure RHCD.6.3. | Relationship of terms for clinical interpretation of assay results for evaluable patients. | 78 |
| Figure RHCD.6.4. | Flow chart of ADA assessment with clinical interpretation of the various result possibilities. | 79 |

# **Table of Contents**

| Appendix | | Page |
|---|---|---|
| Appendix 1. | Concomitant Topical Therapy Definition | 105 |
| Appendix 2. | Anti-infective Treatments and Anatomical Therapeutic Chemical (ATC) Code List | 108 |
| Appendix 3. | Lilly-Defined MedDRA V21.0 Preferred Terms for Opportunistic Infections (OIs) | 113 |
| Appendix 4. | MedDRA Preferred Terms for each Category Associated with<br>Criterion 2 for Anaphylactic Allergic Reactions/Hypersensitivity<br>Events | 123 |
| Appendix 5. | Allergic Reactions/Hypersensitivity MedDRA Preferred Term List | 125 |
| Appendix 6. | Lilly-Defined MedDRA V21.0 Preferred Terms for Inflammatory Bowel Disease (IBD) | 128 |

# 3. Revision History

Statistical analysis plan (SAP) Version 1 was approved prior to unblinding of treatment assignments for Study Period 2.

Statistical Analysis Plan (SAP) Version 2 was approved prior to primary database lock (12 week).

Statistical Analysis Plan (SAP) Version 3 was approved after primary database lock and prior to submission database lock.

#### Revisions since Version 1:

| Section | Action |
|---|---|
| Section 4.1 Study Objectives | Updated time point Week 2 to Week 4. |
| Table 4.1 | |
| Section 6.1.1 Analysis Population | Updated abbreviations for placebo and etanercept arms. |
| Table 6.2 | |
| Section 6.5. Multiple | Updated time point Week 2 to Week 4. |
| Comparisons/Multiplicity | |
| Section 6.8.1 Demographics and | Updated age category criteria. |
| Baseline Characteristics | Removed immunization history. |
| | Updated "Fingernail psoriasis" to "Nail psoriasis". |
| Section 6.8.2 Historical Illness and | Clarified definitions of historical illness and pre-existing conditions. |
| Preexisting Conditions | |
| Section 6.11 Efficacy Analyses | Updated NAPSI definitions with toenail scores added. |
| Table 6.3 | Corrected typo. |
| | Updated PSSI definition. |
| Section 6.11 Efficacy Analyses | Added logistic regression with NRI to categorical endpoints as secondary |
| Table 6.4 | analysis method. |
| Section 6.11.2 Gated Secondary | Updated time point Week 2 to Week 4. |
| Efficacy Analyses | |
| Section 6.12 Health- | Corrected definition of CDLQI question #7. |
| Outcome/Quality-of-Life Analyses | |
| Table 6.5 | |
| Section 6.12 Health- | Added logistic regression with NRI to categorical endpoints as secondary |
| Outcome/Quality-of-Life Analyses | analysis method. |
| Table 6.6 | |
| Section 6.14.1 Extent of Exposure | Removed by-patient listing for extent of exposure. |
| Section 6.14.2.1 Common Adverse | Removed. |
| Events | |
| Section 6.14.3.1 Special Safety | Text updates for definition/derivation of AESIs to be consistent with PSAP |
| Topics Including Adverse Events of | V8 |
| Special Interest | Removed duplicated or unnecessary analyses |
| Table 6.7 | Changed Covance to performing lab reference range |
| | Wording updates per most recent PSAP for Infections, Allergic |
| | Reactions/Hypersensitivities, Injection Site Reactions, IBD, ILD. |

| Section | Action |
|---|---|
| Section 6.14.4 Clinical Laboratory<br>Evaluation | Removed by-patient listings. |
| Section 6.14.9 Tanner Stage Scale | Removed analysis for Period 2. |
| Section 6.15.1 Efficacy Subgroup<br>Analyses | Updated age category criteria. Updated duration of disease category. |
| Section 6.16 Protocol Violations Table 6.12 | Updated important protocol violations per most recent Trial Issue Management Plan. |
| Section 6.17 Interim Analyses and Data Monitoring | Added additional interim analyses to fulfill the need for regulatory interactions or publication purposes. |
| Section 6.18 Planned Exploratory<br>Analyses | Updated psychometric analyses of the Itch NRS. |
| References | Updated references |
| Appendices 3-6 | Updated per PSAP V8. |

# Revisions since Version 2:

| Section | Action |
|---|---|
| Section 6.16 Protocol Violations | Updated important protocol violations per most recent Trial Issue |
| Table 6.12 | Management Plan (to incorporate post-hoc change after the primary |
| | database lock). |

# 4. Study Objectives

Table RHCD.4.1. Study Objectives

| Objectives | Endpoints |
|---|---|
| Co-Primary To assess whether ixekizumab Q4W is superior to placebo at Week 12 (Visit 7) in the treatment of pediatric subjects (children and adolescents) with moderate-to-severe plaque psoriasis as measured by PASI 75 and by sPGA (0,1) | <ul> <li>Proportion of subjects achieving PASI 75 at Week 12</li> <li>Proportion of subjects achieving sPGA (0,1) at Week 12</li> </ul> |
| Gated Secondary To assess whether ixekizumab Q4W is superior to placebo as measured by: PASI 90 sPGA (0) PASI 100 Itch NRS PASI 75 sPGA (0,1) | <ul> <li>Proportion of subjects achieving PASI 90 at Week 12</li> <li>Proportion of subjects achieving sPGA (0) at Week 12</li> <li>Proportion of subjects achieving PASI 100 at Week 12</li> <li>Improvement ≥4 for subjects who had a baseline Itch NRS score ≥4 at Week 12</li> <li>Proportion of subjects achieving PASI 75 at Week 4</li> <li>Proportion of subjects achieving sPGA (0,1) at Week 4</li> </ul> |
| Other Secondary To assess whether ixekizumab Q4W is superior to placebo | The following endpoints will be assessed at Week 12 and at each postbaseline visit during the Double-Blind Treatment Period: • Proportion of subjects achieving PASI 50, PASI 75, PASI 90, and PASI 100 • Proportion of subjects achieving sPGA (0,1) and sPGA (0) • Change from baseline in itching severity (Itch NRS) score • CDLQI/DLQI (0,1) • Change from baseline in NAPSI, PSSI, and/or PPASI score in case of nail, scalp, or hand/feet involvement |
| To summarize the efficacy of ixekizumab Q4W at Week 24 (Visit 10) and Week 48 (Visit 16) as measured by: PASI 75 sPGA (0,1) PASI 90 sPGA (0) PASI 100 | <ul> <li>The following endpoints will be assessed:</li> <li>Proportion of subjects achieving PASI 75 at Weeks 24 and 48</li> <li>Proportion of subjects achieving sPGA (0,1) at Weeks 24 and 48</li> <li>Proportion of subjects achieving PASI 90 at Weeks 24 and 48</li> <li>Proportion of subjects achieving sPGA (0) at Weeks 24 and 48</li> <li>Proportion of subjects achieving PASI 100 at Weeks 24 and 48</li> <li>Proportion of subjects achieving PASI 100 at Weeks 24 and 48</li> </ul> |
| To evaluate the potential development of anti-<br>ixekizumab antibodies and its impact on subject<br>efficacy of ixekizumab To measure ixekizumab exposure and<br>characterize the pharmacokinetics of ixekizumab | <ul> <li>PASI 75 and sPGA(0,1) at Week 12 correlated with treatment-emergent antidrug antibody titer (low, moderate, and high) and by NAb status</li> <li>Serum trough concentrations of ixekizumab</li> </ul> |
| in pediatric subjects To assess the relationship between exposure and efficacy and exposure and immunogenicity | Model parameters for the exposure-response<br>relationship between ixekizumab serum trough<br>concentrations and efficacy endpoints (for example,<br>sPGA, PASI) at Week 12 |

| Objectives | Endpoints |
|---|---|
| | Serum trough concentrations for ixekizumab antibody titer subgroups |
| To assess the safety of ixekizumab | To evaluate the safety of ixekizumab, including but not limited to: infections; injection-site reactions; B-, T-, and NK-cell levels; WBC count; RBC count; and laboratory values (hematology and chemistry [including ALT and AST]) during the course of the study |
| To demonstrate normal growth and pubertal progression in children treated with ixekizumab during the course of the study | <ul> <li>Weight, height, and BMI data will be merged to the Centers for Disease Control and Prevention standard growth data by age and gender to compare subjects' growth with normal values</li> <li>Shift table for Tanner stage from maximum baseline to maximum postbaseline by gender</li> </ul> |
| To evaluate the genital involvement of the subjects per the questionnaire Binary Questions on Psoriasis Location | Proportion of subjects achieving no psoriasis presence in each psoriasis location |
| To evaluate the patient's global assessment of disease severity | <ul> <li>Proportion of subjects achieving patient's global<br/>assessment of disease severity 0 or 1</li> </ul> |
| To evaluate the effect of ixekizumab on maintenance of efficacy and health outcomes during the open-label maintenance period and extension period. | <ul> <li>Proportion of subjects achieving PASI 90</li> <li>Proportion of subjects achieving sPGA (0)</li> <li>Proportion of subjects achieving PASI 100</li> <li>Proportion of subjects achieving PASI 75</li> <li>Proportion of subjects achieving sPGA (0,1)</li> <li>Improvement ≥4 for subjects who had a baseline Itch NRS score ≥4</li> </ul> |

Abbreviations: ALT = alanine aminotransferase; AST = aspartate aminotransferase; BMI = body mass index; CDLQI = Children's Dermatology Life Quality Index; DLQI = Dermatology Life Quality Index; NAb = neutralizing antidrug antibody; NAPSI = Nail Psoriasis Severity Index; NK = natural killer; NRS = numeric rating scale; PASI = Psoriasis Area and Severity Index; PASI 50 = at least a 50% improvement from baseline in PASI score; PASI 75 = at least a 75% improvement from baseline in PASI score; PASI 90 = at least a 90% improvement from baseline in PASI score; PASI = Palmoplantar Psoriasis Severity Index; PSSI = Psoriasis Severity Index; Q4W = every 4 weeks; RBC = red blood cell; sPGA = static Physician's Global Assessment; WBC = white blood cell.

Table RHCD.4.2. Protocol Addendum I1F-MC-RHCD(2) Study Objectives

| Objectives | Endpoints |
|---|---|
| Other Secondary To compare the efficacy of ixekizumab Q4W and etanercept at Week 12 (Visit 7) as measured by PASI 75 and by sPGA (0,1) in countries where etanercept is approved | <ul> <li>Proportion of subjects achieving PASI 75 at Week 12</li> <li>Proportion of subjects achieving sPGA (0,1) at Week 12</li> </ul> |
| To assess whether ixekizumab Q4W is superior to placebo for EU subjects during the Double-Blind, Randomized Withdrawal Period | <ul> <li>Time to relapse to moderate severity (sPGA ≥2) during the Double-Blind, Randomized Withdrawal Period</li> <li>Proportion of subjects achieving sPGA (0,1) at Week 108 (Visit 31)</li> </ul> |

Abbreviations: EU = European Union; PASI 75 = at least a 75% improvement from baseline in Psoriasis Area and Severity Index score; Q4W = every 4 weeks; sPGA = static Physician's Global Assessment.

# 5. Study Design

### 5.1. Summary of Study Design

Study I1F-MC-RHCD (RHCD) is a Phase 3, multicenter, double-blind, randomized, placebo-controlled study examining the effects of ixekizumab versus placebo in subjects from 6 to <18 years of age with moderate-to-severe plaque psoriasis (Ps) (Psoriasis Area and Severity Index [PASI] score ≥12, static Physician's Global Assessment [sPGA] ≥3, and body surface area [BSA] ≥10% at screening and baseline). Protocol Addendum I1F-MC-RHCD(1) specifies the pharmacokinetics (PK) collection schedule and how the data from the approximately 24 subjects participating in the PK addendum will be used. Protocol Addendum I1F-MC-RHCD(2) specifies the details for the active-controlled (etanercept) portion of the study design, as well as a double-blind, randomized withdrawal period for subjects from European Union (EU) countries.

The study consists of 5 periods:

- **Period 1: Screening Period** (Visit 1) will assess subject eligibility and will occur approximately 7 to 30 days before Period 2 (baseline; Week 0; Visit 2).
- **Period 2: Double-Blind Treatment Period** (Induction Period) will occur from Week 0 (baseline; Visit 2) to Week 12 (Visit 7), comparing ixekizumab with placebo in a double-blind fashion. The dose of ixekizumab will not be adjusted during this period. Protocol Addendum I1F-MC-RHCD(2) describes etanercept as a reference control group for countries where etanercept is approved for treatment of chronic severe Ps in children and adolescents from the age of 6 years who are inadequately controlled by, or are intolerant to, other systemic therapies or phototherapies.
- Period 3: 48-Week, Open-Label Maintenance Period will occur from Week 12 (Visit 7) to Week 60 (Visit 19). Subjects randomized to the ixekizumab group during Period 2 will maintain the dose received during the previous period. Subjects randomized to placebo during Period 2 will receive ixekizumab at doses of 20, 40, or 80 mg, based on weight. As part of Protocol Addendum I1F-MC-RHCD(2), subjects randomized to etanercept during the Double-Blind Treatment Period will begin treatment with ixekizumab after an 8-week washout period (to avoid, for safety reasons, increased risk with concurrent etanercept and ixekizumab exposures). If a subject changes weight category following the Double-Blind Treatment Period, the ixekizumab dose associated with that weight will be administered. This may happen at any time during the Maintenance Period.
- **Period 4: Extension Period** will occur from Week 60 (Visit 19) to Week 108 (Visit 31). Subjects will continue with open-label treatment of the ixekizumab dose received during the previous period (Period 3). Protocol Addendum I1F-MC-RHCD(2) describes the 48-week Double-Blind, Randomized Withdrawal Period for subjects from EU countries who meet response criteria during the Maintenance Period (defined as sPGA [0,1]). Subjects who enter the Double-Blind, Randomized Withdrawal Period will be re-randomized to ixekizumab or placebo (1:1 ratio) at Week 60 (Visit 19). Subjects who are re-randomized to

- ixekizumab will receive ixekizumab 20, 40, or 80 mg every 4 weeks (Q4W) according to their weight at the time of re-randomization.
- **Period 5: Post-Treatment Follow-Up Period** is for safety monitoring after treatment discontinuation for any subject receiving at least 1 dose of study drug. This period occurs from the last treatment period visit or Early Termination Visit (ETV) for up to 24 weeks following that visit.

The underlined text in the following sections show the additions and deletions applicable to subjects participating in Protocol Addendum I1F-MC-RHCD(2).

- **Period 2: Double-Blind Treatment Period** (Induction Period) will occur from Week 0 (baseline; Visit 2) to Week 12 (Visit 7), comparing ixekizumab to placebo in a double-blind fashion (all countries) and to etanercept (as a reference arm all countries except North America). The dose will remain the same in this treatment period.
- Period 3: 48-Week, Open-Label Maintenance Period will occur from Week 12 (Visit 7) to Week 60 (Visit 19). Subjects randomized to etanercept during Period 2 will receive ixekizumab at doses of 20, 40, or 80 mg, according to their weight after an etanercept 8-week washout period is complete. The etanercept washout period will be from Week 12 through Week 20. If a subject changes weight category following the Double-Blind Treatment Period, the ixekizumab dose associated with that weight will be administered. This may happen at any time during the Maintenance Period.
- **Period 4: Extension Period** will occur from Week 60 (Visit 19) to Week 108 (Visit 31). Subjects from countries outside of the EU, irrespective of response, and nonresponders from the EU will continue with open-label treatment with the ixekizumab dose received during the previous period (Period 3). Subjects from the EU who meet response criteria at Week 60 (defined as those with sPGA [0,1]) will be re-randomized to ixekizumab or placebo in the Double-Blind, Randomized Withdrawal Period. Subjects will receive the ixekizumab dose according to weight, which will be reassessed during this period.

Figure RHCD.5.1 and Figure RHCD.5.2 illustrate the study design for the main protocol and the protocol addendum (2).



Abbreviations: IXE = ixekizumab (LY2439821); LV = date of last visit; PK = pharmacokinetic(s); Q4W = every 4 weeks; SC = subcutaneous; V = visit; W = week. Footnotes on following page.

Figure RHCD.5.1. Illustration of study design for Clinical Protocol I1F-MC-RHCD.

#### Illustration of study design for Clinical Protocol I1F-MC-RHCD

- a Subjects will be randomized to either ixekizumab or placebo in a 2:1 ratio.
- b Subjects receiving ixekizumab 20 mg or 40 mg will receive 1 SC injection of ixekizumab at Week 0 (Visit 2) and 1 SC injection of ixekizumab Q4W at Weeks 4 and 8. Subjects receiving ixekizumab 80 mg will receive 2 SC injections of ixekizumab at Week 0 (Visit 2) and 1 SC injection of ixekizumab Q4W at Weeks 4 and 8. Subjects receiving placebo for ixekizumab 20 mg or 40 mg will receive 1 SC injection of placebo at Week 0 (Visit 2) and 1 SC injection of placebo Q4W at Weeks 4 and 8. Subjects receiving placebo for ixekizumab 80 mg will receive 2 SC injections of placebo at Week 0 (Visit 2) and 1 SC injection of placebo Q4W at Weeks 4 and 8.
- c Immunogenicity and time-matched PK sample collection will occur as detailed in the Schedule of Activities (Section 2) of the Protocol
- d Subjects randomized to ixekizumab during Period 2 will receive 1 SC injection of ixekizumab and 1 SC injection of placebo at Week 12. Subjects randomized to the placebo group during Period 2 will be assigned to receive ixekizumab at doses of 20, 40, or 80 mg, based on weight. Subjects assigned to 20 mg will receive a starting dose of 40 mg, subjects assigned to 40 mg will receive a starting dose of 80 mg, and subjects assigned to 80 mg will receive a starting dose of 160 mg. All subjects will receive 2 SC injections of ixekizumab at Week 12 and 1 SC injection of ixekizumab Q4W at Week 16 and thereafter. Treatment with ixekizumab is weight-based. If a subject changes weight category during the study, the dose will be adjusted accordingly.
- e All subjects receiving study drug must enter into Period 5, and complete through Visit 802. Subjects may be followed up beyond Visit 802 for continued monitoring of their neutrophil count if determined by the Sponsor/investigator that additional monitoring is needed.
- At Visit 2, randomization will occur based on the following weight groups: 1) <25 kg: randomization to ixekizumab 20 mg, receiving a starting dose of 40 mg; 2) 25 kg to 50 kg: randomization to ixekizumab 40 mg, receiving a starting dose of 80 mg; and 3) >50 kg: randomization to 80 mg, receiving a starting dose of 160 mg. A staggered approach to enrollment by weight group will be implemented with subjects >12 years and >50 kg enrolling initially to the study. If no safety concern is identified after an initial safety analysis of the first 12 weeks of treatment in the first 15 subjects >50 kg, subjects will start to enroll in the 25- to 50-kg group. Once data are obtained to Week 12 for approximately 15 subjects in the 25- to 50-kg group, an interim analysis of PK, safety, and efficacy data in all subjects in the study at that point will be performed to confirm doses for the remaining subjects in the study. Once confirmed, all weight groups will be open for enrollment.



Abbreviations: EU = European Union; LV = date of last visit; OEU = outside the European Union; PASI = Psoriasis Area and Severity Index PK = pharmacokinetic(s); Ps = plaque psoriasis; Q1W = every week; Q4W = every 4 weeks; RW = randomized withdrawal; SC = subcutaneous; sPGA = static Physician's Global Assessment; V = visit; W = weeks. Footnotes on following page.

Figure RHCD.5.2. Illustration of study design for Protocol Addendum I1F-MC-RHCD(2).

- a Randomization will be stratified by region (United States/Canada, EU countries, and rest of the world) and by etanercept approval status: 1) Subjects with severe pediatric Ps (PASI ≥20 or sPGA ≥4) who are from countries where etanercept is approved for the treatment of severe pediatric Ps will be randomized to ixekizumab, etanercept, or placebo in a 2:2:1 ratio. 2) Per the main protocol, all other subjects (including those with moderate-to-severe Ps [PASI ≥12 and sPGA ≥3] from countries where etanercept is not approved for the treatment of severe pediatric Ps, and subjects with moderate pediatric Ps [12 ≤PASI <20 and sPGA = 3] in countries where etanercept is approved for the treatment of severe pediatric Ps) will be randomized to either ixekizumab or placebo in a 2:1 ratio.
- b At Visit 2, randomization will occur according to the following weight groups: 1) <25 kg: randomization to ixekizumab 20 mg, receiving a starting dose of 40 mg; 2) 25 kg to 50 kg: randomization to ixekizumab 40 mg, receiving a starting dose of 80 mg; 3) >50 kg: randomization to 80 mg, receiving a starting dose of 160 mg. A staggered approach to enrollment by weight group will be implemented, with subjects aged >12 years and weighing >50 kg enrolling initially to the study. After an initial safety analysis of the first 12 weeks of treatment of 15 subjects weighing >50 kg, and if no safety concern is identified, subjects will start to enroll in the 25- to 50-kg group. Once data for Week 12 for approximately 15 subjects in the 25- to 50-kg group is gathered, an interim analysis of PK, safety, and efficacy data for all subjects in the study at that point will be performed to confirm doses for future subjects in the study. Once confirmed, all weight groups will be open for enrollment.
- c Subjects receiving ixekizumab 20 mg or 40 mg will receive 1 SC injection of ixekizumab at Week 0 (Visit 2) and 1 SC injection of ixekizumab Q4W at Weeks 4 and 8. Subjects receiving ixekizumab 80 mg will receive 2 SC injections of ixekizumab at Week 0 (Visit 2) and 1 SC injection of ixekizumab Q4W at Weeks 4 and 8.
- d Subjects receiving placebo for ixekizumab 20 mg or 40 mg will receive 1 SC injection of placebo at Week 0 (Visit 2) and 1 SC injection of placebo Q4W at Weeks 4 and 8. Subjects receiving placebo for ixekizumab 80 mg will receive 2 SC injections of placebo at Week 0 (Visit 2) and 1 SC injection of placebo Q4W at Weeks 4 and 8.
- e Subjects will be randomized to receive etanercept 0.8 mg/kg and up to a maximum of 50 mg per dose. All subjects will receive etanercept SC Q1W at Week 0 through Week 11.
- f Unblinded site personnel will prepare the doses of ixekizumab and placebo.
- g Subjects will initiate Maintenance Period as follows: (1) Subjects randomized to the ixekizumab arm during Period 2 will receive 1 SC injection of ixekizumab and 1 SC injection of placebo at Week 12. (2) Subjects randomized to the placebo arm during Period 2 will be assigned to receive ixekizumab at doses of 20, 40, or 80 mg, according to weight, and will receive 2 ixekizumab injections as follows—subjects assigned to 20 mg will receive a starting dose of 40 mg; subjects assigned to 40 mg will receive a starting dose of 80 mg; subjects assigned to 80 mg will receive a starting dose of 160 mg. All subjects will be assigned to receive ixekizumab at doses of 20, 40, or 80 mg, according to their weight. Subjects assigned to 20 mg will receive a starting dose of 40 mg. Subjects assigned to 40 mg will receive a starting dose of 80 mg. Subjects assigned to 80 mg will receive a starting dose of 160 mg. Treatment with ixekizumab is weight-based. If a subject changes weight category during the study and after the Double-Blind Treatment Period, the dose will be adjusted accordingly.
- h All subjects will receive 1 SC injection of ixekizumab Q4W.
- i Subjects from EU countries who meet the response criterion at Week 60 (defined as sPGA [0,1]) will be re-randomized to ixekizumab or placebo (1:1 ratio). Subjects from EU countries who do not meet response criteria and subjects from non-EU countries will continue with open-label treatment with ixekizumab.
- j Subjects will receive ixekizumab upon disease relapse to Ps (sPGA  $\geq$ 2).
- k All subjects receiving investigational product must enter into the Post-Treatment Follow-Up Period (Period 5) and complete through Visit 802. Subjects may be followed beyond Visit 802 for continued monitoring of their neutrophil counts if needed or if determined by the Sponsor/investigator that additional monitoring is needed.

### 5.2. Determination of Sample Size

#### 5.2.1. Clinical Protocol RHCD

Sample size of this study is based on the regulatory requirements from the European Medicine's Agency Paediatric Investigation Plan for ixekizumab. The regulatory requirements for the number of subjects in each treatment group were: (1) at least 170 randomized subjects (at least 90 to ixekizumab, at least 25 to etanercept, and at least 55 to placebo); and (2) at least 30% of subjects from the EU.

In the main protocol RHCD, approximately 165 subjects will be randomized in a 2:1 ratio to receive ixekizumab (110 subjects) or placebo (55 subjects) during the Double-Blind Treatment Period. The study will have >99% power to test the superiority of ixekizumab to placebo for PASI 75 and for sPGA (0,1) at Week 12, based on the 2-sided Fisher's exact test at a significance level of 0.05. The following assumptions were used for the power calculations for both sPGA (0,1) and PASI 75 responses rates, based on ixekizumab clinical studies in adult subjects with moderate-to severe Ps efficacy data (Griffiths et al. 2015; Gordon et al. 2016): 80% response for ixekizumab and 10% response for placebo for both PASI 75 and sPGA (0,1).

## 5.2.2. Protocol Addendum RHCD(2)

During the Double-Blind Treatment Period, approximately 75 subjects with severe Ps from etanercept-approved countries will be randomized to ixekizumab (30 subjects), etanercept (30 subjects), and placebo (15 subjects) with 2:2:1 ratio.

Study RHCD(2) will have approximately 85% power to test the superiority of ixekizumab to etanercept for sPGA (0,1) and at least a 75% improvement from baseline in PASI score (PASI 75) at Week 12, based on the 2-sided Fisher's exact test at significance level of 0.05. The study will have approximately 45% power to test the superiority of etanercept to placebo for PASI 75 at Week 12, based on the 2-sided Fisher's exact test at significance level of 0.05. The following assumptions were used for the power calculations for both sPGA (0,1) and PASI 75 response rates, based on ixekizumab clinical studies in adult subjects with moderate-to-severe Ps efficacy data (Griffiths et al. 2015; Gordon et al. 2016): 80% responders for ixekizumab, 40% responders for etanercept, and 10% for placebo.

During the Double-Blind, Randomized Withdrawal Period (Period 4), approximately 40 subjects from EU countries will be re-randomized to ixekizumab (20 subjects) and placebo (20 subjects) with a 1:1 ratio. The response criterion for re-randomization is sPGA (0,1) at Week 60. The study will have approximately 95% power to test the superiority of ixekizumab to placebo in time to relapse, based on the 2-sided log-rank test at significance level of 0.05. The following assumptions were used for the power calculations: 20% relapse for ixekizumab; and 85% relapse for placebo. Relapse rates were estimated, based on ixekizumab clinical studies in adult subjects with moderate-to-severe Ps efficacy data (Griffiths et al. 2015; Gordon et al. 2016).

### 5.3. Method of Assignment to Treatment

Assignment to treatment groups will be determined by a computer-generated random sequence using an interactive web-response system (IWRS). The IWRS will be used to assign cartons containing double-blind study drug to each subject. Study site personnel will confirm that they have located the correct carton by entering a confirmation number into the IWRS.

#### 5.3.1. Clinical Protocol RHCD

Subjects who meet all enrollment criteria at Visit 1 and Visit 2 will be randomized in a 2:1 ratio to double-blind treatment with ixekizumab or placebo at Week 0 (Visit 2).

To achieve between-group comparability for region, the randomization will be stratified by region (United States/Canada, European countries, and the rest of the world).

During the Maintenance and Extension periods, all subjects will receive open-label treatment with ixekizumab.

### 5.3.2. Protocol Addendum RHCD(2)

Subjects from countries where etanercept is approved for severe pediatric Ps treatment only who meet all criteria for enrollment at Visit 1 and Visit 2 will be randomized to double-blind treatment at Week 0 (Visit 2) in a 2:2:1 ratio to ixekizumab, etanercept, or placebo.

Subjects who meet response criteria (sPGA 0,1) from EU countries will enter the Double-Blind Randomized Withdrawal Period and will be re-randomized to double-blind treatment at Week 60 (Visit 19) in a 1:1 ratio to ixekizumab or placebo. Subjects who are re-randomized to ixekizumab will receive ixekizumab 20, 40, or 80 mg every 4 weeks (Q4W) according to their weight at the time of re-randomization. Subjects from EU countries who relapse (sPGA  $\geq$ 2) during the Double-Blind Randomized Withdrawal Period will receive open-label treatment with ixekizumab according to their weight at the time of relapse.

### 6. A Priori Statistical Methods

#### 6.1. General Considerations

Statistical analysis of this study will be the responsibility of Eli Lilly and Company (hereafter, Lilly, or its designee). The statistical analyses will be performed using SAS® Version 9.2 or higher.

Continuous data will be summarized in terms of the number of observations, mean, standard deviation (SD), minimum, median, and maximum. The minimum and maximum will be reported to the same number of decimal places as the raw data recorded in the database. The mean and median will be reported to 1 more decimal place than the raw data recorded in the database. The SD will be reported to 2 more decimal places than the raw data recorded in the database. In general, the maximum number of decimal places reported shall be 4 for any summary statistic.

Categorical data will be summarized in terms of the number of patients in the Analysis Population, the number of patients providing data at the relevant time point, frequency counts, and the percentages corresponding to the appropriate method. Percentages will be presented to 1 decimal place. Percentages will not be presented for zero counts.

All confidence intervals (CIs) and statistical tests will be 2-sided unless, otherwise, specified. P-values which are greater than or equal to  $(\ge)$  0.001, and less than or equal to  $(\le)$  0.999, will be presented to 3 decimal places. All other p-values which are less than 0.001 will be presented as <0.001, while p-values greater than 0.999 will be presented as >0.999. Confidence intervals will be presented to 1 more decimal place than the raw data.

Age, gender, and race will be reported on all by-patient listings unless, otherwise, specified. Gender will be abbreviated as follows: female (F); and male (M). Race will be abbreviated as follows: American Indian or Alaska Native (AI), Asian (AS), Black or African American (BL), Native Hawaiian or other Pacific Islander (NH), White (WH), and Multiple (MU).

# 6.1.1. Analysis Population

Table RHCD.6.1 provides the definitions for each analysis population for specific treatment periods. Table RHCD.6.2 summarizes the treatment groups and comparisons for each study period and analysis population.

Unless, otherwise, specified, efficacy and health-outcome analyses will be conducted for the Intent-to-treat (ITT) Population (per the main study) in Double-Blind Treatment Period (Period 2). In addition, the co-primary endpoints will be analyzed using the per-protocol set (PPS).

Select efficacy analyses will be conducted on the ITT Population-Etanercept Approved Countries (per Protocol Addendum[2]) in Double-Blind Treatment Period (Period 2).

Safety analyses for the Double-Blind Treatment Period (Period 2) will be conducted on the Safety Population. There are 2 safety populations: Safety Population (per the main study); and Safety Population-Etanercept Approved Countries (per Protocol Addendum[2]).

Unless, otherwise, specified, the efficacy and safety analyses for the Double-Blind, Randomized Withdrawal Period will be conducted on the Double-Blind, Randomized Withdrawal Period Population (per Protocol Addendum[2]).

Unless, otherwise, specified, during the Combined Treatment Periods (Periods 2, 3, and 4), efficacy and health-outcome analysis will be conducted on the ixekizumab Efficacy Primary Population.

Safety analyses during the Combined Treatment Periods (Periods 2, 3, and 4) will be conducted on the All Ixekizumab Safety Population

Unless, otherwise, specified, during Combined Treatment Periods 3 and 4, efficacy analysis will be conducted on the Ixekizumab Efficacy Secondary Population.

Safety analyses for the Post-Treatment Follow-Up Period (Period 5) will be conducted on the Follow-Up Population.

Table RHCD.6.1. Analysis Populations

| Population | Period | Description |
|---|---|---|
| Intent-to-Treat (ITT) | Double-Blind Treatment Period (Period 2) | All randomized subjects, even if the subject |
| Population (per main | | does not take the assigned treatment, does |
| study) | | not receive the correct treatment, or, |
| | | otherwise, does not follow the protocol. |
| | | Unless, otherwise, specified, efficacy and |
| | | health-outcome analyses will be conducted |
| | | on the ITT Population during Double-Blind |
| | | Treatment Period (Period 2). Subjects will |
| | | be analyzed according to the treatment to |
| | | which they were assigned. |
| Intent-to-Treat (ITT) | Double-Blind Treatment Period (Period 2) | All randomized subjects per Protocol |
| - Etanercept | | Addendum(2) in etanercept-approved |
| Approved Countries | | countries (that is, subjects with severe |
| (per Protocol | | psoriasis in countries where etanercept is |
| Addendum[2]) | | used as a reference arm), even if the subject |
| | | does not take the assigned treatment, does |
| | | not receive the correct treatment, or, |
| | | otherwise, does not follow the protocol. |
| | | Subjects will be analyzed according to the |
| D D : 10 : / | D 11 DI 17 | treatment to which they were assigned. |
| Per-Protocol Set (per | Double-Blind Treatment Period (Period 2) | All randomized subjects who do not have |
| main study) | | significant protocol violations (refer to |
| | | Section 6.16). Subjects will be analyzed |
| | | according to the treatment to which they |
| Cofety Domilation | Double Dind Treatment Donied (Donied 2) | were assigned. |
| Safety Population | Double-Blind Treatment Period (Period 2) | All randomized subjects who take at least |
| (per main study) | | 1 dose of double-blind study treatment. |
| | | Subjects will be analyzed according to the |
| | | treatment to which they were assigned. |

| Population | Period | Description |
|---|---|---|
| • | | • |
| Safety Population – | Double-Blind Treatment Period (Period 2) | All randomized subjects in Protocol |
| Etanercept-Approved | per Protocol Addendum(2) | Addendum(2) in etanercept countries who |
| Countries (per | | take at least 1 dose of double-blind study |
| Protocol | | treatment per Protocol Addendum(2). |
| Addendum[2]) | | Subjects will be analyzed according to the |
| | | treatment to which they were assigned. |
| Double-Blind, | Randomized-Withdrawal Period (Period 4) | All re-randomized patients (that is, subjects |
| Randomized | per Protocol Addendum(2) | from countries in the EU who were |
| Withdrawal Period | | re-randomized at Week 60) who received at |
| Population | | least 1 dose of study treatment during |
| | | Double-Blind, Randomized Withdrawal |
| | | Period. |
| Ixekizumab Efficacy | Combined Treatment Periods (Periods 2, 3, | All subjects randomized to ixekizumab at |
| Primary Population | and 4) | Week 0 (Visit 2) and who received |
| | | ixekizumab throughout their study |
| | | participations. The following subjects are |
| | | not included in this analysis population: |
| | | (1) patients randomized to etanercept or |
| | | placebo at Week 0; and (2) patients who are |
| | | re-randomized to placebo during Period 4 |
| | | per Protocol Addendum(2). |
| Ixekizumab Efficacy | Combined Treatment Periods 3 and 4 | Patients initially randomized to placebo or |
| Secondary | | etanercept who switch to ixekizumab during |
| Population | | Period 3. The following data is not included |
| | | in this analysis population: (1) patients |
| | | initially randomized ixekizumab; |
| | | (2) Period 4 data for patients re-randomized |
| | | to placebo at Week 60. |
| All Ixekizumab | Combined Treatment Periods. | All subjects who have at least 1 dose of |
| Safety Population | | ixekizumab, including patients in main |
| | | protocol and Protocol Addendum(2). |
| Follow-Up | Post-Treatment Follow-Up Period (Period 5) | Safety analyses for Post-Treatment Follow- |
| Population | | Up Period will be conducted on the Follow- |
| | | Up Population, defined as all randomized |
| | | subjects who received at least 1 dose of |
| | | study treatment and have entered the Post- |
| | | Treatment Follow-Up Period. Patients will |
| | | be analyzed according to the last treatment |
| A11 '' EVI I | | they received before entering Period 5. |

Abbreviations: EU = European Union.

Table RHCD.6.2. Treatment Groups and Comparisons for Each Study Period and Analysis Population

| Study Period | Analysis Population | Treatment<br>Group | Abbreviation | Comparison |
|---|---|---|---|---|
| Double-Blind<br>Treatment Period<br>(Period 2) | Intent-to-Treat Population; Per-Protocol Set; Safety Population | Ixekizumab Q4W | IXEQ4W | IXEQ4W vs. PBO |
| | | Etanercept Q1W | ETN | IXEQ4W vs. ETN |
| | | Placebo Q4W | PBO | ETN vs. PBO |
| Randomized-<br>Withdrawal Period | Double-Blind,<br>Randomized Withdrawal<br>Period Population | Ixekizumab Q4W | IXEQ4W | IXEQ4W vs. PBO |
| (Period 4) | | Placebo Q4W | PBO | |
| Combined Treatment Periods (Period 2, 3, 4) | Ixekizumab Efficacy<br>Primary Population, All<br>Ixekizumab Safety<br>Population | Ixekizumab Q4W | IXEQ4W | NA |
| Combined Treatment Periods 3 and 4 | Ixekizumab Secondary<br>Primary Population | Placebo<br>Q4W/ixekizumab<br>Q4W | PBO/IXE | NA |
| | | Etanercept<br>Q4W/ixekizumab<br>Q4W | ETN/IXE | |
| Post-Treatment Follow-Up Period (Period 5) | Follow-Up Population | Ixekizumab Q4W | IXEQ4W | No comparison |
| | | Etanercept | ETN | |
| | | Placebo Q4W | РВО | |

Abbreviations: ETN = etanercept; IXE = ixekizumab; NA = not applicable; PBO = placebo; Q1W = every week; Q4W = every 4 weeks; vs. = versus.

#### 6.1.2. Baseline Definition

For the Double-Blind Treatment Period (Period 2; ITT Populations), as well as the Combined Treatment Periods (Ixekizumab Efficacy Primary Population and Ixekizumab Efficacy Secondary Population), the baseline for efficacy and health-outcome analyses will be defined as the last available value before the first injection. In most cases, this will be the measure recorded at Week 0 (Visit 2). For efficacy and health-outcome measures, if the patient does not take any injection, the last available value on or prior to randomization date will be used.

Unless, otherwise, specified, baseline for safety during Period 2 is defined as follows: for categorical data, baseline includes all available values before the first injection at Week 0; for continuous data, baseline is the last available value before the first injection at Week 0.

Protocol Addendum I1F-MC-RHCD(2), for the Double-Blind Randomized Withdrawal Period in Subjects in EU Countries, the baseline for efficacy and health-outcome analyses will be defined as the measure recorded at Week 0 (Visit 2). For safety analysis, the baseline is defined as the last available values before the re-randomization (Week 60).

For safety analysis during the Combined Treatment Periods (Periods 2, 3, and 4; Ixekizumab Safety Population): patients who were initially randomized to ixekizumab at Week 0, baseline period is defined as the time from Visit 1 to the date/time of the first injection. For patients initially randomized to placebo or etanercept, baseline is defined as last available value prior to first dose of ixekizumab. For patients who get re-randomized to placebo during the Double-Blind Randomized Withdrawal Period (Protocol Addendum RHCD[2]), they may enter the rescue arm on ixekizumab after relapse. The baseline for this second ixekizumab exposure period will be the last nonmissing value during the placebo exposure period and prior to the ixekizumab injection. For patients who had 2 separate ixekizumab exposures, the baseline for the shift tables and standardized growth analyses in both exposure periods will be defined as the baseline for the first ixekizumab exposure period.

For the Post-Treatment Follow-Up Period (Period 5), the baseline is defined as the last nonmissing assessment on or prior to entering Period 5, that is, on or prior to Week 108, or ETV.

Change from baseline will be calculated as the visit value of interest minus the baseline value. If all baseline values are missing for a particular variable, then the change from baseline and the percent improvement from baseline will not be calculated.

# 6.1.3. Analysis Methods

#### 6.1.3.1. Double-Blind Treatment Period (Period 2): Main Protocol

The primary analysis method for categorical data for treatment group comparisons will be Fisher's exact test. The difference of the proportions and the 95% CI of the difference will be included.

Secondary analyses for the primary efficacy measures, PASI 75 and sPGA(0,1), and other categorical efficacy and health outcome measures, will be conducted using a logistic regression analysis with treatment group, region, baseline sPGA score (severity of Ps), and baseline weight category (<25 kg,  $\ge25$  to  $\le50$  kg, or >50 kg) as factors. The odds ratio and the corresponding 95% CI will be reported.

The analyses for the continuous efficacy and health-outcome variables will be made using analysis of covariance (ANCOVA) and mixed model for repeated measures (MMRM) analysis. The ANCOVA model includes treatment group, region, baseline sPGA score, baseline weight category, and baseline value. Type III sums of squares for the least-squares means will be used for the statistical comparison; the 95% CI will be reported.

When the MMRM is used, the model will include treatment, region, baseline sPGA score, baseline weight category, baseline value, visit, treatment-by-visit, and baseline-by-visit interactions as fixed factors. The covariance structure to model the within-subject errors will be unstructured. The Kenward-Roger method will be used to estimate the denominator degrees of freedom. Type III tests for the least-squares means will be used for the statistical comparison; the 95% CI will be reported. Treatment comparisons at Week 12 and all other postbaseline visits will be reported.

If the unstructured covariance matrix results in a lack of convergence, the heterogeneous Toeplitz covariance structure, followed by the heterogeneous autoregressive covariance structure, followed by the compound symmetry will be used. This order is specified according to a decreasing number of covariance parameters in the structure. The sandwich estimator (Diggle et al. 1994) for the covariance estimation will be used by specifying the EMPIRICAL option in SAS PROC MIXED. When sandwich estimation is used, the Kenward-Roger approximation for denominator degrees of freedom cannot be used. Instead, the DDFM= BETWITHIN option will be used to estimate denominator degrees of freedom.

Fisher's exact test will be used for all adverse events (AEs), baseline characteristics, discontinuation, and other categorical safety data. The continuous baseline characteristics will be analyzed using an analysis of variance (ANOVA) model with treatment as a factor. Continuous vital sign data and laboratory values will be analyzed by an ANCOVA with treatment and baseline value in the model.

### 6.1.3.2. Double-Blind Treatment Period (Period 2): Protocol Addendum(2)

The analysis method for categorical data for treatment group comparisons will be Fisher's exact test. The difference of the proportions and the 95% CI of the difference will be included.

Fisher's exact test will be used for all AEs, baseline characteristics, discontinuation, and other categorical safety data. The continuous baseline characteristics will be analyzed using an ANOVA model with treatment as a factor. Continuous vital sign data and laboratory values will be analyzed by an ANCOVA with treatment and baseline value in the model.

#### 6.1.3.3. Combined Treatment Periods

Data for the combined treatment periods will be summarized using descriptive statistics.

#### 6.1.3.4. Double-Blind Randomized Withdrawal Period (Period 4)

The time to relapse (loss of response;  $sPGA \ge 2$ ) during Double-Blind, Randomized Withdrawal Period (Period 4) is defined as:

Time to relapse (days)

=  $date\ of\ first\ sPGA \ge 2\ during\ Period\ 4 - date\ of\ Week\ 60\ rerandomization\ +\ 1$ 

If a patient has not experienced relapse by completion or early discontinuation of Period 4, the patient will be censored at the date of his/her last visit during Period 4.

The number of patients at risk and experiencing a relapse event by each scheduled visit during Period 4 will be presented by treatment group. The Kaplan-Meier estimate of the proportion of patients relapsing will be presented for each visit. Treatment group comparisons will be performed using the log-rank test. For each treatment group, a Kaplan-Meier plot of the time to relapse will be provided.

The analysis method for categorical data for treatment group comparisons will be Fisher's exact test. The difference of the proportions and the 95% CI of the difference will be included.

Fisher's exact test will be used for all AEs, baseline characteristics, discontinuation, and other categorical safety data. The continuous baseline characteristics will be analyzed using an ANOVA model with treatment as a factor. Continuous vital sign data and laboratory values will be analyzed by an ANCOVA with treatment and baseline value in the model.

### 6.2. Adjustments for Covariates

Clinical Protocol RHCD (main study), the randomization at the beginning of the Double-Blind Treatment Period (Period 2) is stratified by geographic region. With the exception of the primary analysis (that is, Fisher's exact test), efficacy and health-outcome analyses during Period 2 will include geographic region and baseline weight category in the analysis models.

In general, when an MMRM is to be used for analyses, baseline value and baseline-by-visit interactions will be included as covariates; when an ANCOVA is to be used for analyses, baseline value will be included as a covariate.

Protocol Addendum RHCD(2), for the double-blind randomized withdrawal period (Period 4), subjects were re-randomized to ixekizumab according to their weight at the time of re-randomization. The stratification factor, weight at the time of re-randomization, will not be included in the analysis models.

# 6.3. Handling of Dropouts or Missing Data

The methods for imputation of missing data to be used in this study are in accordance with the precedent set in other Phase 3 Ps trials (Leonardi et al. 2008; Papp et al. 2008) and ixekizumab Phase 3 pivotal studies (RHAZ, RHBA, and RHBC).

# 6.3.1. Nonresponder Imputation (NRI)

Analysis of categorical efficacy and health-outcome variables will be assessed using a NRI method. Subjects will be considered nonresponders for the NRI analysis if they do not meet the clinical response criteria or have missing clinical response data at the analysis time point. Randomized patients without at least 1 postbaseline observation will also be defined as nonresponders for the NRI analysis.

# 6.3.2.Last Observation Carried Forward (LOCF)

An LOCF analysis will be performed on all continuous efficacy and health-outcome variables as a secondary analysis. For patients having missing data at the visit, the last nonmissing postbaseline observation before the missing data will be carried forward to the corresponding

time point for evaluation. Subjects who have a baseline and at least 1 postbaseline observation will be included for evaluation.

#### 6.4. Multicenter Studies

This study will be conducted by multiple investigators at multiple sites internationally. Data from the sites are pooled within geographic region. Unless, otherwise, specified, geographic region will be included in the statistical analysis models. The co-primary endpoints at Week 12 will be summarized by center using descriptive statistics only.

### 6.5. Multiple Comparisons/Multiplicity

A multiple testing strategy for the primary and major secondary objectives will be implemented to control the family-wise type I error rate at a 2-sided  $\alpha$  level of 0.05. The primary and key secondary comparisons will be tested by using the primary analysis method, Fisher's exact test, with an NRI missing-data imputation approach.

A gatekeeping approach will be used for multiple comparisons to control the family-wise error rate. To assess whether ixekizumab Q4W is superior to placebo, the following endpoints will be tested:

- Primary 1: Proportion of subjects achieving PASI 75 at Week 12
- Primary 2: Proportion of subjects achieving sPGA (0,1) at Week 12
- Secondary 1: Proportion of subjects achieving PASI 90 at Week 12
- Secondary 2: Proportion of subjects achieving sPGA (0) at Week 12
- Secondary 3: Proportion of subjects achieving PASI 100 at Week 12
- Secondary 4: Proportion of subjects achieving ≥4 point improvement for subjects who had a baseline Itch numeric rating scale (NRS) ≥4 at Week 12
- Secondary 5: Proportion of subjects achieving PASI 75 at Week 4
- Secondary 6: Proportion of subjects achieving sPGA (0,1) at Week 4

The Primary 1 will first be tested at 2-sided  $\alpha$ =0.05. If successful, the test for Primary 2 will be performed at 2-sided  $\alpha$ =0.05. Otherwise, the test will stop. If the Primary 2 endpoint is successful, the Secondary 1 endpoint will be tested. The test will continue to the last endpoint if all the prior tests are successful. If a test is not successful, all subsequent tests will not be tested.

# 6.6. Use of an "Efficacy Subset" of Patients

The PPS is defined above in Section 6.1.1 and is an efficacy subset of patients. The analysis of the co-primary endpoints will be repeated using the PPS.

# 6.7. Patient Disposition

Patient flow will be summarized from entered to randomized to completion, and analysis populations will be listed and summarized by treatment group.

Patient disposition from study will be listed and summarized with reasons for disposition for the ITT Population and the Follow-Up Population, respectively.

Patient disposition from study treatment will be listed and summarized for the ITT Population for the Double-Blind Treatment Period (Period 2) and the ITT Population of etanercept approved countries for the Double-Blind Treatment Period (Period 2) in Protocol Addendum RHCD(2) with reasons for disposition, which will be compared between and among treatment groups using Fisher's exact test.

Time to study treatment discontinuation due to any reason (in weeks) will be summarized by treatment group and graphically presented using Kaplan-Meier technique. The log-rank test will be used to compare time to study treatment discontinuation between treatment groups. Time to study treatment discontinuation will be calculated as:

$$\frac{\textit{Date of study treatment discontinuation} - \textit{Date of first dose} + 1}{7}$$

If the date of first dose is missing, the date of randomization will be used. Patients completing the study treatment will be censored at the date of completion.

Patient allocation by region, country, and center/site will be summarized with number of patients who entered the study, number of ITT patients for each dosing regimen, number of patients discontinued from study treatment, and number of patients discontinued from study.

#### 6.8. Patient Characteristics

### 6.8.1. Demographics and Baseline Characteristics

Patient demographic variables and baseline characteristics will be summarized by treatment group and, overall, for the ITT Population and the ITT Population – etanercept-approved countries and the Double-Blind, Randomized Withdrawal Period Population. The continuous variables will be summarized using descriptive statistics, and the categorical variables will be summarized using frequency counts and percentages. The comparisons between treatment groups will be conducted using the Fisher's exact test for categorical data, and an analysis of variance model with treatment group as a factor for continuous data.

The following demographic variables and baseline characteristics will be summarized:

- Age (years)
- Age category: <12 years; and ≥12 years
- Gender
- Ethnicity
- Race
- Weight (kg): measured at Visit 2
- Weight Category:  $\langle 25 \text{ kg}; \geq 25 \text{ to } \leq 50 \text{ kg}; \text{ and } \rangle \leq 50 \text{ kg}$
- Height (cm): measured at Visit 1
- Body mass index (BMI) (kg/m²): BMI will be calculated as:

$$BMI(kg/m^2) = \frac{Weight(kg)}{(Height(m))^2}$$

• Habits (only for subjects ≥12 years old)

- o Caffeine consumption: never; current; former
- o Alcohol consumption: never; current; former
- o Tobacco consumption: never; current; former
- Country: Argentina, Canada, Czech Republic, France, Germany, Hungary, Mexico, Netherlands, Poland, Russia, Spain, United States
- Geographic region:
  - o United States/Canada (United States, Canada)
  - European Union (Czech Republic, France, Germany, Hungary, Netherlands, Poland, Spain)
  - o Rest of the world (Argentina, Mexico, Russia)
- Geographic region:
  - United States/Canada (United States, Canada)
  - o Other
- Previous systemic therapy: never used; nonbiologic only; biologic only; biologic and nonbiologic.
  - o Nonbiologics are defined as: methotrexate; cyclosporine; corticosteroids; acitretin; fumaric-acid derivatives; apremilast; or other nonbiologics
  - O Biologics are defined as: efalizumab; ustekinumab; infliximab; etanercept; alefacept; adalimumab; golimumab; certolizumab pegol; secukinumab; or other biologics
- Tuberculosis (TB) exposure: positive; negative
- Age at Ps onset (in years)
- Duration of Ps (in years): will be calculated using the date of Ps onset (as recorded on the Prespecified Medical History Psoriasis electronic case report form [eCRF] page) as follows:

 $Duration of psoriasis (years) = \frac{Date of informed consent - Date of psoriasis onset}{365.25}$ 

- Age at psoriasis diagnosis (in years)
- Duration of psoriasis diagnosis (in years): will be calculated using the date of psoriasis diagnosis (as recorded on the Prespecified Medical History Psoriasis eCRF page) as follows:

Duration of psoriasis diagnosis (years)  $= \frac{Date\ of\ Visit\ 2 - Date\ of\ psoriasis\ diagnosis}{365.25}$ 

- Baseline sPGA
- Baseline sPGA category: 3; 4; and 5
- Baseline sPGA category: 3; and combined 4 or 5
- Baseline PASI score
- Baseline PASI category: <20; and  $\ge 20$
- Baseline BSA (%)
- Baseline BSA category: <20%; and ≥20%
- Nail psoriasis: yes; and no

- Baseline Nail Psoriasis Severity Index (NAPSI) score
- Scalp psoriasis: yes; and no
- Baseline Psoriasis Severity Index (PSSI) score
- Palmoplantar psoriasis: yes; and no
- Baseline Palmoplantar Psoriasis Severity Index (PPASI) score
- Baseline Itch NRS score
- Baseline Itch NRS category: <4; and ≥4
- Baseline Children's Dermatology Life Quality Index (CDLQI) total score
- Baseline Dermatology Life Quality Index (DLQI) total score
- Patient's Global Assessment of Disease Severity (PatGA)
- PatGAcategory: 0; 1; 2; 3; 4; and 5
- Baseline Children's Depression Rating Scale, Revised (CDRS-R)
- Baseline CDRS-R category: ≤28; 29-39; and ≥40
- Baseline Columbia Suicide Severity Rating Scale (C-SSRS)
- Binary questions on psoriasis location
- Tanner Stage Scale

By-patient listings of demographic and baseline characteristics, respectively, for the ITT Population will be provided.

## 6.8.2. Historical Illnesses and Preexisting Conditions

Historical illnesses and preexisting conditions will be classified using the latest version of the Medical Dictionary for Regulatory Activities (MedDRA).

Historical illness/condition is defined as the condition/event recorded on the Pre-Existing Conditions and Medical History eCRF page or on the Prespecified Medical History eCRF page with an end date prior to the date of informed consent.

A preexisting condition is defined as the condition/event recorded on the Pre-Existing Conditions and Medical History eCRF page or on the Prespecified Medical History eCRF page with a start date prior to the date of informed consent, and no end date (that is, the event is ongoing) or an end date on or after the date of informed consent. Adverse events occurring prior to the date of first study injection will also be reported. Note that, if a preexisting condition worsens in severity on or after the date of informed consent, it will be recorded as an AE on Adverse Events eCRF page from the date of worsening onward.

The following summaries will be provided for both ITT Populations:

- The number and percentage of patients with historical illnesses by treatment group and overall, by System Organ Class (SOC) and preferred term (PT).
- The number and percentage of patients with preexisting conditions and adverse events occurring prior to the first dose, by treatment group and overall, by SOC and PT.
- The number and percentage of patients with prespecified medical history (hypertension; diabetes mellitus, Type I; diabetes mellitus, Type II; dyslipidemia; psoriatic arthritis;

inflammatory bowel disease [Crohn's disease and uncreative colitis]), by treatment group and overall.

For a condition/event that is gender-specific (as defined by MedDRA), the denominator and computation of the percentage will include only patients from the given gender. The comparisons among treatment groups will be conducted using Fisher's exact test.

By-patient listings of historical illnesses and preexisting conditions, respectively, for the ITT Populations will be provided.

### 6.9. Treatment Compliance

By-patient listings of randomization schedules and study drug dispensed (include the clinical trial (CT) Lot number), respectively, for the ITT Populations will be provided.

Throughout treatment periods, randomized patients will record information in a Study Drug Administration Log (captured in the Exposure as Collected eCRF page), including the date, time, and anatomical location of administration of investigational product, syringe number, who administered the investigational product, and the reason if the investigational product was not fully administered.

Treatment compliance for each patient per period will be calculated as:

Treatment compliance (%) = 
$$100 \times \frac{Total\ number\ of\ injections\ administered}{Total\ number\ of\ injections\ prescribed}$$

#### Clinical Protocol RHCD:

- For patients who complete Period 2 and receive ixekizumab 20 mg or 40 mg or placebo for ixekizumab 20 mg or 40 mg, the number of injections prescribed (that is, expected) during Period 2 will be equal to 3 (1 injection at Week 0 and 1 injection at Weeks 4 and 8). For patients who complete Period 2 and receive ixekizumab 80 mg or placebo for ixekizumab 80 mg, the number or injections prescribed during Period 2 will be equal to 4 (2 injections at Week 0 and 1 injection at Weeks 4 and 8).
- For patients who discontinue during Period 2, the number of injections prescribed during Period 2 can be derived from the IWRS study drug dispense dataset.

#### Protocol Addendum RHCD(2):

- The number of injections for ixekizumab group and placebo group are the same as in the main study ITT Population. For patients who complete Period 2 and receive etanercept, the number of injections prescribed during period 2 will be equal to 12 (1 injection every week from Week 0 to Week 11).
- For patients who discontinue during Period 2, the number of injections prescribed during Period 2 can be derived from the IWRS study drug dispense dataset.

A patient will be considered overall compliant with study treatment within each treatment period if he/she misses no more than 20% of the expected doses, does not miss 2 consecutive doses, and

does not overdose (that is, take more injections at the same time point than specified in the protocol).

Patient treatment compliance, by Period 2, will be summarized. The comparisons between treatment groups during Period 2 will be conducted using Fisher's exact test.

A by-patient listing of study treatment administration and compliance for the ITT Population will be provided.

## 6.10. Previous and Concomitant Therapy

Medication/therapy will be classified into Anatomical Therapeutic Chemical (ATC) drug classes using the latest version of the World Health Organization (WHO) Drug Dictionary.

A by-patient listing of previous and concomitant therapy, and a by-patient listing of previous Ps therapy for the ITT Population will be provided.

## 6.10.1. Previous Therapy

Previous therapy is defined as therapy that starts and ends prior to the date of first dose of study treatment in the Double-Blind Treatment Period (Period 2). If therapy start and/or end dates are missing or partial, the dates will be compared as far as possible with the date of first dose of study treatment in Period 2. If there is clear evidence to suggest that the therapy stopped prior to the first dose of study treatment in Period 2, the therapy will be assumed to be previous dose only. The comparisons will be conducted using Fisher's exact test.

The following summaries will be provided for both ITT populations:

- Previous therapy (captured in the Prior Therapy: Psoriasis eCRF page and Concomitant Therapy eCRF page) by WHO ATC Level 4 and WHO PT.
- Previous Ps therapy captured in the Prior Therapy: Psoriasis eCRF page to be summarized according to type (topical prescription therapy, topical nonprescription therapy, nonbiologic systemic agent, biologic agent, nonbiologic nonsystemic agent, phototherapy) and therapy. The previous biologic agent will be further classified as tumor necrosis factor- (TNF-) α inhibitor (includes infliximab, etanercept, adalimumab, golimumab, certolizumab pegol), interleukin- (IL-) 12/23 inhibitor (includes ustekinumab), IL-17 inhibitor (includes secukinumab and brodalumab), and other (includes efalizumab, alefacept, or other biological agents).
- The number and percentage of patients with each reason for discontinuation of previous Ps therapy to be summarized by type and therapy.

# 6.10.2. Concomitant Therapy

Concomitant therapy is defined as the therapy that starts before, on, or after the first day of study treatment in the defined treatment period and before the last visit date in the treatment period, and continues into the treatment period, that is, either no end date (the therapy is ongoing) or an end date on or after the first day of study treatment in treatment period. Note, concomitant

therapy will belong to a treatment period if the therapy starts and ends on the exact same day as the first day of study treatment of the treatment period.

Concomitant therapy during period 2 will be summarized by both ITT populations. Concomitant therapy for Period 2 is defined as the therapy that starts before, on, or after the first day of study treatment of Period 2 and before the last visit date of Period 2, and continues into Period 2, that is, there is either no end date (the therapy is ongoing) or there is an end date on or after the first day of study treatment of Period 2. Note that concomitant therapy will belong to Period 2 if the therapy starts and ends on the exact same day as the first day of study treatment of Period 2.

Concomitant therapy during period 4 will be summarized by the Double-Blind Randomized Withdrawal Period Population. Concomitant therapy for Period 4 is defined as the therapy that starts before, on, or after the first day of study treatment of Period 4 and before the last visit date of Period 4, and continues into Period 4, that is, there is either no end date (the therapy is ongoing) or there is an end date on or after the first day of study treatment of Period 4. Note that concomitant therapy will belong to Period 4 if the therapy starts and ends on the exact same day as the first day of study treatment of Period 4.

The comparisons will be conducted using Fisher's exact test.

The following summaries will be provided:

- Concomitant therapy by WHO ATC Level 4 and WHO PT
- The number and percentage of patients taking concomitant therapy of a topical product to be summarized for topical and topical steroid therapies, respectively, by WHO ATC Level 4 and WHO PT. The definition of concomitant topical therapy can be found in Appendix 1. Please refer to I1F-MC-RHCD Clinical Protocol Section 7.7 for concomitant therapies permitted during the study.
- The number and percentage of patients who received premedication for allergic reaction/hypersensitivity captured in the Allergic/Hypersensitivity Reaction Follow-Up eCRF page.

If a partial or completely missing medication start date/time or end date/time is present, the following imputation rules will be utilized in the analysis:

- For the start date:
  - o If year, month, and day are missing, then use the earlier of the patient's first visit date or the consent date.
  - o If either month or month and day are missing, then use January 1.
  - o If only day is missing, impute the first day of the month.
- For the start time:
  - o Impute as 23:59
- For the end date:
  - o If year, month, and day are missing, then use the patient's last visit date.
  - o If either month or month and day are missing, then use December 31.
  - o If only day is missing, then use the last day of the month.

- o The imputed date will not be beyond the patient's last visit date.
- For the end time:
  - o Impute as 23:59.
- If there is any doubt, the medication will be flagged as concomitant.

# 6.11. Efficacy Analyses

Table RHCD.6.3 includes the description and derivation of the primary and secondary efficacy outcomes. Table RHCD.6.4 includes the description of primary and secondary efficacy analyses.

 Table RHCD.6.3.
 Description and Derivation of Primary and Secondary Efficacy Outcomes

| Measure | Description | Variable | Derivation / Comment | Imputation Approach if with Missing Components |
|---|---|---|---|---|
| PASI | Psoriasis Area and Severity Index (PASI): | PASI score | The composite PASI score is calculated by multiplying | If any individual score |
| | combines assessments of the extent of body- | | the sum of the individual-severity scores for each area | is missing, the PASI |
| | surface involvement in 4 anatomical regions | | by the weighted area-of-involvement score for that | score will not be |
| | (head and neck, trunk, arms, and legs) and | | respective area, and then summing the 4 resulting | calculated, hence, |
| | the severity of scaling (S), redness (R), and | | quantities as follows: | missing. |
| | plaque induration/infiltration (thickness, T) | | PASI = 0.1(Rh + Th + Sh)Ah + 0.2(Ru + Tu + Su)Au + | |
| | in each region, yielding an overall score of 0 | | 0.3(Rt + Tt + St)At + 0.4(Rl + Tl + Sl)Al, where: | |
| | for no psoriasis to 72 for the most severe | | Rh, Ru, Rt, Rl = redness score of plaques on the | |
| | disease (Fredriksson and Pettersson 1978). | | head, upper limb, trunk, and lower limb, scored | |
| | Severity is rated for each index (R, S, T) on a | | 0-4 respectively; | |
| | 0-4 scale (0 for no involvement up to 4 for | | Th, Tu, Tt, Tl = thickness score of plaques on the | |
| | severe involvement): | | head, upper limb, trunk, and lower limb, scored | |
| | 0 = none | | 0-4 respectively; | |
| | 1 = slight | | Sh, Su, St, $Sl = scaliness$ score of plaques on the | |
| | 2 = mild | | head, upper limb, trunk, and lower limb, scored | |
| | 3 = moderate | | 0-4 respectively; | |
| | 4 = severe | | Ah, Au, At, Al = numerical value translation of % | |
| | The body is divided into four anatomical | | area of psoriatic involvement score for the head, | |
| | regions comprising the head (h), upper limb | | upper limb, trunk, and lower limb, respectively. | |
| | (u), trunk (t), and lower limb (l). In each of | | PASI scores are treated as a continuous score, with | |
| | these areas, the fraction of total body surface | | 0.1 increments within these values. | |
| | area affected is graded on a 0-6 scale (0 for | PASI change | Calculated as: observed PASI – baseline PASI | Missing if baseline or |
| | no involvement up to 6 for 90% - 100% | from baseline | | observed value is |
| | involvement): | | | missing. |
| | 0 = 0% (clear) | PASI percent | Calculated as: | Missing is baseline or |
| | 1 = >0% to < 10% 2 = 10% to < 30% | improvement | D | observed value is |
| | 2 = 10% to < 30%<br>3 = 30% to < 50% | from baseline | Percent improvement from baseline $= 100 \times \frac{Baseline\ PASI - Observed\ PASI}{Baseline\ PASI}$ | missing |
| | 4 = 50% to $< 70%$ | | = 100 × ————————————————————————————————— | 6 |
| | 5 = 70% to < 90% | | If a patient has experienced an improvement, this | |
| | 6 = 90% to 100% | | measure will be positive. If a patient has experienced a | |
| | The various body regions are weighted to | | worsening in the condition, this measure will be | |
| Measure | Description | Variable | Derivation / Comment | Imputation Approach if with Missing Components |
|---|---|---|---|---|
| | reflect their respective proportions of body | | negative. | |
| | surface area (BSA). | PASI 75 (coprimary) | A clinically meaningful response; at least a 75% improvement in PASI score from baseline. | Missing is baseline or observed value is missing |
| | | PASI 90 | Higher level of clearance; at least a 90% improvement in PASI score from baseline. | Missing is baseline or observed value is missing |
| | | PASI 100 | Complete resolution of plaque psoriasis; a 100% improvement in PASI score from baseline. | Missing is baseline or observed value is missing |
| sPGA | Static Physician Global Assessment (sPGA):<br>the physician's global assessment of the<br>patient's psoriasis lesions at a given time | sPGA score | Range from 0 to 5: clear (0); minimal (1); mild (2); moderate (3); severe (4); or very severe (5). | Single item, missing if missing |
| | point (EMA 2004 [WWW]). Plaques are assessed for induration, erythema, and scaling, and an overall rating of psoriasis | sPGA (0,1) (coprimary) | An sPGA assessed as either 0 or 1, which represents a clinically meaningful response of minimal plaque severity or complete resolution of plaque psoriasis. | Missing if sPGA is missing |
| (0 | severity is given using the anchors of clear (0), minimal (1), mild (2), moderate (3), severe (4), or very severe (5). | sPGA (0) | An sPGA assessed as 0, which represents a clinically important endpoint indicating complete resolution of plaque psoriasis. | Missing if sPGA is missing |
| BSA | Percentage of BSA: The investigator will evaluate the percentage involvement of psoriasis on each patient's BSA on a continuous scale from 0% (no involvement) | BSA | Collected as a single scale as part of PASI electronic case report form (eCRF) page. Range from 0% to 100%. | Missing is baseline or observed value is missing |
| | to 100% (full involvement), in which 1% corresponds to the size of the patient's hand (including the palm, fingers, and thumb) (Van Voorhees et al. 2009). | BSA change from baseline | Calculated as: observed BSA – baseline BSA | Missing is baseline or observed value is missing |

| Measure | Description | Variable | Derivation / Comment | Imputation Approach if with Missing Components |
|---|---|---|---|---|
| NAPSI | | NAPSI score | The NAPSI score of a nail is the sum of scores in nail bed and nail matrix from each quadrant (maximum of 8). Each nail is evaluated, and the sum of all the fingernails and toenails is the total NAPSI score (range, 0 to 160), usually indicated as NAPSI score. | For each nail, if either bed or matrix score is missing or not done, the score for that nail is missing. If <50% of the nail scores from 20 nails are missing, the imputation will be performed by using the average score of the remaining nails. If ≥50% of the nail scores are missing, the NAPSI score will be left as missing. |
| | | NAPSI score<br>change from<br>baseline<br>NAPSI score = 0 | Calculated as: observed NAPSI – baseline NAPSI A NAPSI response is defined as a NAPSI score of 0, which is also referred to as nail clearance. | Missing if baseline or observed value is missing Missing if NAPSI score is missing. |
| PSSI* | Psoriasis Scalp Severity Index (PSSI): will be used if the patient has scalp psoriasis at baseline. The scalp will be assessed for erythema (redness), induration (hardness), and desquamation (shedding of skin) and percentage of area affected as follows: Erythema, Induration and Desquamation: 0 = Absent | PSSI score | The PSSI score is a composite score derived from the sum of the scores for erythema, induration and desquamation multiplied by the score for the extent of scalp area involved (percent of scalp involved). The range is 0 to 72. | If any individual score is missing, the PSSI score will not be calculated, hence, missing. |

| Measure | Description | Variable | Derivation / Comment | Imputation Approach if with Missing Components |
|---|---|---|---|---|
| | 1 = Slight | PSSI score | Calculated as: observed PSSI – baseline PSSI | Missing if baseline or |
| | 2 = Moderate | change from | | observed value is |
| | 3 = Severe | baseline | | missing |
| | 4 = Severest Possible | | | |
| | Percent of Scalp Involved: | | | |
| | 1 = <10% | PSSI score = 0 | A DCCI magnetic defined as a DCCI sages of 0 which | Missing if DCCI asons |
| | 2 = 10% - 29% | PSS1 score = 0 | A PSSI response is defined as a PSSI score of 0, which is also referred to as scalp clearance. | Missing if PSSI score is missing. |
| | 3 = 30% - 49% | | is also referred to as scarp clearance. | is missing. |
| | 4 = 50% - 69% | | | |
| | 5 = 70% - 89% | | | |
| | 6 = 90% - 100% | | | |
| PPASI | Palmoplantar Psoriasis Area and Severity | PPASI score | The PPASI score is a composite score derived from the | If any individual score |
| | Index (PPASI): will be used if the patient has | | sum scores for erythema, induration, and desquamation | is missing, the PPASI |
| | palmoplantar psoriasis at baseline. Both the | | multiplied by a score for the extent of palm and sole | score will not be |
| | palms and soles on each hand and foot will | | area involvement. The range is 0 to 72. | calculated, hence, |
| | be individually assessed for erythema, | | PPASI = 0.2(Erp + Irp + Drp)Arp + 0.2(Elp | missing. |
| | induration, desquamation and percentage of | | +Ilp+Dlp)Alp + 0.3(Ers + Irs+Drs)Ars + 0.3(Els | |
| | area affected as follows: | | +Ils+Dls)Als, where: | |
| | Erythema (E), Induration (I), and | | Erp, Elp, Ers, Els = Erythema score of plaques on | |
| | Desquamation (D): | | the right palm (rp), left palm (lp), right sole (rs), | |
| | 0 = None | | left sole (ls), scored 0-4 respectively; | |
| | 1 = Slight | | Irp, Ilp, Irs, Ils = Induration score of plaques on the | |
| | 2 = Moderate | | right palm (rp), left palm (lp), right sole (rs), left | |
| | 3 = Severe | | sole (ls), scored 0-4 respectively; | |
| | 4 = Very Severe | | Drp, Dlp, Drs, Dls = Desquamation score of plaques | |
| | Percent of Palm and Sole Area Covered: | | on the right palm (rp), left palm (lp), right sole | |
| | 0 = None | | (rs), left sole (ls), scored 0-4 respectively; | |
| | 1 = <10% | | Arp, Alp, Ars, Als = numerical value translation of | |
| | 2 = 10% - 29% | | % area covered for the right palm, left palm, right | |
| | 3 = 30% - 49% | | sole, and left sole, respectively. | |
| | 4 = 50% - 69% | | | |
| | 5 = 70% - 89% | PPASI change | Calculated as: observed PPASI – baseline PPASI | Missing if baseline or |

| Measure | Description | Variable | Derivation / Comment | Imputation Approach if with Missing Components |
|---|---|---|---|---|
| | 6 = 90% - 100% | from baseline | | observed value is missing |
| | | PPASI percent improvement from baseline | Calculated as: Percent improvement from baseline $= 100 \times \frac{Baseline\ PPASI - Observed\ PPASI}{Baseline\ PPASI}$ If a patient has experienced an improvement, this measure will be positive. If a patient has experienced a worsening in the condition, this measure will be negative. | Missing is baseline or observed value is missing |
| | | PPASI 50 | At least a 50% improvement in PPASI score from baseline. | Missing is baseline or observed value is missing |
| | | PPASI 75 | At least a 75% improvement in PPASI score from baseline. | Missing is baseline or observed value is missing |
| | | PPASI 100 | A 100% improvement in PPASI score from baseline. | Missing is baseline or observed value is missing |
| Binary<br>questions<br>on<br>psoriasis<br>location | The presence of visible psoriasis on the following locations will be noted: 1. Face 2. Nail 3. Axilla 4. Genitals 5. Perianal region | Binary<br>questions on<br>psoriasis<br>location | Binary responses (yes/no) will be noted to determine the presence of visible psoriasis on each of the 5 locations. | Missing if the response is missing |

<sup>\*</sup> A previous version of PSSI questionnaire was sent to the sites with percent of scalp involved range 1 to 6. Some sites still enter 0 to represent none scalp psoriasis involvement. The range of the total score is still 0-72, so that there is no impact on planned analyses.

 Table RHCD.6.4.
 Description of Primary and Secondary Efficacy Analyses

| Measure | Variable | Analysis<br>(Method) | Population | Comparison/Time Point | Analysis Type |
|---|---|---|---|---|---|
| PASI | PASI 75 (co-primary) | Fisher's exact test<br>with NRI (primary<br>analysis)<br>Logistic regression<br>with NRI | ITT Population | Ixekizumab Q4W vs. placebo<br>at Week 12 and all other<br>postbaseline visits during<br>Period 2. | Primary analysis is Fisher's exact test with NRI for ITT Population comparing ixekizumab and placebo at Week 12. Secondary analysis is logistic regression with NRI for ITT Population comparing ixekizumab and placebo at Week 12. |
| | | Fisher's exact test<br>with NRI<br>Logistic regression<br>with NRI | Per-Protocol Set | Ixekizumab Q4W vs. placebo<br>at Week 12 and all other<br>postbaseline visits during<br>Period 2. | Additional analysis for co-primary outcomes. |
| | PASI 75 | Fisher's exact test with NRI | ITT Population | Ixekizumab Q4W vs. placebo at Week 4. | Gated secondary analysis |
| | | Logistic regression with NRI | ITT Population -<br>Etanercept-approved<br>countries | All pairwise comparisons at Week 12 and all other postbaseline visits during Period 2. | Other secondary analysis |
| | PASI 90 | Fisher's exact test<br>with NRI<br>Logistic regression<br>with NRI | ITT Population | Ixekizumab Q4W vs. placebo<br>at Week 12 and all other<br>postbaseline visits during<br>Period 2. | Gated secondary analysis comparing ixekizumab Q4W vs. Placebo at Week 12. |
| | PASI 100 | Fisher's exact test<br>with NRI<br>Logistic regression<br>with NRI | ITT Population | Ixekizumab Q4W vs. placebo<br>at Week 12 and all other<br>postbaseline visits during<br>Period 2. | Gated secondary analysis comparing ixekizumab Q4W vs. Placebo at Week 12. |
| | PASI 50 | Fisher's exact test<br>with NRI<br>Logistic regression<br>with NRI | ITT Population | Ixekizumab Q4W vs. placebo<br>at Week 12 and all other<br>postbaseline visits during<br>Period 2. | Other secondary analysis |

| Measure | Variable | Analysis<br>(Method) | Population | Comparison/Time Point | Analysis Type |
|---|---|---|---|---|---|
| | Change from baseline, percent improvement | ANCOVA with<br>LOCF;<br>MMRM | ITT Population | Ixekizumab Q4W vs. placebo<br>at Week 12 and all other<br>postbaseline visits during<br>Period 2. | Other secondary analysis |
| | PASI 75<br>PASI 90<br>PASI 100 | Summarize | Ixekizumab Efficacy<br>Primary Population | At all postbaseline visits during the Combined Treatment Periods (Periods 2, 3, and 4). | Other secondary analysis/<br>Exploratory analysis |
| | | | Ixekizumab Efficacy<br>Secondary Population | At all postbaseline visits during the Combined Treatment Periods (Periods 3 and 4). | Exploratory analysis |
| | | Fisher's exact test | Double-Blind,<br>Randomized<br>Withdrawal<br>Population | Ixekizumab Q4W vs. placebo at all postbaseline visits during Period 4. | Other secondary analysis |
| sPGA | sPGA (0,1)<br>(co-primary) | Fisher's exact test<br>with NRI (primary<br>analysis);<br>Logistic regression<br>with NRI | ITT Population | Ixekizumab Q4W vs. placebo<br>at Week 12 and all other<br>postbaseline visits during<br>Period 2. | Primary analysis is Fisher's exact test with NRI for ITT Population comparing ixekizumab and placebo at Week 12. Secondary analysis is logistic regression with NRI for ITT Population comparing ixekizumab and placebo at Week 12. |
| | | Fisher's exact test<br>with NRI<br>Logistic regression<br>with NRI | Per-Protocol Set | Ixekizumab Q4W vs. placebo<br>at Week 12 and all other<br>postbaseline visits during<br>Period 2. | Additional analysis for co-primary outcomes. |
| | sPGA (0,1) | Fisher's exact test with NRI | ITT Population | Ixekizumab Q4W vs. placebo at Week 4. | Gated secondary analysis |
| | | Logistic regression with NRI | ITT Population -<br>Etanercept approved | Ixekizumab Q4W vs. etanercept at Week 12 and all | Other secondary analysis |

| Measure | Variable | Analysis<br>(Method) | Population | Comparison/Time Point | Analysis Type |
|---|---|---|---|---|---|
| | | | countries | other postbaseline visits during Period 2. | |
| | | | Double-Blind,<br>Randomized<br>Withdrawal Period<br>Population | Ixekizumab Q4W vs. placebo<br>at Week 108 and all other<br>postbaseline visits during<br>Period 4. | Other secondary analysis |
| | sPGA (0) | Fisher's exact test<br>with NRI<br>Logistic regression<br>with NRI | ITT Population | Ixekizumab Q4W vs. placebo<br>at Week 12 and all other<br>postbaseline visits during<br>Period 2. | Gated secondary analysis |
| | sPGA (0,1)<br>sPGA (0) | Fisher's exact test<br>with NRI<br>Logistic regression<br>with NRI | ITT Population | Ixekizumab Q4W vs. placebo<br>at Week 12 and all other<br>postbaseline visits during<br>Period 2. | Other secondary analysis |
| | sPGA (0,1)<br>sPGA (0) | Summarize | Ixekizumab Efficacy<br>Primary Population | At all postbaseline visits during the Combined Treatment Periods (Periods 2, 3, and 4). | Other secondary analysis/<br>Exploratory analysis |
| | | | Ixekizumab Efficacy<br>Secondary Population | At all postbaseline visits<br>during the Combined<br>Treatment Periods (Periods 3<br>and 4) | Exploratory analysis |
| | Time to relapse to sPGA ≥2 | Log-rank test<br>Kaplan-Meier<br>estimate | Double-Blind,<br>Randomized<br>Withdrawal Period<br>Population | Ixekizumab Q4W vs. placebo<br>during the Double-Blind<br>Randomized Withdrawal<br>Period. | Other secondary analysis |
| BSA | Change from baseline | ANCOVA with<br>LOCF;<br>MMRM | ITT Population | Ixekizumab Q4W vs. placebo<br>at Week 12 and all other<br>postbaseline visits during<br>Period 2. | Other secondary analysis |

| Measure | Variable | Analysis<br>(Method) | Population | Comparison/Time Point | Analysis Type |
|---|---|---|---|---|---|
| NAPSI | Change from baseline | ANCOVA with<br>LOCF<br>MMRM | ITT Population – patients with baseline nail involvement (NAPSI baseline score >0) | Ixekizumab Q4W vs. placebo<br>at Week 12 and all other<br>postbaseline visits during<br>Period 2. | Other secondary analysis |
| | NAPSI score = 0 | Fisher exact test<br>with NRI<br>Logistic regression<br>with NRI | ITT Population – patients with baseline nail involvement (NAPSI baseline score >0) | Ixekizumab Q4W vs. placebo<br>at Week 12 and all other<br>postbaseline visits during<br>Period 2. | Exploratory analysis |
| PSSI | Change from baseline | ANCOVA with<br>LOCF;<br>MMRM | ITT Population – patients with baseline scalp involvement (PSSI baseline score >0) | Ixekizumab Q4W vs. placebo<br>at Week 12 and all other<br>postbaseline visits during<br>Period 2. | Other secondary analysis |
| | PSSI score = 0 | Fisher's exact test<br>with NRI<br>Logistic regression<br>with NRI | ITT Population – patients with baseline scalp involvement (PSSI baseline score >0) | Ixekizumab Q4W vs. placebo<br>at Week 12 and all other<br>postbaseline visits during<br>Period 2. | Exploratory analysis |
| PPASI | Change from baseline | ANCOVA with<br>LOCF;<br>MMRM | ITT Population – patients with baseline palmoplantar involvement (PPASI baseline score >0) | Ixekizumab Q4W vs. placebo<br>at Week 12 and all other<br>postbaseline visits during<br>Period 2. | Other secondary analysis |
| | PPASI 50<br>PPASI 75<br>PPASI 100 | Fisher's exact test<br>with NRI<br>Logistic regression<br>with NRI | ITT Population – patients with baseline palmoplantar involvement (PPASI baseline score >0) | Ixekizumab Q4W vs. placebo<br>at Week 12 and at each<br>postbaseline visit during<br>Period 2. | Exploratory analysis |
| Binary questions<br>on psoriasis<br>location | Proportion of patients with no psoriasis presence on face | Fisher's exact test<br>with NRI<br>Logistic regression<br>with NRI | ITT Population – patients with psoriasis presence on face at baseline | Ixekizumab Q4W vs. placebo at Week 12. | Other secondary analysis |

| Measure | Variable | Analysis<br>(Method) | Population | Comparison/Time Point | Analysis Type |
|---|---|---|---|---|---|
| | Proportion of patients with no psoriasis presence on nail | Fisher's exact test<br>with NRI<br>Logistic regression<br>with NRI | ITT Population – patients with psoriasis presence on nail at baseline | Ixekizumab Q4W vs. placebo at Week 12. | |
| | Proportion of patients with no psoriasis presence on axilla | Fisher's exact test<br>with NRI<br>Logistic regression<br>with NRI | ITT Population – patients with psoriasis presence on axilla at baseline | Ixekizumab Q4W vs. placebo at Week 12. | |
| | Proportion of patients with no psoriasis presence on genital | Fisher's exact test<br>with NRI<br>Logistic regression<br>with NRI | ITT Population – patients with psoriasis presence on genital at baseline | Ixekizumab Q4W vs. placebo at Week 12. | |
| | Proportion of patients<br>with no psoriasis<br>presence on perianal<br>region | Fisher's exact test<br>with NRI<br>Logistic regression<br>with NRI | ITT Population – patients with psoriasis presence on perianal region at baseline | Ixekizumab Q4W vs. placebo at Week 12. | |

Abbreviations: ANCOVA = analysis of covariance; BSA = body surface area; ITT = intent-to-treat; LOCF = last observation carried forward; MMRM = mixed-effects model of repeated measures; NAPSI = Nail Psoriasis Severity Index; NRI = nonresponder imputation; PASI = Psoriasis Area and Severity Index; PASI 50/75/90 = at least a 50%/75%/90% improvement from baseline in PASI score; PASI 100 = a 100% improvement from baseline in PASI score; PPASI = Palmoplantar Psoriasis Area and Severity Index; PPASI 50/75 = at least a 50%/75% improvement from baseline in PPASI score; P)PASI 100 = a 100% improvement from baseline in PPASI score; PSSI = Psoriasis Scalp Severity Index; Q4W = every 4 weeks; sPGA = static Physician Global Assessment; vs. = versus.

#### 6.11.1. Co-Primary Outcome and Primary Analysis Methodology

The co-primary outcomes are:

- Proportion of patients achieving PASI 75
- Proportion of patients achieving sPGA (0,1)

The primary analysis will be based on the ITT Population for the Double-Blind Treatment Period (Period 2) comparing ixekizumab versus placebo at Week 12. The primary analysis is Fisher's exact test. Missing data will be imputed using the NRI method. The secondary analyses for the primary efficacy measures will be conducted using a logistic regression with treatment group, region, baseline sPGA score (severity of the Ps), and baseline weight category (<25kg; ≥25 to ≤50 kg; or >50 kg) as factors. Missing data will be imputed using the NRI method.

#### 6.11.2. Gated Secondary Efficacy Analyses

The gated secondary outcomes are:

- Proportion of patients achieving PASI 90 at Week 12
- Proportion of patients achieving an sPGA (0) at Week 12
- Proportion of patients achieving PASI 100 at Week 12
- Proportion of subjects achieving ≥4-point improvement for subjects who had a baseline Itch NRS ≥4 at Week 12
- Proportion of patients achieving PASI 75 at Week 4
- Proportion of patients achieving sPGA (0,1) at Week 4

The gated secondary analyses will be based on ITT Population for the Double-Blind Treatment Period (Period 2) comparing ixekizumab versus placebo. The analysis will be Fisher's exact test. Missing data will be imputed using the NRI method.

# 6.11.3. Additional Analyses of the Co-Primary Outcome

There will be no adjustment for multiple comparisons for additional analyses of the co-primary outcomes.

To support the primary efficacy analysis, the co-primary outcomes, PASI 75 and sPGA (0,1), will be analyzed based on the PPS Population for the Double-Blind Treatment Period (Period 2), comparing ixekizumab versus placebo at Week 12 using Fisher's exact test with NRI.

# 6.11.4. Other Secondary Efficacy Analyses

There will be no adjustment for multiple comparisons for other secondary analyses.

The other secondary efficacy variables include:

• PASI 50, PASI 90, PASI 100, PASI change from baseline percent improvement

- sPGA (0)
- NAPSI change from baseline
- PSSI change from baseline
- PPASI change from baseline

The other secondary analyses for the Double-Blind Treatment Period (Period 2) will be based on the ITT Population, except (refer to Table RHCD.6.4):

- NAPSI: based on ITT Population patients with baseline nail involvement (NAPSI baseline score >0)
- PSSI: based on ITT Population patients with baseline scalp involvement (PSSI baseline score >0)
- PPASI: based on ITT Population patients with baseline palmoplantar involvement (PPASI baseline score >0)
- Binary questions on psoriasis locations

The other secondary analyses are detailed in Table RHCD.6.4. Comparisons of ixekizumab versus placebo at Week 12 and all other postbaseline visits will be provided.

Efficacy measures PASI 75, PASI 90, PASI 100, sPGA (0,1), and sPGA (0) at Week 24 and Week 48 will be summarized based on the ITT Population. The immunogenicity impact on efficacy is described in Section 6.14.11.2.2.

#### **Protocol Addendum I1F-MC-RHCD(2)**

The other secondary efficacy variables include:

- Period 2: ITT Population Etanercept-Approved Countries
  - o PASI50, PASI75, PASI90 and PASI100
  - o sPGA (0,1) and sPGA (0)
- Double-Blind Randomized Withdrawal Period (Period 4): Randomized Withdrawal Population
  - Time to relapse to moderate severity (sPGA ≥2) during the Double-Blind, Randomized Withdrawal Period
  - $\circ$  sPGA(0,1) and sPGA (0)
  - o PASI 50, PASI 75, PASI 90 and PASI 100

The other secondary analyses are detailed in Table RHCD.6.4. Analysis methods are detailed in Section 6.1.3.1.

#### 6.12. Health-Outcome/Quality-of-Life Analyses

The health-outcome and quality-of-life (QOL) measures are Itch NRS, CDLQI/DLQI, and Patient's global assessment of disease severity. Table RHCD.6.5 and Table RHCD.6.6 include the description and derivation of the health-outcome and QOL measures. There will be no adjustment for multiple comparisons.

The analyses of health-outcome variables for Period 2 will be based on the ITT Population, except:

• Itch NRS ≥4 improvement from baseline: based on ITT Population - patients with baseline Itch NRS score ≥4

Table RHCD.6.6 provides the detailed analyses including analysis type, method and imputation, population, time point, and dosing regimen comparisons for health-outcome and QOL analyses.

 Table RHCD.6.5.
 Description and Derivation of Health-Outcome and Quality-of-Life Measures

| Measure | Description | Variable | Derivation / Comment | Imputation Approach if with Missing Components |
|---|---|---|---|---|
| Itch NRS | Itch Numeric Rating Scale (NRS): is a single-<br>item, patient-reported outcome (PRO) measure<br>designed to capture information on the overall | Itch NRS score | Range from 0 to 10. | Single item, missing if missing |
| | severity of a patient's itching due to his/her psoriatic skin condition by having the patient | Itch NRS change from baseline | Calculated as: observed Itch NRS – baseline Itch NRS | Missing if baseline or observed value is missing |
| | circle the integer that best describes the worst<br>level of itching in the past 24 hours on an<br>11-point NRS anchored at 0 representing "no<br>itching" and 10 representing "worst itch | Itch NRS ≥4 improvement from baseline | Reduced/decreased of ≥4 point from baseline | Missing if baseline or observed value is missing |
| | imaginable." | Itch NRS = 0 | Defined as a postbaseline Itch NRS score of 0 | Missing if Itch NRS score is missing |
| DLQI | Dermatology Life Quality Index (DLQI): is a validated, dermatology-specific, patient-reported measure that evaluates patient's health-related quality of life. This questionnaire has 10 items that are grouped in | DLQI symptoms<br>and feelings<br>domain | Sum of responses of questions #1 and #2:<br>#1. How itchy, sore, painful or stinging<br>has your skin been?<br>#2. How embarrassed or self-conscious<br>have you been because of your skin? | If one question in a domain is missing, that domain is missing. |
| | 6 domains, including symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. The recall period of this scale is over the "last week." Response categories and corresponding scores are: | DLQI daily<br>activities domain | Sum of responses of questions #3 and #4:<br>#3. How much has your skin interfered<br>with you going shopping or looking after<br>your home or garden?<br>#4. How much has your skin influenced<br>the clothes you wear? | If one question in a domain is missing, that domain is missing. |
| | Very much = 3 A lot = 2 A little = 1 Not at all = 0 Not relevant = 0 | DLQI leisure<br>domain | Sum of responses of questions #5 and #6:<br>#5. How much has your skin affected any<br>social or leisure activities?<br>#6. How much has your skin make it<br>difficult for you to do any sport? | If one question in a domain is missing, that domain is missing. |
| | | DLQI work and school domain | Sum of responses of questions question #7A and #7B: #7A. Has your skin prevented you from working or studying? #7B. If No: how much has your skin been | If the answer to question #7A is missing, this domain is missing. If #7A is No, and #7B is missing, this domain is missing. |

| Measure | Description | Variable | Derivation / Comment | Imputation Approach if with Missing Components |
|---|---|---|---|---|
| | • | | a problem at work or studying? | g 1 |
| | | DLQI personal<br>and relationships<br>domain | Sum of responses of questions #8 and #9: #8. How much has your skin created problems with your partner or any of your close friends or relatives? #9. How much has your skin caused any sexual difficulties? | If 1 question in a domain is missing, that domain is missing. |
| | | DLQI treatment | Response of question #10:<br>#10. How much of a problem has the<br>treatment for your skin been, for example<br>by making your home messy, or by<br>taking up time? | If 1 question in a domain is missing, that domain is missing. |
| | | DLQI total score | A DLQI total score is calculated by summing all 10 question responses, and has a range of 0 to 30 (less to more impairment) (Finlay and Khan 1994; Basra et al. 2008). | If 2 or more questions are missing, the total score is missing. Note: #7B could be a valid missing while #7A is not "No." That is, #7 should be considered as 1 question. |
| | | DLQI (0,1) | A DLQI (0,1) response is defined as a postbaseline DLQI total score of 0 or 1. A DLQI total score of 0 to 1 is considered as having no effect on a patient's health-related quality of life (HRQoL) (Khilji et al. 2002; Hongbo et al. 2005). | Missing if DLQI total score is missing |
| CDLQI | Children's Dermatology Life Quality Index (CDLQI): is designed for use in children (subjects form age 4 to age 16 years) (Lewis-Jones and Finlay 1995; Waters et al. 2010; Salek et al. 2013). It consists of 10 items, of | CDLQI symptoms<br>and feelings<br>domain | Sum of responses of questions #1 and #2:<br>#1. How itchy, "scratchy," sore, or<br>painful has your skin been?<br>#2. How embarrassed or self-conscious,<br>have you been because of your skin? | If 1 question in a domain is missing, that domain is missing. |
| | which there are 6 headings, including<br>symptoms and feelings, leisure, school or<br>holidays, personal relationships, sleep, and<br>treatment. The recall period of this scale is | CDLQI leisure | Sum of responses of questions #4, #5, and #6:<br>#4. How much have you changed or worn different or special clothes/shoes because | If 1 question in a domain is missing, that domain is missing. |

| Measure | Description | Variable | Derivation / Comment | Imputation Approach if with Missing Components |
|---|---|---|---|---|
| | over the "last week." Response categories and | | of your skin? | 9 |
| | corresponding scores are: | | #5. How much has your skin trouble | |
| | 0-1 = no effect on child's life | | affected going out, playing, or doing | |
| | 2-6 = small effect | | hobbies? | |
| | 7-12 = moderate effect | | #6. How much have you avoided | |
| | 13-18 = very large effect | | swimming or other sports because of your | |
| | 19-30 = extremely large effect | | skin trouble? | |
| | 3 6 | CDLQI school or | Response of question | If 1 question in a domain is |
| | | holidays | #7A or #7B: | missing, that domain is |
| | | | #7A. If school time, how much did your | missing. If both parts of |
| | | | skin problem affect your school work? | Question 7 are answered, the |
| | | | #7B. If holiday time, how much has your | higher of the 2 scores should |
| | | | skin problem interfered with your | be counted. |
| | | | enjoyment of the holiday? | |
| | | CDLQI personal | Sum of responses of questions #3 and #8: | If 1 question in a domain is |
| | | relationships | #3. How much has your skin affected | missing, that domain is |
| | | _ | your friendships? | missing. |
| | | | #8. How much trouble have you had | |
| | | | because of your skin with other people | |
| | | | calling you names, teasing, bullying, | |
| | | | asking questions, or avoiding you? | |
| | | CDLQI sleep | Response of question #9: | If 1 question in a domain is |
| | | | #9. How much has your sleep been | missing, that domain is |
| | | | affected by your skin problem? | missing. |
| | | CDLQI treatment | Response of question #10: | If 1 question in a domain is |
| | | | #10. How much of a problem has the | missing, that domain is |
| | | | treatment for your skin been? | missing. |
| | | CDLQI total score | A CDLQI total score is calculated by | If 2 or more questions are |
| | | | summing all 10 question responses, and | missing, the total score is |
| | | | has a range of 0 to 30 (less to more | missing. |
| | | | impairment) (Lewis-Jones and Finlay | |
| | | | 1995; Basra et al. 2008). | |

| Measure | Description | Variable | Derivation / Comment | Imputation Approach if with Missing Components |
|---|---|---|---|---|
| | | CDLQI (0,1) | A CDLQI (0,1) response is defined as a postbaseline CDLQI total score of 0 or 1. | Missing if CDLQI total score is missing |
| Patient's<br>Global | Patient's Global Assessment of Disease<br>Severity (PatGA): is a subject-administered | PatGA (0,1) | A PatGA (0,1) response is defined as a postbaseline PatGA score of 0 or 1. | Missing if the item is missing |
| Assessment<br>of Disease<br>Severity | single-item scale on which subjects are asked to rank by circling a number on a 0 to 5 numerical rating scale (NRS) the severity of their psoriasis today from 0 (clear) = no psoriasis to 5 (severe) = the worst their psoriasis has ever been. | Change from baseline | Calculated as: observed PatGA – baseline PatGA | Missing if baseline or observed value is missing |

Table RHCD.6.6. Description of Health-Outcomes and Quality-of-Life Analyses

| Measure | Variable | Analysis (Method) | Population | Comparison/Time Point |
|---|---|---|---|---|
| Itch NRS | Itch NRS ≥4 improvement from | Fisher's exact test with NRI | ITT Population – | Ixekizumab Q4W vs. placebo at Week 12 and |
| | baseline | Logistic regression with NRI | patients with | all other postbaseline visits during Period 2 |
| | (Gated secondary) | | baseline value ≥4 | |
| | Change from baseline | MMRM | ITT Population | Ixekizumab Q4W vs. placebo at Week 12 and |
| | | | | all other postbaseline visits during Period 2 |
| | | ANCOVA with LOCF | ITT Population | Ixekizumab Q4W vs. placebo at Week 12 and |
| | | | | all other postbaseline visits during Period 2 |
| CDLQI/DLQI | CDLQI/DLQI (0,1) | Fisher's exact test with NRI | ITT Population | Ixekizumab Q4W vs. placebo at Week 12 and |
| | | Logistic regression with NRI | | all other postbaseline visits during Period 2 |
| PatGA | PatGA (0,1) | Fisher's exact test with NRI | ITT Population | Ixekizumab Q4W vs. placebo at Week 12 and |
| | | Logistic regression with NRI | | all other postbaseline visits during Period 2 |
| | Change from baseline | ANCOVA with LOCF | ITT Population | Ixekizumab Q4W vs. placebo at Week 12 and |
| | | | | all other postbaseline visits during Period 2 |

Abbreviations: ANCOVA = analysis of covariance; CDLQI = Children's Dermatology Life Quality Index; DLQI = Dermatology Life Quality Index; ITT = intent-to-treat; LOCF = last observation carried forward; MMRM = mixed-effects model of repeated measures; NRI = nonresponder imputation; NRS = Numeric Rating Scale; PatGA = Patient's Global Assessment of Disease Severity; Q4W = every 4 weeks; vs. = versus.

#### 6.13. Pharmacokinetic/Pharmacodynamic Methods

More details of the pharmacokinetic/pharmacodynamic (PK/PD) analyses can be found in a separate PK/PD analysis plan.

Briefly, observed ixekizumab serum trough concentrations will be summarized by time point across the study. The PK parameters of ixekizumab in pediatric subjects will be determined using population PK methods. The exposure-response relationship will be investigated between steady-state trough concentrations of ixekizumab and clinically important efficacy measures (for example, sPGA and PASI endpoints) at Week 12 using graphical methods and, if appropriate, modeling methods. If applicable, the potential impact of immunogenicity on ixekizumab exposure and/or exposure or efficacy responses may be evaluated by graphical assessments, as appropriate, to compare drug exposure or efficacy responses between antidrug antibody- (ADA-) negative and ADA-positive subjects at corresponding visits, or before and after ADA development for subjects who developed ADA. Both treatment-emergent only and all ADA-positive/negative subjects may be explored. A similar approach may be taken if subjects become neutralizing antibody positive.

Additional analyses may be performed upon receipt of the data. The data from this study may be combined with data from previous adult studies, if needed, for model development.

#### 6.14. Safety Analyses

Safety will be assessed by summarizing and analyzing AEs, laboratory analytes, including neutrophil counts and immunogenicity; vital signs, CDRS, and C-SSRS. The duration of dosing exposure will also be summarized. Immunization history will be summarized at baseline, and any unexpected outcomes or effects related to standard-of-care vaccination will be summarized.

For Period 2 in Main Protocol RHCD, the safety data will be summarized and analyzed for the safety population with treatment comparisons of ixekizumab versus placebo. This population will be abbreviated as "P2 Main Study Safety Population."

For Period 2 in Protocol Addendum RHCD(2), the select safety data will be summarized and analyzed for the safety population etanercept-approved countries with all pairwise comparisons. This population will be abbreviated as "P2 Addendum Safety Population."

For Period 4 in Protocol Addendum RHCD(2), the select safety data will be summarized and analyzed for the Double-Blind, Randomized Withdrawal Period Population with treatment comparisons of ixekizumab versus placebo. This population will be abbreviated as "P4 Randomized Withdrawal Population."

For all ixekizumab treatment periods combined (Period 2, 3, and 4), the safety data will be summarized to all ixekizumab population. This population will be abbreviated as "All Ixekizumab Safety Population."

For Period 5, safety data will be summarized using Follow-Up Population.

#### 6.14.1. Extent of Exposure

Duration of exposure to study drug will be summarized by treatment group using descriptive statistics, the summary will also include the total exposure in patient years, mean, and median total dose. Exposure of the following safety population will be summarized:

- P2 Main Study Safety Population
- P2 Addendum Safety Population
- P4 Randomized Withdrawal Population
- All Ixekizumab Safety Population

The duration of exposure will be calculated as:

- Duration of exposure (days) =
   Date of last visit (scheduled or unscheduled) in the treatment period Date of first dose in the treatment period + 1
- Total exposure in patient years will be calculated as:

```
Total exposure in patient years
= \frac{Sum \ of \ duration \ (days) \ of \ exposures \ for \ all \ patients \ in \ treatment \ group}{365.25}
```

• Total dose (in mg) is calculated by the summation of dose for each active injection taken during the treatment period. Dose for placebo injection will be 0.

For P2 Main Study and P2 Addendum Safety Populations, the number and percentage of patients in each of the following categories will be included in the summaries:

- $>0, \ge 7$  days,  $\ge 14$  days,  $\ge 30$  days,  $\ge 60$  days,  $\ge 84$  days, and  $\ge 90$  days. Note that patients may be included in more than 1 category.
- >0 to <7 days, ≥7 to <14 days, ≥14 to <30 days, ≥30 to <60 days, ≥60 to <84 days, ≥84 to <90 days, and ≥90 days.

For P4 Randomized Withdrawal Population, the number and percentage of patients in each of the following categories will be included in the summaries:

- $>0, \ge 7$  days,  $\ge 14$  days,  $\ge 30$  days,  $\ge 60$  days,  $\ge 84$  days,  $\ge 90$  days,  $\ge 120$  days,  $\ge 183$  days, and  $\ge 365$  days. Note that patients may be included in more than 1 category.
- >0 to <7 days, ≥7 to <14 days, ≥14 to <30 days, ≥30 to <60 days, ≥60 to <84 days, ≥84 to <90 days, ≥90 to <120 days, ≥120 to <183 days, ≥183 to <365 days, and ≥365 days

For the All Ixekizumab Safety Population, duration of exposure for each uninterrupted ixekizumab treatment period will be calculated as:

*Duration of ixekizumab exposure (days)* 

- = Date of last visit of ixekizumab treatment period
- Date of first dose of ixekizumab treatment period +1

If a patient had more than 1 uninterrupted ixekizumab treatment periods, patients who re-randomized to placebo during the Double-Blind, Randomized Withdrawal Period (Period 4) and relapsed, the duration of total ixekizumab exposure is the sum of durations of both uninterrupted ixekizumab exposure.

The number and percentage of patients in each of the following categories will be included in the summaries for the All Ixekizumab Safety Population:

- >0, ≥7 days, ≥14 days, ≥30 days, ≥60 days, ≥84 days, ≥90 days, ≥120 days, ≥183 days, ≥365 days, ≥548 days, and ≥730 days. Note that patients may be included in more than 1 category.
- >0 to <7 days, ≥7 to <14 days, ≥14 to <30 days, ≥30 to <60 days, ≥60 to <84 days, ≥84 to <90 days, ≥90 to <120 days, ≥120 to <183 days, ≥183 to <365 days, ≥365 days to <548 days, ≥548 days to <730 days, and ≥730 days.

#### 6.14.2. Adverse Events

Adverse events will be classified based upon the latest version of the MedDRA. Adverse events will be recorded at every study visit. Any condition starting on or after the date of informed consent will be considered an AE. Any preexisting condition which worsens in severity on or after the date of informed consent will be considered and recorded as an AE on the Adverse Event (AE) eCRF page from the date of worsening onward.

A treatment-emergent adverse event (TEAE) is defined as an event that first occurred or worsened in severity after baseline and on or prior to the date of the last visit within the defined treatment period. Both the date/time of the event and the date/time of the dose (that is, injection) are considered when determining TEAEs. Treatment-emergent AEs will be assigned to the study period to which it is considered treatment-emergent:

- The MedDRA lowest level term (LLT) will be used when classifying AEs as treatmentemergent.
- The maximum severity recorded for each LLT prior to the first dose date/time in the treatment period will be used as the pre-treatment severity for that LLT. If an event during the baseline period has missing severity, and the event persists during the treatment period, then it will be considered as treatment-emergent, regardless of the postbaseline level of severity. Events with a missing severity during the treatment period will be considered treatment-emergent.
- AEs with a particular LLT will be classified as treatment-emergent if they first start on or after the first dose date/time in the treatment period (that is, a patient has no preexisting conditions with that LLT), or if the severity is greater than the pre-treatment severity for that LLT. If a partial AE start date/time is present, the date/time will be compared as far as possible to the treatment start date/time in order to determine whether the event is treatment-emergent. If there is any doubt, the event will be flagged as treatment-emergent.

A follow-up-emergent adverse event (FEAE) is defined as an event that first occurred or worsened in severity after the date of Visit 31 (that is, Week 108) or the ETV:

- The MedDRA LLT will be used when classifying AEs as follow-up-emergent.
- For AEs that are ongoing at the date of Visit 31 or ETV, the maximum severity recorded for each LLT on or prior to the date of Visit 31 or ETV will be used as the follow-up baseline severity for that LLT.

If a partial or completely missing AE start date/time or end date/time is present the following imputation rules will be utilized in the analysis:

- For the start date:
  - o If year, month, and day are missing, then use the earlier of the patient's first visit date or the consent date.
  - o If either month or month and day are missing, then use January 1.
  - o If only day is missing, impute the first day of the month.
- For the start time:
  - o Impute as 23:59
- For the end date:
  - o If year, month, and day are missing, then use the patient's last visit date in the follow-up period.
  - o If either month or month and day are missing, then use December 31.
  - o If only day is missing, then use the last day of the month.
  - The imputed date will not be beyond the patient's last visit date in the follow-up period.
- For the end time:
  - o Impute as 23:59.
- If there is any doubt, the event will be flagged as treatment-emergent or follow-up-emergent, according the corresponding study period. If a follow-up-emergent event was already counted as treatment-emergent during the prior treatment period, it will not be counted as a follow-up-emergent event.

Adverse events and TEAEs will be summarized for the following study periods and analysis populations; treatment comparisons between treatment groups will be conducted using a Fisher's exact test.

The following summaries/analyses will be performed for P2 Main Study Safety Population and All Ixekizumab Safety Population:

- An overall summary of AEs, including the number and percentage of patients who experienced TEAE, TEAE by maximum severity, death, serious adverse event (SAE), TEAE possibly related to study treatment, discontinuations from the treatment due to an AE, and TEAEs of special interest.
- TEAE by SOC and PT.
- TEAE by maximum severity, SOC, and PT.

The following summaries/analyses will be performed for P2 Addendum Safety Population and P4 Randomized Withdrawal Population:

- An overall summary of AEs, including the number and percentage of patients who
  experienced TEAE, TEAE by maximum severity, death, SAE, TEAE possibly related to
  study treatment, discontinuations from the treatment due to an AE, and TEAEs of special
  interest.
- TEAE by SOC and PT.

Follow-up emergent adverse events will be summarized for the Follow-Up Population for Period 5:

• FEAE by SOC and PT.

In general, for all AE-related summaries, the number and percentage of patients experiencing the events will be presented by treatment group. In general, events will be ordered by decreasing frequency in the total ixekizumab group, followed in the order of ixekizumab Q4W, etanercept, and placebo (when applicable) group, within SOC and/or PT for sorting. For events that are gender-specific (as defined by MedDRA), the denominator and computation of the percentage will include only patients from the given gender.

A by-patient listing of all AEs will be provided.

# 6.14.3. Deaths, Other Serious Adverse Events, and Other Notable Adverse Events

By-patient listings of deaths, SAEs, and AEs leading to discontinuation will be provided, respectively.

All deaths will be included, regardless of the investigator's or the Sponsor's judgment about causality, including:

- any deaths occurring during participation in the study in the database for which data are being presented
- any deaths occurring after a patient leaves (is discontinued from or completed) the study in the database for which data are being presented if the death is:
  - o the result of a process initiated during the study, regardless of when it actually occurred
  - o occurs during the Period 5 after discontinuation of study drug

An SAE is any AE that results in one of the following outcomes: death, life-threatening, initial or prolonged hospitalization, disability or permanent damage, congenital anomaly or birth defect, or any other serious/important medical events.

The following summary tables (including treatment group comparison for Period 2) will be provided for P2 Main Study Safety Population and All Ixekizumab Safety Population:

- SAEs by SOC and PT
- AEs that lead to treatment discontinuation (including death) by SOC and PT

The following summary tables (including treatment group comparisons for Period 2 and Period 4) will be provided P2 Addendum Safety Population and P4 Randomized Withdrawal Population:

• SAEs by SOC and PT

# **6.14.3.1.** Special Safety Topics including Adverse Events of Special Interest Safety information on special topics including AEs of special interest (AESIs) will be presented by treatment group for P2 Main Study Safety Population and All Ixekizumab Safety Population.

Table RHCD.6.7 provides the definitions/derivations and analyses methods (including analyses, summaries and by-patient listings) of special safety topics including AESIs.

Potential AESIs will be identified by a standardized MedDRA query (SMQ) or a Lilly-defined MedDRA PT listing. Preferred terms within an SMQ will be classified as broad and narrow. In the Lilly-defined MedDRA PT listings, Lilly has provided the broad and narrow classification. The Lilly-defined broad terms are for a more sensitive search of potential events of interest, and the Lilly-defined narrow terms are for a more specific search. Therefore, the summaries will include the classifications of broad term (same as pooling narrow and broad terms together) and narrow term.

In the event that the listing of terms or analysis changes for a special safety topic, it will be documented in the most current program safety analysis plan (PSAP) which will supersede this document; it will not warrant an amendment to the individual study SAP.

Fisher's exact tests will be used to compare the treatment groups.

In general, AESI summary will not be provided for Follow-Up Population during Period 5 except for cytopenia and hepatic laboratory tests.

Table RHCD.6.7. Definitions and Analyses of Special Safety Topics including Adverse Events of Special Interest

| Special Safety<br>Topic | Definition/Derivation | Analysis/Summary/Listing |
|---|---|---|
| Hepatic | Hepatic AE analysis will include events that are potentially drug-related hepatic disorders by using the MedDRA PTs contained in any of the following SMQs: • Broad and narrow terms in the Liver related investigations, signs and symptoms (20000008) • Broad and narrow terms in the Cholestasis and jaundice of hepatic origin (20000009) • Broad and narrow terms in the Hepatitis, non-infectious (20000010) • Broad and narrow terms in the Hepatic failure, fibrosis and cirrhosis and other liver damage (20000013) • Narrow terms in the Liver-related coagulation and bleeding disturbances (20000015) | P2 Main Study Safety Population (Fisher's exact test) and All Ixekizumab Safety Population (Summary): TEAE by PT within SMQ or sub-SMQ Listing: TEAE (display in Spotfire) |
| | <ul> <li>Elevations in hepatic laboratory tests (ALT, AST, ALP, total bilirubin) using Performing Laboratory Reference Ranges are defined as:</li> <li>Include scheduled visits, unscheduled visits, and repeat measurements.</li> <li>ALT or AST: maximum postbaseline measurement ≥3 times (3×), 5 times (5×), 10 times (10×), and 20 times (20×) the Performing Lab ULN for all patients with a postbaseline value.</li> <li>The analysis of 3× ULN will contain 4 subsets: patients whose nonmissing maximum baseline value is ≤1× ULN, patients whose maximum baseline is &gt;1× ULN but &lt;3× ULN, patients whose maximum baseline value is ≥3× ULN, and patients whose baseline values are missing.</li> <li>The analysis of 5× ULN will contain 5 subsets: patients whose nonmissing maximum baseline value is ≤ to 1× ULN, patients whose maximum baseline is &gt;1× ULN but &lt;3× ULN, patients whose maximum baseline value is ≥5× ULN, and patients whose baseline values are missing.</li> <li>The analysis of 10× ULN will contain 6 subsets: patients whose nonmissing maximum baseline value is ≤1× ULN, patients whose maximum baseline is &gt;1× ULN but &lt;3× ULN, patients whose maximum baseline is ≥5× ULN but &lt;10× ULN, patients whose maximum baseline value is ≥10× ULN, and patients whose baseline value is ≤1× ULN, patients whose maximum baseline value is ≤1× ULN, patients whose maximum baseline is &gt;1× ULN but &lt;3× ULN, patients whose maximum baseline value is ≥10× ULN but &lt;3× ULN, patients whose maximum baseline is ≥3× ULN but &lt;5× ULN, patients whose maximum baseline is ≥5× ULN but &lt;10× ULN, patients whose maximum baseline is ≥10× ULN but &lt;20× ULN, patients whose maximum baseline value is ≥5× ULN but &lt;10× ULN, patients whose maximum baseline is ≥10× ULN but &lt;20× ULN, patients whose maximum baseline value is ≥10× ULN but &lt;20× ULN, patients whose maximum baseline value is ≥10× ULN but &lt;10× ULN, patients whose maximum baseline value is ≥10× ULN but &lt;10× ULN, patients whose maximum baseline value is ≥10× ULN but &lt;10× ULN, patients whose maximum baseline value is ≥10× U</li></ul> | Listing: Elevations in hepatic laboratory tests (display in Spotfire) |

| Special Safety | | |
|---|---|---|
| Topic | Definition/Derivation | Analysis/Summary/Listing |
| | $\geq$ 2×) the Performing Lab ULN during the treatment period will be summarized for all patients with a | |
| | postbaseline value. | |
| | o The analysis of 1.5× ULN will contain 4 subsets: patients whose nonmissing maximum baseline | |
| | value is $\leq 1 \times$ ULN, patients whose maximum baseline is $\geq 1 \times$ ULN but $\leq 1.5 \times$ ULN, patients whose | |
| | maximum baseline value is $\ge 1.5 \times$ ULN, and patients whose baseline values are missing. | |
| | o The analysis of 2× ULN will contain 5 subsets: patients whose nonmissing maximum baseline | |
| | value is $\leq 1 \times$ ULN, patients whose maximum baseline is $\geq 1 \times$ ULN but $\leq 1.5 \times$ ULN, patients whose | |
| | maximum baseline is $\ge 1.5 \times$ ULN but $\le 2 \times$ ULN, patients whose maximum baseline value is $\ge 2 \times$ | |
| | ULN, and patients whose baseline values are missing. | |
| | • ALP: The number and percentages of patients with an ALP measurement >1.5× the Performing Lab | |
| | ULN during the treatment period will be summarized for all patients with a postbaseline value, and | |
| | divided into 4 subsets: patients whose nonmissing maximum baseline value is ≤1× ULN, patients whose | |
| | maximum baseline is >1× ULN but ≤1.5× ULN, patients whose maximum baseline value is >1.5× ULN, | |
| | and patients whose baseline values are missing. | |
| | • The number and percentages of patients meeting the following elevated hepatic criteria: maximum ALT | |
| | $\geq$ 3× ULN and maximum total bilirubin $\geq$ 2× ULN during the treatment period will be summarized. | |
| | Shift for ALT, AST, and total bilirubin from maximum baseline to maximum postbaseline will be produced | |
| | with the requirements using Performing Lab Reference Ranges: | |
| | Include scheduled visits, unscheduled visits, and repeat measurements. | |
| | Use the maximum nonmissing value in the baseline period. | |
| | Use the maximum nonmissing postbaseline value within each study period. | |
| | Categories are: | |
| | $\circ \text{ALT: } \leq 1 \times \text{ULN}, > 1 \text{ to } < 3 \times \text{ULN}, \geq 3 \text{ to } < 5 \times \text{ULN}, \geq 5 \text{ to } < 10 \times \text{ULN}, \geq 10 \text{ to } < 20 \times \text{ULN}, \text{ and } \geq 20 \times 10 \times 10^{-5} \text{ to } < 10^{-5} \text{ to } <$ | |
| | ULN | |
| | $\circ AST: \ \le 1 \times \ ULN, \ >1 \ to \ <3 \times \ ULN, \ \ge 3 \ to \ <5 \times \ ULN, \ \ge 5 \ to \ <10 \times \ ULN, \ \ge 10 \times \ to \ <20 \times \ ULN \ and \ \ge 20 \times \ ULN \ and \ \ge 10 \times \ ULN \ and \ B$ and \ B\ B | |
| | ULN | |
| | ○ Total bilirubin: $\leq 1 \times ULN$ , $\geq 1$ to $\leq 1.5 \times ULN$ , $\geq 1.5$ to $\leq 2 \times ULN$ , $\geq 2 \times ULN$ | |
| | $\circ \text{ALP:} \le 1 \times \text{ULN,} > 1 \text{ to } \le 1.5 \times \text{ULN,} > 1.5 \times \text{ULN}$ | |
| | With additional categories: | |
| | <ul> <li>Decreased: postbaseline category &lt; baseline category</li> </ul> | |
| | <ul> <li>Increased: postbaseline category &gt; baseline category</li> </ul> | |
| | o Same: postbaseline category = baseline category | |
| | Elevated hepatic criteria: maximum ALT $\ge 3 \times$ ULN, maximum total bilirubin $\ge 2 \times$ ULN. | |

| Special Safety | | |
|---|---|---|
| Topic | <b>Definition/Derivation</b> | Analysis/Summary/Listing |
| | Listing of patients who meet any of the following criteria: | |
| | • Elevated hepatic criteria: defined as maximum ALT ≥3× ULN, maximum total bilirubin ≥2× ULN | |
| | An ALT or AST ≥3× ULN | |
| | • An ALP $\geq 1.5 \times$ ULN | |
| | A total bilirubin ≥2× ULN | |
| | The listing will include: patient demographics, concomitant medications, ALT/AST/ALP/total | |
| | bilirubin/GGT by visit, treatment start and stop dates, and reason for treatment discontinuation | |
| | Evaluation of Drug-Induced Serious Hepatotoxicity (eDISH) plot: use maximum ALT measurement and | P2 Main Study Safety |
| | maximum total bilirubin measurement with patients having at least 1 postbaseline ALT and total bilirubin, | Population and All |
| | which contributes 1 point to the plot. The measurements do not need to be taken at the same blood draw. | Ixekizumab Safety Population: eDISH plot (display in |
| | | Spotfire) |
| Cytopenias | Cytopenias are defined using the PTs from the following 2 sub-SMQs of the Haematopoietic cytopenias | P2 Main Study Safety |
| - | SMQ (20000027) as defined in MedDRA version: | Population (Fisher's exact |
| | Broad and narrow terms in the Haematopoietic leukopenia (20000030) | test) and All Ixekizumab |
| | Broad and narrow terms in the Haematopoietic thrombocytopenia (20000031) | Safety Population |
| | | (Summary): |
| | | TEAE by PT within sub-SMQ |
| | | Period 5 (Summary): |
| | | FEAE by PT within sub-SMQ |
| | | Listing: |
| | | TEAE (display in Spotfire) |
| Infections | Infections are events including all infections (defined using all the MedDRA PTs from the Infections and | P2 Main Study Safety |
| | infestations SOC), serious infections, potential opportunistic infections, and infections resulting in anti- | Population (Fisher's exact |
| | infective medication administration (i.e., antibacterial, antiviral, antifungals, antiparasitic treatment.). | test) and All Ixekizumab |
| | The relationship between TEAEs-infections and other clinical, laboratory, and hematology parameters will | Safety Population |
| | be examined using Spotfire tool. | (Summary): |
| | | TEAE by PT* |
| | | SAE by PT* |
| | | DCAE by PT* |
| | | * Included in overall TEAE |
| | | tables. |

| Special Safety<br>Topic | Definition/Derivation | Analysis/Summary/Listing |
|---|---|---|
| | | Listing: TEAE (display in Spotfire) |
| | Anti-infective medications are defined in Appendix 2 including antibiotics, antifungals, antivirals, or antiprotozoals. | |
| | The opportunistic infections (OI) are defined in Appendix 3. This list contain PTs as contained within Categories (narrow or broad) from the Infections and Infestations SOC and from the Investigations SOC which can assist in identifying potential OIs. The narrow terms are considered opportunistic infections unless medical review determines that the reported term is not consistent with the patient's clinical history/presentation/course. Medical review of broad terms is needed for final determination of patients meeting the program definition of OIs. The number and percentage of patients with TEAEs that represent potential OIs and as potential OIs will be summarized by treatment group using MedDRA PT nested within categories. Events will be ordered by decreasing frequency in the ixekizumab group (or combined ixekizumab group in the event of multiple cohorts/doses) nested within categories. | P2 Main Study Safety Population (Fisher's exact test) and All Ixekizumab Safety Population (Summary): TEAE of OIs Listing: TEAE of OIs (display in Spotfire) |
| | The duration of each common TEAE PT of Infections and narrow terms for Opportunistic infections is defined as: Duration of treatment-emergent AE Infections (in weeks) = (End date of AE – Start date of AE + 1) / 7. Patients who do not have the PT will not be included in the analysis. If the TEAE has not ended by the date of completion from the study, or date of early discontinuation, it will be censored as of that date. If a patient has multiple episodes of the same TEAE, the episode with the greatest severity will be used for the duration of event calculation. If a patient has multiple episodes of the same TEAE with the same severity, the episode with the longest duration will be used for the duration of event calculation. | P2 Main Study Safety Population and All Ixekizumab Safety Population (Summary): Duration of Common TEAE – Infections (display in Spotfire) |
| Allergic<br>Reactions/<br>Hypersensitiv-<br>ities | Allergic reactions/hypersensitivity events will be categorized as either anaphylaxis or nonanaphylaxis events (these will refer to events that are not localized to the site of injection) and summarized separately. Allergic Reactions/Hypersensitivity Events, Anaphylaxis: Anaphylaxis has been broadly defined as "a serious allergic reaction that is rapid in onset and may cause death" (Sampson et al. 2006). Identification of cases of potential anaphylaxis from the clinical trial data involves 2 screening criteria: | P2 Main Study Safety Population (Fisher's exact test) and All Ixekizumab Safety Population (Summary): |

| Special Safety | | |
|---|---|---|
| Topic | Definition/Derivation | Analysis/Summary/Listing |
| | 1) Designed to specifically identify cases (following Criterion 1) based on narrow terms from the MedDRA | TEAE by PT within Category, |
| | SMQ for anaphylactic reaction (20000021). Criterion 1 for anaphylaxis is defined by the presence of a | SAE by PT within Category, |
| | TEAE based on the following MedDRA PTs from the anaphylactic reaction SMQ: | AE leading to treatment |
| | Anaphylactic reaction | discontinuation by PT within |
| | Anaphylactic shock | Category. |
| | Anaphylactoid reaction | |
| | Anaphylactoid shock | Listing: |
| | Kounis Syndrome | TEAE (display in Spotfire) |
| | Type 1 hypersensitivity | |
| | 2) To identify possible cases, following Criterion 2 as defined by Sampson et al. (2006). Criterion 2 for | |
| | anaphylaxis requires having TEAEs from 2 or more of 4 categories of AEs as described by Sampson et | |
| | al. (2006). Occurrence of these events should be nearly coincident; based on recording of events or | |
| | CRFs. All qualifying events must be within 1 day of study drug injection. | |
| | The 4 categories to be considered in Criterion 2 are: | |
| | Category A: Involvement of the skin-mucosal tissue | |
| | Category B: Respiratory compromise | |
| | Category C: Reduced blood pressure or associated symptoms | |
| | Category D: Persistent gastrointestinal symptoms | |
| | The specific MedDRA PTs covered by each of these Criterion 2 categories are shown in Appendix 4. | |
| | Summaries of Criterion 2 anaphylactic TEAEs will be provided by the specific combination of categories as | |
| | follows: | |
| | AB: events based on meeting Category A and Category B (but no other category) | |
| | AC: events based on meeting Category A and Category C (but no other category) | |
| | AD: events based on meeting Category A and Category D (but no other category) | |
| | BC: events based on meeting Category B and Category C (but no other category) | |
| | BD: events based on meeting Category B and Category D (but no other category) | |
| | CD: events based on meeting Category C and Category D (but no other category) | |
| | ABC: events based on meeting Category A, Category B and Category C (but no other category) | |
| | ABD: events based on meeting Category A, Category B and Category D (but no other category) | |
| | ACD: events based on meeting Category A, Category C and Category D (but no other category) | |
| | BCD: events based on meeting Category B, Category C and Category D (but no other category) | |
| | ABCD: events based on meeting each of the 4 Criterion 2 categories. | |
| | Summaries of treatment-emergent anaphylactic AEs will be provided for patients meeting each of the | |
| | 2 criteria and for patients who meet either criteria, overall. Separate summaries will be provided for TEAEs | |

| Special Safety | | |
|---|---|---|
| Topic | Definition/Derivation | Analysis/Summary/Listing |
| | by maximum severity, SAEs, and AEs resulting in study drug discontinuation. Severity of treatment- | |
| | emergent Criterion 2 anaphylactic AEs will be based on the maximum severity of the specific events met by | |
| | the patient. Maximum severity of an (overall) treatment-emergent anaphylactic AE will be based on the | |
| | maximum severity within Criterion 1 and/or Criterion 2. | |
| | Allergic Reactions/Hypersensitivity Events, Nonanaphylaxis: TEAEs of allergic reaction/hypersensitivity | |
| | categorized as nonanaphylaxis events are defined by the narrow terms within Hypersensitivity SMQ | |
| | (20000214) excluding the PTs noted in Appendix 5 and excluding the anaphylactic events as defined above. | |
| Injection Site | Injection site reaction is defined using the PTs from the MedDRA HLT of Injection site reactions as defined | P2 Main Study Safety |
| Reactions | by MedDRA, excluding the following 10 PTs: | Population (Fisher's exact |
| | 1) Embolia cutis medicamentosa | test) and All Ixekizumab |
| | 2) Injection site joint discomfort | Safety Population |
| | 3) Injection site joint effusion | (Summary): |
| | 4) Injection site joint redness | TEAE by PT within HLT, |
| | 5) Injection site joint infection | SAE by PT within HLT |
| | 6) Injection site joint inflammation | (display in Spotfire), |
| | 7) Injection site joint movement impairment | AE leading to treatment |
| | 8) Injection site joint pain | discontinuation by PT within |
| | 9) Injection site joint swelling | HLT (display in Spotfire) |
| | 10) Injection site joint warmth. | |
| | Patients with TEAE of injection site reactions will be categorized into 3 groups: patients with 1 TEAE of | |
| | injection site reaction event, patients with 2 or 3 events, and patients with $\geq$ 4 events. | Listing: |
| | Redness (Scored 0-4) | TEAE (display in Spotfire) |
| | • [0] Subject's normal skin color, no increased redness | |
| | • [1] Noticeable, but very mild redness | |
| | • [2] Clearly red | |
| | • [3] Bright red | |
| | • [4] Dark with some scar formation | |
| | Swelling (Scored 0-4 after running a finger over injected area) | |
| | • [0] No bump | |
| | • [1] Barely noticeable | |
| | • [2] Clear bump but very thin | |
| | • [3] Clear bump 1-mm thick | |
| | • [4] Clear bump 2-mm thick or more | |

| Special Safety | | |
|---|---|---|
| Topic | Definition/Derivation | Analysis/Summary/Listing |
| | Pain (including burning) (Scored 0-3) • [1] Mild • [2] Moderate • [3] Severe | |
| Malignancies | Malignancy is defined using PTs from the Malignant or unspecified tumors SMQ as defined in MedDRA (SMQ: 20000091, which includes the sub-SMQs: [1] 20000194 [Malignant tumours], including sub-SMQs of 20000227 [Haematological malignant tumours] and 20000228 [Non-haematological malignant tumours]; [2] 20000195 [Tumours of unspecified malignancy], including sub-SMQs of 20000229 [Haematological tumours of unspecified malignancy] and 20000230 [Non-haematological tumours of unspecified malignancy]. Events will be summarized by the following categories: • Nonmelanoma Skin Cancer (NMSC) • Basal Cell Carcinoma, PTs include: • Basosquamous carcinoma • Basosquamous carcinoma • Basosquamous carcinoma of skin • Squamous Cell Carcinoma, PTs include: • Squamous cell carcinoma of skin • Bowen's disease • Lip squamous cell carcinoma • Skin squamous cell carcinoma metastatic • Keratoacanthoma • Malignancies excluding NMSC: all PTs in the Malignant or unspecified tumors SMQ excluding the 8 defined NMSC PTs. | P2 Main Study Safety Population (Fisher's exact test) and All Ixekizumab Safety Population (Summary): TEAE by PT within category Listing: TEAE (display in Spotfire) |
| Depressions | Depression and suicide/self-injury is defined using the PTs from the Depression and suicide/self-injury SMQ as specified in MedDRA (SMQ: 20000035, which includes the sub-SMQs: 20000037 [Suicide/self-injury] and 20000167 [Depression (excl suicide and self-injury)]). | P2 Main Study Safety Population (Fisher's exact test) and All Ixekizumab Safety Population (Summary): TEAE by PT within SMQ and sub-SMQ Listing: TEAE (display in Spotfire) |
| Inflammatory | Inflammatory Bowel Disease (IBD) will be identified using the following subcategory and MedDRA PTs. | P2 Main Study Safety |
| Bowel Disease | The narrow terms are considered IBD. Medical reviews of patients identified with broad terms are needed | Population (Fisher's exact |

| <b>Special Safety</b> | | |
|---|---|---|
| Topic | Definition/Derivation | Analysis/Summary/Listing |
| (IBD) | for final determination of patients with IBD. | test) and All Ixekizumab |
| | IBD Specific Terms (Narrow terms) | Safety Population |
| | Inflammatory Bowel Disease: Inflammatory bowel disease | (Summary): |
| | Crohn's Disease: Crohn's disease | IBD confirmed by |
| | Ulcerative Colitis: Acute haemorrhagic ulcerative colitis; Colitis ulcerative; Proctitis ulcerative | adjudication (included in AE |
| | IBD Non-Specific Terms: The PTs in this category are listed in Appendix 6. | overview) |
| | | Listing: |
| | | TEAE (display in Spotfire) |
| Interstitial | ILD is defined using the following terms: | Listing: |
| Lung Disease | Narrow terms in the Interstitial lung disease SMQ (20000042) | TEAE (display in Spotfire) |
| (ILD) | Additional 6 PTs from Eosinophilic pneumonia SMQ (20000157): | |
| | <ul> <li>Angiolymphoid hyperplasia with eosinophilia (Narrow)</li> </ul> | |
| | o Eosinophilic bronchitis (Narrow) | |
| | Hypereosinophilic syndrome (Narrow) | |
| | o Loeffler's syndrome (Narrow) | |
| | o Pulmonary eosinophilia (Narrow) | |
| | o Pulmonary vasculitis (Narrow) | |

Abbreviations: AE = adverse event; AESI = adverse event of special interest; ALP = alkaline phosphatase; ALT = alanine aminotransferase; AST = aspartate aminotransferase; DCAE = adverse event leading to discontinuation; eCRF = electronic case report form; FEAE = follow-up emergent adverse event; GGT = gamma-glutamyltransferase; HLT = high-level term; MedDRA = Medical Dictionary for Regulatory Activities; PT = preferred term; SAE = serious adverse event; SMQ = standardized MedDRA query; SOC = System Organ Class; TB = tuberculosis; TEAE = treatment emergent adverse event; ULN = upper limit of normal.

#### 6.14.4. Clinical Laboratory Evaluation

Clinical laboratory assessments include hematology, serum chemistry, urinalysis, and safety-related immune markers, such as neutrophil counts.

Laboratory test observed values at each visit (starting at baseline) and change from baseline to each scheduled visit, respectively, will be displayed in box plots for patients in the P2 of the Main Study Safety Population who have both a baseline and at least 1 postbaseline result. These box plots will be used to evaluate trends over time and to assess a potential impact of outliers on central tendency summaries.

- The scheduled visits/measurements will be included. The unscheduled visits and the repeat measurements will be excluded.
- The displays with both SI and conventional units will be provided, when different.
- The following summary statistics will be included as a table below the box plot: number of patients with a baseline and at least 1 postbaseline result, mean, SD, minimum, Q1, median, Q3, and maximum.
- Data will be summarized based on original scale.
- On the box plots of the laboratory test observed values, the lines of the reference ranges/limits (by using the large clinical trial population-based reference limits, that is, Lilly reference ranges) will be added. In cases where limits vary across age and gender, the lowest of the high limits and the highest of the low limits will be used.

The number and percentage of patients with a treatment-emergent or follow-up emergent abnormal high or low for laboratory tests will be summarized by treatment group for each safety population. The comparisons between treatment groups will be conducted using Fisher's exact test.

- All scheduled, unscheduled and repeated measurements will be included.
- In general, performing lab reference ranges will be used to define the low and high limits. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, and alkaline phosphatase (ALP) will not be included in the treatment-emergent abnormal high or low summary as a separate analysis addressing the risk of liver injury is described in Table RHCD.6.7.
- Note that the ranges are defined by a lower limit of normal (LLN) and an upper limit of normal (ULN). A result that is greater than or equal to the LLN and less than or equal to the ULN is considered to be within the normal ranges.
- For categorical laboratory tests:
  - Treatment-emergent abnormal value is defined as a change from normal at all baseline visits to abnormal at any time postbaseline during the treatment period.
  - o Follow-up emergent abnormal result is defined as a change from normal at baseline to abnormal at any time during the follow-up period.

- For continuous laboratory tests:
  - o Treatment-emergent high value is defined as a change from a value less than or equal to the ULN at all baseline visits to a value greater than the ULN at any time postbaseline during the treatment period.
  - Treatment-emergent low value is defined as a change from a value greater than or equal to the LLN at all baseline visits to a value less than the LLN at any time postbaseline during the treatment period.
  - Follow-up emergent high value is defined as a change from a value less than or equal to the ULN at baseline to a value greater than the ULN at any time postbaseline during the follow-up period.
  - o Follow-up emergent low value is defined as a change from a value greater than or equal to the LLN at baseline to a value less than the LLN at any time postbaseline during the follow-up period.

#### 6.14.4.1. Leukocytes (White Blood Cells [WBCs]) and Platelets

Further analyses will be conducted for total leukocytes, neutrophils, platelets, lymphocytes, monocytes, eosinophils, and basophils. Neutrophils will include both segmented neutrophils and absolute neutrophils (derived by adding segmented neutrophils and band neutrophil). The segmented neutrophils and absolute neutrophils will be summarized using the same categories.

Shift table will be produced showing the number and percentage of patients shifting from baseline to a minimum postbaseline result in each relevant category by treatment groups P2 Main Study Safety Population, All Ixekizumab Safety Population, and Follow-Up Safety Population:

- Scheduled visits, unscheduled visits, and repeat measurements will be included.
- Baseline is defined as the minimum result during the defined baseline period or baseline.
- Use the minimum nonmissing postbaseline value within each study period.
- The parameters and categories are:
  - <u>Leukocytes</u>:  $\ge 1 \times$  LLN, < LLN to  $\ge 3.0 \times 10^9$ /L,  $< 3.0 \times 10^9$ /L to  $\ge 2.0 \times 10^9$ /L,  $< 2.0 \times 10^9$ /L to  $\ge 1.0 \times 10^9$ /L, and  $< 1.0 \times 10^9$ /L
  - Neutrophils: segmented neutrophils and absolute neutrophils;  $\ge 1 \times LLN$ , < LLN to  $\ge 1.5 \times 10^9/L$ ,  $< 1.5 \times 10^9/L$  to  $\ge 1.0 \times 10^9/L$ ,  $< 1.0 \times 10^9/L$  to  $\ge 0.5 \times 10^9/L$ , and  $< 0.5 \times 10^9/L$
  - <u>Platelets</u>:  $\ge 1 \times LLN$ , < LLN to  $\ge 75.0 \times 10^9/L$ ,  $< 75.0 \times 10^9/L$  to  $\ge 50.0 \times 10^9/L$ ,  $< 50.0 \times 10^9/L$  to  $\ge 25.0 \times 10^9/L$ , and  $< 25.0 \times 10^9/L$
  - <u>Lymphocytes</u>:  $\ge 1 \times LLN$ , < LLN to  $\ge 0.8 \times 10^9/L$ ,  $< 0.8 \times 10^9/L$  to  $\ge 0.5 \times 10^9/L$ ,  $< 0.5 \times 10^9/L$  to  $\ge 0.2 \times 10^9/L$ , and  $< 0.2 \times 10^9/L$
- The LLNs are defined by as follow:
  - Leukocytes: LLN =  $4.0 \times 10^9$ /L
  - Neutrophils: LLN =  $2.0 \times 10^9$ /L
  - $\circ$  Lymphocytes: LLN =  $1.1 \times 10^9$ /L
  - $\circ$  Platelets: LLN =  $150 \times 10^9$ /L
- With additional categories:

- o Decreased; postbaseline category < baseline category
- o Increased; postbaseline category > baseline category
- o Same; postbaseline category = baseline category.

The change from minimum baseline to minimum postbaseline result for each of these leukocytes and platelets will be summarized graphically using a box plot for P2 Main Study Safety Population.

#### 6.14.4.2. Neutrophil Follow-Up

Neutrophil counts will be followed throughout the study. Patients will continue in Period 5 until their neutrophil counts have recovered.

The neutrophil follow-up analysis will be conducted on the Neutrophil Follow-Up Population defined as patients who have an absolute neutrophil count <1500 cells/ $\mu$ L (SI units: <1.5× 10<sup>9</sup>/L) at the last scheduled visit or early termination visit prior to entering the Post-Treatment Follow-Up Period (Period 5) and less than the patient's baseline absolute neutrophil count (that is, prior to first injection at Week 0). These patients are monitored during the Period 5 until neutrophil recovery.

Neutrophil clinical recovery is defined as an absolute neutrophil count  $\geq 1500$  cells/ $\mu$ L (SI units:  $\geq 1.5 \times 10^9$ /L) or greater than or equal to a patient's minimum absolute neutrophil count prior to first study drug injection at Week 0.

If a patient's neutrophil count has not recovered, within 12 weeks after entering the follow-up period (Visit 802), the patient will return for Visit 803 (12 weeks after Visit 802). Additional visits may be required for appropriate patient management depending upon the degree of neutropenia. If at Visit 802, a patient's has met the criteria for neutrophil recovery, the patient's participation in the study will be considered complete, unless the investigator deems additional follow-up may be necessary.

The number and percentage of patients achieving neutrophil clinical recovery will be presented by dosing regimen and week interval for Neutrophil Follow-Up Population for Post-Treatment Follow-Up Period (Period 5). The number and percentage of patients with an absolute neutrophil cell count that is at least 25%, 50%, 75%, or 100% of the patient's baseline absolute neutrophil count (that is, prior to first injection at Week 0), irrespective of absolute neutrophil minimum, will be included in the summary.

# 6.14.5. Vital Signs and Other Physical Findings

Analyses will be conducted on vital signs and physical characteristics including systolic blood pressure (mmHg), diastolic blood pressure (mmHg), pulse (bpm), weight (kg), BMI (kg/m²), and by-patient listing of vital signs and physical characteristics will be provided.

For vital signs and physical characteristics, the observed values at each visit (starting at baseline) and change from baseline to each scheduled visit, respectively, will be displayed in box plots for patients in P2 Main Study Safety Population who have both a baseline and at least 1 postbaseline result. These box plots will be used to evaluate trends over time and to assess a potential impact of outliers on central tendency summaries.

- The scheduled visits/measurements will be included. The unscheduled visits and the repeat measurements will be excluded.
- The following summary statistics will be included as a table below the box plot: number of patients with a baseline and at least 1 postbaseline result, mean, SD, minimum, Q1, median, Q3, and maximum.
- Data will be summarized based on original scale.

To assess the effect of administration of study drug on vital signs (blood pressures and pulse rate) among patients, at Weeks 0 and 12, vital signs will be measured before the first injection and 1 hour after the injection. The box plots will be produced for predose and postdose vital signs at Week 0 (Visit 2) and Week 12 (Visit 7).

The number and percentage of patients with treatment-emergent high blood pressure and pulse at any time for P2 Main Study Safety Population and All Ixekizumab Safety Population will be summarized. The comparisons between treatment groups will be conducted using Fisher's exact test.

- Table RHCD.6.8 and Table RHCD.6.9 define the limits of each category that are specified as treatment-emergent.
- All postbaseline scheduled, unscheduled and repeated measurements will be included.
- For treatment-emergent high blood pressure:
  - A treatment-emergent prehypertension is defined as a change from a value less than the low limit of prehypertension at all baseline visits to a value that is within the limits of prehypertension at any time postbaseline during the treatment period.
  - A treatment-emergent stage 1 hypertension is defined as a change from a value less than the low limit of stage 1 hypertension at all baseline visits to a value that is within the limits of stage 1 hypertension at any time postbaseline during the treatment period.
  - O A treatment-emergent stage 2 hypertension is defined as a change from a value less than the low limit of stage 2 hypertension at all baseline visits to a value that is greater than or equal to the limits of stage 2 hypertension at any time postbaseline during the treatment period.
- Treatment-emergent high or low value in pulse rate:
  - A treatment-emergent high value is defined as a change from a value less than or equal to the high limit at all baseline visits to a value greater than the high limit at any time postbaseline during the treatment period.
  - o Treatment-emergent low value is defined as a change from a value greater than or equal to the low limit at all baseline visits to a value less than the low limit at any time postbaseline during the treatment period.

Table RHCD.6.8. Blood Pressure Levels for Children by Age and Gender (Median Height)

| | | Boy | | G | irl |
|---|---|---|---|---|---|
| Ago | Hypertension | Systolic BP (mmHg) (supine or sitting – forearm at heart | Diastolic BP<br>(mmHg)<br>(supine or sitting –<br>forearm at heart | Systolic BP<br>(mmHg)<br>(supine or sitting –<br>forearm at heart | Diastolic BP<br>(mmHg)<br>(supine or sitting –<br>forearm at heart |
| Age<br>(Year) | Stage | level) | level) | level) | level) |
| (1011) | Prehypertension | $\geq 110 \text{ and } < 114$ | $\geq$ 70 and $\leq$ 74 | $\geq 108 \text{ and } < 111$ | $\geq$ 70 and $\leq$ 74 |
| 6 | Stage 1 | ≥114 and <126 | ≥74 and <87 | ≥111 and <124 | ≥74 and <86 |
| | Stage 2 | ≥126 | ≥87 | ≥124 | ≥86 |
| | Prehypertension | ≥111 and <115 | ≥72 and <76 | ≥109 and <113 | ≥71 and <75 |
| 7 | Stage 1 | ≥115 and <127 | ≥76 and <89 | ≥113 and <125 | ≥75 and <87 |
| | Stage 2 | ≥127 | ≥89 | ≥125 | ≥87 |
| | Prehypertension | ≥112 and <116 | ≥73 and <78 | ≥111 and <115 | ≥72 and <76 |
| 8 | Stage 1 | ≥116 and <128 | ≥78 and <91 | ≥115 and <127 | ≥76 and <88 |
| | Stage 2 | ≥128 | ≥91 | ≥127 | ≥88 |
| | Prehypertension | ≥114 and <118 | ≥75 and <79 | ≥113 and <117 | ≥73 and <77 |
| 9 | Stage 1 | ≥118 and <130 | ≥79 and <92 | ≥117 and <129 | ≥77 and <89 |
| | Stage 2 | ≥130 | ≥92 | ≥129 | ≥89 |
| | Prehypertension | ≥115 and <119 | ≥75 and <80 | ≥115 and <119 | ≥74 and <78 |
| 10 | Stage 1 | ≥119 and <132 | ≥80 and <93 | ≥119 and <131 | ≥78 and <91 |
| | Stage 2 | ≥132 | ≥93 | ≥131 | ≥91 |
| | Prehypertension | ≥117 and <121 | ≥76 and <80 | ≥117 and <121 | ≥75 and <79 |
| 11 | Stage 1 | ≥121 and <134 | ≥80 and <93 | ≥121 and <133 | ≥79 and <92 |
| | Stage 2 | ≥134 | ≥93 | ≥133 | ≥92 |
| | Prehypertension | ≥120 and <123 | ≥76 and <81 | ≥119 and <123 | ≥76 and <80 |
| 12 | Stage 1 | ≥123 and <136 | ≥81 and <94 | ≥123 and <135 | ≥80 and <93 |
| | Stage 2 | ≥136 | ≥94 | ≥135 | ≥93 |
| | Prehypertension | ≥120 and <126 | ≥77 and <81 | ≥120 and <124 | ≥77 and <81 |
| 13 | Stage 1 | ≥126 and <138 | ≥81 and <94 | ≥124 and <137 | ≥81 and <94 |
| | Stage 2 | ≥138 | ≥94 | ≥137 | ≥94 |
| | Prehypertension | ≥120 and <128 | ≥78 and <82 | ≥120 and <126 | ≥78 and <82 |
| 14 | Stage 1 | ≥128 and <141 | ≥82 and <95 | ≥126 and <138 | ≥82 and <95 |
| | Stage 2 | ≥141 | ≥95 | ≥138 | ≥95 |
| | Prehypertension | ≥120 and <131 | ≥79 and <83 | ≥120 and <127 | ≥79 and <83 |
| 15 | Stage 1 | ≥131 and <143 | ≥83 and <96 | ≥127 and <139 | ≥83 and <96 |
| | Stage 2 | ≥143 | ≥96 | ≥139 | ≥96 |
| | Prehypertension | ≥120 and <134 | ≥80 and <84 | ≥120 and <128 | ≥80 and <84 |
| 16 | Stage 1 | ≥134 and <146 | ≥84 and <97 | ≥128 and <140 | ≥84 and <96 |
| | Stage 2 | ≥146 | ≥97 | ≥140 | ≥96 |
| | Prehypertension | ≥120 and <136 | ≥80 and <87 | ≥120 and <129 | ≥80 and <84 |
| 17 | Stage 1 | ≥136 and <148 | ≥87 and <99 | ≥129 and <141 | ≥84 and <96 |
| | Stage 2 | ≥148 | ≥99 | ≥141 | ≥96 |
Abbreviations: BP = blood pressure; mmHg = millimeters of mercury.

Source: [NIH] The Fourth report on the Diagnosis, Evaluation, and Treatment of High Blood Pressure in Children

and Adolescents. Revised May 2005

Table RHCD.6.9. Categorical Criteria for Abnormal Treatment-Emergent Pulse Rate in Children and Adolescents Requiring Evaluation and Potential Intervention by a Health Care Professional

| Parameter | Age (year) | Low | High |
|---------------|------------|-----|------|
| Pulse (bpm) a | 6 - 9 | <60 | >150 |
| | 10 - 11 | <60 | >140 |
| | 12 - 14 | <50 | >120 |
| | 15 - 17 | <50 | >100 |

Abbreviations: bpm = beats per minute.

Source: See the Selected Reference Limits for Pulse/Heart Rate, Arterial Blood Pressure [Including Orthostasis], and Electrocardiogram Numerical Parameters for Use in Analyses of Phase 2-4 Clinical Trials guidance, located on the CV SAC Collaboration site.

### 6.14.6. Standardized Growth

Weight, height, and BMI data will be merged to the Centers for Disease Control and Prevention (CDC) standard growth data (released in 2000) by age and gender in order to compare patients' growth with the standard. Z-score and standardized percentile of weight, height, and BMI at each visit will be calculated and compared to the 2000 CDC growth charts.

The z-score and percentile calculations are based on algorithms and data provided by the National Center for Health Statistics. The details are provided in the CDC website (https://www.cdc.gov/nccdphp/dnpao/growthcharts/resources/sas.htm).

The following summaries will be provided for All Ixekizumab Safety Population:

- Baseline, endpoint and mean change of actual measure, z-score and standardized percentile of weight, height, and BMI will be summarized by month of ixekizumab exposure..
- Patient's mean weight, height, and BMI standardized percentile will be plotted versus ixekizumab exposure time.

By-patient listings of actual measures, z-scores, standardized percentiles in weight height, BMI for each visit will be provided.

# 6.14.7. Children's Depression Rating Scale, Revised (CDRS-R)

The Children's Depression Rating Scale–Revised (CDRS-R) (Poznanski and Mokros 1996) is the most widely used rating scale for assessing severity of depression and change in depressive symptoms for clinical research studies in children and adolescents with depression.

The CDRS-R was originally developed as a rating scale for children aged 6 to 12 years. It is a 17-item scale, with items ranging from 1 to 5 or 1 to 7 (the total score is the sum of the 17 items

<sup>&</sup>lt;sup>a</sup> Baseline abnormal values are defined by the value presented.

and ranges from 17-113, with higher scores indicating more depressive symptoms) and is rated by a clinician via interviews with the child and parent or legal guardian. A score of  $\geq$ 40 is indicative of depression, whereas, a score  $\leq$ 28 is often used to define remission (minimal or no symptoms) (Mayes et al. 2010).

Change from baseline to each postbaseline visits in CDRS-R total score will be analyzed using MMRM methods for P2 Main Study Safety Population.

A shift table will be produced showing the number and percentage of patients shifting from maximum baseline score to a maximum postbaseline score in categories of  $\leq$ 28,  $\geq$ 28 and  $\leq$ 40, and  $\geq$ 40 for P2 Main Study Safety Population and All Ixekizumab Safety Population.

By-patient listing of CDRS-R data will be provided.

## 6.14.8. Columbia-Suicide Severity Rating Scale (C-SSRS)

The Columbia-Suicide Severity Rating Scale (C-SSRS) is an assessment tool that evaluates suicidal ideation and behavior. Information on the C-SSRS scale can be found through the following link: http://www.cssrs.columbia.edu.

Specifically, the following outcomes are C-SSRS categories and have binary responses (yes/no). The categories have been re-ordered from the actual scale to facilitate the definitions of the composite and comparative endpoints, and to enable clarity in the presentation of the results.

Category 1 – Wish to be Dead

Category 2 – Non-specific Active Suicidal Thoughts

Category 3 – Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act

Category 4 – Active Suicidal Ideation with Some Intent to Act, without Specific Plan

Category 5 – Active Suicidal Ideation with Specific Plan and Intent

Category 6 – Preparatory Acts or Behavior

Category 7 – Aborted Attempt

Category 8 – Interrupted Attempt

Category 9 – Actual Attempt (non-fatal)

Category 10 – Completed Suicide

Self-injurious behavior without suicidal intent is also a C-SSRS outcome (although not suicide-related) and has a binary response (yes/no).

Composite endpoints based on the above categories are defined below.

- Suicidal ideation: A "yes" answer at any time during treatment to any 1 of the 5 suicidal ideation questions (Categories 1-5) on the C-SSRS.
- **Suicidal behavior:** A "yes" answer at any time during treatment to any 1 of the 5 suicidal behavior questions (Categories 6-10) on the C-SSRS.
- Suicidal ideation or behavior: A "yes" answer at any time during treatment to any 1 of the 10 suicidal ideation and behavior questions (Categories 1-10) on the C-SSRS.

The Self-Harm Supplement Form is a 1-question form that is completed, at any visit, including baseline visit, that asks for the number of suicidal behaviors, possible suicidal behaviors, or nonsuicidal self-injurious behaviors the patient has experienced since the last assessment. For each unique event identified, a questionnaire (Self-Harm Follow-up Form) which collects supplemental information on the self-injurious behavior is to be completed.

Given that few or no suicidal ideation or behaviors are anticipated, C-SSRS will be listed by patient and visit. Only patients that show suicidal ideation/behavior or self-injurious behavior without suicidal intent will be displayed (that is, if a patient's answers are all "no" for the C-SSRS, then that patient will not be displayed). However, if a patient reported any suicidal ideation/ behavior or self-injurious behavior without suicidal intent at any time point, then all his/her ideation and behavior will be displayed, even if not positive. Note that missing data should not been imputed.

The Self-Harm data will be listed by patient and visit if number of events on Self-Harm Supplement Form is not zero in the eCRF Self Harm Questionnaire Supplement.

## 6.14.9. Tanner Stage Scale

The Tanner Stage Scales are a series of line drawings that are designed to aid the investigator in appropriately assessing the sexual maturity of the subject. Data gathered will be assessed to determine that no pubertal disruption has occurred during the study. Although the line drawings were originally intended for child self-assessment, evidence suggests that pubertal assessment by the child or the parents/legal guardian is not a reliable measure of exact pubertal staging, and should be augmented by a physical examination (Rasmussen et al. 2015). The drawings will be used by the dermatologist investigator as an aid.

Shift table will be produced showing the number and percentage of patients shifting from the highest stage score at baseline to the highest postbaseline stage score by gender for each scale item for All Ixekizumab Safety Population.

A by-patient listing of Tanner stage data will be provided.

#### 6.14.10. Immunization

A by-patient listing of all immunization data will be provided. The listing will include any TEAEs occurring within 30 days after the vaccinations.

# 6.14.11. Immunogenicity

#### 6.14.11.1. Definitions and Terms

The following sample- and patient-related definitions and parameters will be used to describe the immunogenicity data.

## 6.14.11.1.1. Sample Category Definitions

Samples are classified into the following categories:

- Unevaluable sample: Sample could not be tested for ADA due to sample loss, mishandling, or errors in collection, processing, storage, and so on.
- Anti-drug antibody (ADA) Positive sample: The presences of ADA is detected and confirmed. The samples are reported as positive. If the sample is positive, a titer value is reported.
- Neutralizing anti-drug antibody (NAb) Positive sample: NAb are reported as detected.
- Anti-drug antibody (ADA) Negative sample: The presence of ADA is not detected and the assay drug tolerance level is not exceeded.
- NAb Negative sample: The presence of NAb is not detected and the assay drug tolerance level is not exceeded.
- **Inconclusive sample:** ADA/NAb is not detected in a sample, but the drug is present in the same sample at a level that can cause interference in the ADA/NAb detection method. The negative ADA/NAb result cannot be confirmed, and the sample was considered inconclusive.
  - Confirmation of a negative ADA result was based on expected ixekizumab concentrations based on PK modeling.
  - Confirmation of negative NAb results was based on ixekizumab concentrations

Figure RHCD.6.1 illustrates the relationship of some of the above terms.



Abbreviation: ADA = anti-drug antibody.

Figure RHCD.6.1. Sample definitions.

#### 6.14.11.1.2. Patient Category Definitions

The following categories are applied to patients, based on the classification of their samples:

- Unevaluable patient: a) a patient with no evaluable baseline sample and/or no evaluable postbaseline samples; b) a patient with an evaluable baseline sample, but no evaluable postbaseline sample; c) a patient with no evaluable baseline sample, but whose evaluable postbaseline values are all ADA-positive or a mix of positive and negative. Note: If all postbaseline samples are negative, the patient is considered "evaluable" and will be classified as ADA-negative.
- Evaluable patient: a) Patient with an evaluable baseline sample and at least 1 evaluable postbaseline sample (that is, sample after administration of study drug); b) patient with no evaluable baseline sample whose evaluable postbaseline samples are all ADA negative.

Figure RHCD.6.2 illustrates the relationship of the above terms.



Abbreviation: ADA = anti-drug antibody.

Figure RHCD.6.2. Patient categories (evaluable/unevaluable) based on sample status at baseline and postbaseline.

#### 6.14.11.1.3. Definitions for Clinical Interpretation of Assay Results

• Baseline: For immunogenicity analyses during Period 2, baseline is the last nonmissing observation on, or prior to, the date of the first injection of study treatment of ixekizumab (Week 0). Unless, otherwise, specified, the baseline for Overall Ixekizumab Treatment Period (Period 2, 3, and 4 combined) is defined as the last nonmissing observation on, or prior to, the date of first injection of ixekizumab. For patients originally randomized to ixekizumab during Period 2, baseline is the last nonmissing observation on, or prior to, the date of the first injection of study treatment for Period 2 (Week 0). For patients who are not originally randomized to ixekizumab in Period 2, baseline is the last nonmissing observation on, or prior to, the date of the first injection of ixekizumab (see Table RHCD.6.10 for further details).

Table RHCD.6.10. Baseline Definition for Immunogenicity Analyses for Overall Ixekizumab Treatment Period

| Treatment Assignment<br>for Double-Blind<br>Treatment Period<br>(Period 2) | Treatment Assignment<br>for Maintenance Period<br>(Period 3) and Extension<br>Period (Period 4) or<br>Period 3 Only (Protocol<br>Addendum RHCD[2]) | Treatment Assignment<br>for 48-Week Double-<br>Blind, Randomized<br>Withdrawal Period<br>(Protocol Addendum<br>RHCD[2] Period 4) | Baseline for Overall<br>Ixekizumab Treatment<br>Period Analysis <sup>a</sup> |
|---|---|---|---|
| Ixekizumab | Ixekizumab | NA | Week 0 |
| Placebo | Ixekizumab | NA | Week 12 |
| Ixekizumab | Ixekizumab | Ixekizumab | Week 0 |
| Ixekizumab | Ixekizumab | Placebo | Week 0 |
| Etanercept | Ixekizumab | Ixekizumab | Week 20 |
| Etanercept | Ixekizumab | Placebo | Week 20 |
| Placebo | Ixekizumab | Ixekizumab | Week 12 |
| Placebo | Ixekizumab | Placebo | Week 12 |

Abbreviations: NA = not applicable.

- Baseline ADA-positive (preexisting antibody): ADA detected in a sample collected at baseline.
- **Baseline ADA-negative:** ADA is not detected in a sample collected at baseline.
- Treatment-emergent-(TE-) ADA positive: a) a patient with a  $\geq$ 4-fold increase over a positive baseline antibody titer (Tier 3); or b) for a negative baseline titer, a patient with an increase from the baseline to a level of  $\geq$ 1:10.
- **TE-ADA inconclusive:** A patient without a TE-ADA positive sample and with at least 1 sample for which drug levels may interfere with the ADA assay.
- **TE-ADA negative:** A patient who is evaluable for TE-ADA and is not either TE-ADA positive or TE-ADA inconclusive.

<sup>&</sup>lt;sup>a</sup> Last non-missing observation on, or prior to, the date of the first injection of study treatment at the defined week.



Figure RHCD.6.3 illustrates the relationship of some of these terms.

Abbreviation: ADA = anti-drug antibody.

Figure RHCD.6.3. Relationship of terms for clinical interpretation of assay results for evaluable patients.

- **Incidence of TE-ADA:** Patients with TE-ADA as a proportion of the evaluable patient population during the treatment period. This excludes unevaluable patients.
- Follow-up-emergent ADA: ADA is first detected during the follow-up period, after study drug administration is discontinued. This category includes patients negative at baseline who increased to ≥1:10 titer (4-fold increase/ 2 dilutions) after baseline in the follow-up period or patients ADA positive at baseline and increased at least 4-fold (2 dilutions) over baseline for the first time in the follow-up period.
- **Incidence of follow-up emergent ADA:** Patients with follow-up-emergent ADA as a proportion of the follow-up evaluable patient population. This excludes unevaluable patients.

All ADA positive samples will be evaluated for NAb. Definitions for NAb patient status will be defined as follows:

- **NAb-positive:** A patient where a NAb positive result is detected for ≥1 TE-ADA positive samples.
- NAb-inconclusive: A patient without a NAb positive sample and with at least 1 sample for which drug levels may interfere with the NAb assay.
- **NAb-negative:** A patient who is evaluable for NAb and is not either NAb positive or NAb inconclusive.

A flow chart that reflects the connection between the analytical test results and the clinical interpretation based on the definitions is shown in Figure RHCD.6.4.



Figure RHCD.6.4. Flow chart of ADA assessment with clinical interpretation of the various result possibilities.

#### 6.14.11.2. Immunogenicity Analyses

Immunogenicity evaluable patients will be identified as TE-ADA positive, TE-ADA negative, or TE-ADA inconclusive, according to the definitions provided in Section 6.14.11.1.2 and further grouped into TE-ADA status groups and time-varying TE-ADA status groups:

#### **TE-ADA Status Groups:**

- TE-ADA status (positive, negative, or inconclusive)
- NAb status (positive, negative, or inconclusive) for TE-ADA positive patients
- TE-ADA titer groups for TE-ADA positive patients:
  - o Low Titer: TE-ADA titer value (LOCF) <1:160
  - o Moderate Titer: TE-ADA titer value (LOCF) ≥1:160 and <1:1280
  - o High Titer: TE-ADA titer value (LOCF) ≥1:1280

### **Time-Varying TE-ADA Status Groups:**

Individual ADA samples will be ascribed into 3 different dichotomous variables as explained in Table RHCD.6.11. Each variable has possible values of a "greater-TE-ADA status" or a "lesser-TE-ADA status," in the sense that the level of TE-ADA detected in the greater-TE-ADA category is higher than in the lesser-TE-ADA category.

Table RHCD.6.11. TE-ADA Status Dichotomous Variables for AE Analysis

| <b>TE-ADA Status Dichotomous</b> | | |
|---|---|---|
| Variable | Greater-TE-ADA Status | Lesser-TE-ADA Status |
| TE-ADA positive | TE-ADA positive | not TE-ADA positive |
| TE-ADA moderate-to-high | TE-ADA positive with moderate | not TE-ADA positive, or TE-ADA positive |
| | titer or high titer | with low titer |
| TE-ADA high status | TE-ADA positive with high titer | not TE-ADA positive, or TE-ADA positive |
| | | with low or moderate titer |

Abbreviations: TE-ADA = treatment-emergent antidrug antibodies/

Note: for purpose of this analysis, TE-ADA Inconclusive is taken to be "not TE-ADA positive." A TE-ADA low is defined as a TE-ADA positive with a titer value <1:160; a TE-ADA moderate is defined as a TE-ADA positive with a titer value ≥1:160 and <1:1280; and a TE-ADA high is defined as a TE-ADA positive with a titer value ≥1:1280.

For each TE-ADA status dichotomous variable, a time-varying TE-ADA status will be computed. At time *t*, the TE-ADA status is taken to be the highest of the TE-ADA values bracketing time *t*. More formally, the TE-ADA status at time *t* is given by the greater of: (a) the TE-ADA status at the most-recent postbaseline measurement prior to *t*; and (b) the TE-ADA status at the first TE-ADA postbaseline measurement at or after time *t*. In this computation, "greater" is given by the greater-TE-ADA status of Table RHCD.6.11. If there is no value satisfying criterion (a), then the value (b) is used. Similarly, if there is no value (b), then the value (a) is used.

For each TE-ADA status dichotomous variable, patients will be categorized according to whether they were: (1) always in lesser-TE-ADA status postbaseline; or (2) at some point postbaseline, were in greater-TE-ADA status.

## 6.14.11.2.1. Analyses of Characteristics of ADA Immune Response

The analyses of ADA effects will be conducted on all evaluable patients within the defined Safety Population for Period 2, All Ixekizumab Population for Combined Treatment Period (Period 2, 3, and 4 combined), and Follow-Up Population for Period 5.

The overall frequency and percentage (incidence) of patients will be summarized for the TE-ADA status groups and the time-varying TE-ADA status groups. Scheduled visits, unscheduled visits, and repeat measurements will be included.

The time to the development of TE-ADAs (TE-ADA positive, low titer, moderate titer, high titer, and NAb positive) will be calculated as follows:

Time to development of TE-ADAs/NAb (in weeks) = (Date of development of TE-ADAs/NAb – Date of first injection of study treatment + 1) / 7.

If a patient has not developed TE-ADAs/NAbs, he/she will be censored at the date of the last immunogenicity assessment. If a patient does not have any postbaseline assessments for immunogenicity, he/she will be censored at the date of randomization.

Descriptive statistics, including 25th percentile, 50th percentile (median), 75th percentile, and corresponding 95% CIs, as well as probability of TE-ADA/NAb positive by endpoint summarized by treatment group, will also be provided if sufficient data is present. A Kaplan-Meier plot of the time to development of treatment-emergent ADA/NAb will be presented by treatment group, also if sufficient data is present. Caution should be exercised in the interpretation of time-to-event analyses and related statistics, given the limited sampling scheme for immunogenicity testing.

For each TE-ADA status dichotomous variable (as defined in Table RHCD.6.11), summaries will be provided of the total postbaseline time in the greater-TE-ADA status for patients who were at some point postbaseline in the greater-TE-ADA status group. Postbaseline time in greater-TE-ADA status for each patient will be aggregated.

A by-patient listing to include treatment, visit date, visit, ADA result, TE-ADA result, NAb result, ADA titer value, ixekizumab concentration, and ADA and NAb inconclusive results will also be provided, for patients with any one sample of ADA (or NAb) positive or inconclusive.

## 6.14.11.2.2. Analyses of Treatment-Emergent ADA Effects on Efficacy

Efficacy analyses for Period 2 will be conducted on all evaluable patients within the ITT Population.

Analyses will be performed to examine how patient TE-ADA effects PASI 75 and sPGA(0,1) response rates at week 12 with NRI by the TE-ADA status groups as described in Section 6.14.11.1.2.

A logistic regression model with treatment group, TE-ADA status and the interaction of treatment group-by-TE-ADA status included as factors will be used to test the interaction of treatment group -by-TE-ADA status for ITT Population during Period 2. The p-value associated

with the interaction term will be used to assess if the treatment groups effect is consistent across TE-ADA status groups. When the interaction term is statistically significant, the association between responder status and treatment groups depends, in some manner, on the status. The interaction will be tested at the 10% significance level. Treatment group differences will be evaluated within each TE-ADA subgroup using Fisher's exact test, regardless of whether the interaction is statistically significant.

## 6.14.11.2.3. Analyses of Treatment-Emergent ADA on Specific Adverse Events

The analyses of TE-ADA effects on safety will be conducted on all evaluable patients within the defined Safety Population for Period 2 and All Ixekizumab Population for combined Periods 2, 3, and 4.

Adverse events of special interest of allergic reaction/hypersensitivity (anaphylaxis and nonanaphylaxis) and of injection-site reactions will be included in an assessment of AE to TE-ADA over time. See Section 6.14.3.1 for the definitions of the AESIs. Timing of an AE will be taken to be the reported AE start date.

For each TE-ADA status dichotomous variable (as defined in Table RHCD.6.11), patients will be categorized according to whether they were: (1) always in lesser-TE-ADA status postbaseline; or (2) at some point postbaseline, were in greater-TE-ADA status. For each AESI, within the time-varying TE-ADA status groups, a summary will be provided of the number of patients who had no event, events only while in lesser-TE-ADA status for group (1), or – for group (2) – at least 1 event while in greater-TE-ADA status.

Additionally, summaries will be provided of the total number of AESI events (with unique start dates) by time-varying TE-ADA status groups at the event date. The summaries will aggregate time respectively in greater-TE-ADA status and in lesser-TE-ADA status, along with the event rates (rates per 100 patient-years) relative to those aggregate times.

By-patient listings will be provided of patients with TE-ADA who experience a treatmentemergent allergic reaction/hypersensitivity reaction or an injection site reaction.

## 6.15. Subgroup Analyses

# 6.15.1. Efficacy Subgroup Analyses

Subgroup analysis will be conducted for the co-primary endpoints of proportion of patients achieving PASI 75 and sPGA (0,1) response using the ITT Population for Period 2.

Subgroups to be evaluated may include gender, age, weight, ethnicity, region, geographic region, baseline disease severity, duration of disease, previous nonbiologic systemic therapy, and previous biologic therapy.

A logistic regression model with treatment, subgroup, and interaction of subgroup-by-treatment included as factors will be used. The subgroup-by-treatment interaction will be tested at the significance level of 0.10. Treatment group differences will be evaluated within each category of the subgroup using the Fisher's exact test, regardless of whether the interaction is statistically

significant. Missing data will be imputed using NRI. If any group within the subgroup is <10% of the Total ITT Population, only summaries of the efficacy data will be provided (that is, no inferential testing).

The following subgroups will be analyzed:

- Patient Demographics Subgroups:
  - o Gender
  - o Age Group (years): <12; and  $\ge 12$
  - Weight Category: <25 kg;  $\ge 25 \text{ to } \le 50 \text{ kg}$ ; and >50 kg (only summary statistics)
  - o Ethnicity
- Geographic Region Subgroups:
  - o Geographic Region: North America; Europe Union; and Rest of the World
- Baseline Severity of Disease Subgroups:
  - o Baseline PASI category: <20; and ≥20
  - o Baseline sPGA category: 3; 4; and 5
  - o Baseline sPGA category: 3; and combined 4 or 5
  - o Baseline BSA category: <20%; and ≥20%
- Previous Psoriasis Therapy Subgroups:
  - Previous Nonbiologic Systemic Therapy (methotrexate, cyclosporine, retinoids, corticosteroid, fumaric acid derivatives, apremilast, psoralen and ultraviolet A [PUVA]): never used; and ever used
  - o Previous Biologic Systemic Therapy: never used; and ever used
- Other Patient Characteristics Subgroups:
  - Duration of Disease (in years): >0.5 and <=1; >1 and <=1.5; >1.5 and <=2; and >2

Additional subgroup analyses on efficacy may be performed, as deemed appropriate and necessary.

# 6.15.2. Safety Subgroup Analyses

Safety subgroup analysis for common TEAEs and AESI of infections and injection site reactions will be summarized for P2 Main Study Safety Population. The common TEAEs will be presented by decreasing frequency of PT within SOC. The infections and injection site reactions will be presented by decreasing frequency of PT

A logistic regression model with treatment, subgroup, and the interaction of subgroup-by-treatment included as factors will be used. The subgroup-by- treatment interaction will be tested at the significance level of 0.10. The response variable will be each AE. Treatment group differences will be evaluated within each category of the subgroup using Fisher's exact test, regardless of whether the interaction is statistically significant. If any group within the subgroup is <10% of the total population, only the descriptive statistics will be provided for that subgroup (that is, no inferential testing).

The following subgroups will be analyzed:

- Weight Category:  $<25 \text{ kg}; \ge 25 \text{ to } \le 50 \text{ kg}; \text{ and } >50 \text{ kg}$
- Geographic Region: North America; Europe Union; and Rest of the World

Additional subgroup analyses on safety may be performed, as deemed appropriate and necessary.

### 6.16. Protocol Deviations

Protocol deviations will be identified throughout the study. Important protocol deviations are defined as those deviations from the protocol likely to have a significant impact on the completeness, accuracy, and/or reliability of the study data, or that may significantly affect subject's rights, safety, or well-being.

The major protocol deviations, which are the subset of the important protocol deviations, are the protocol deviations that might have impact on the efficacy and/or safety results. The impact of major protocol deviations on the efficacy results will be investigated by assessing the robustness of the study results and conclusions to the choice of analysis population, both by including and excluding the data potentially affected by major protocol deviations. As specified in Section 6.1.1, the PPS Population is defined as all randomized patients who do not have major protocol deviations.

Table RHCD.6.12 includes the categories and subcategories of important protocol deviations, whether or not these deviations are major protocol violations, the action to be taken regarding the exclusion of patients from PPS, the source of the deviation identified, and the statistical programming guidance for the clinical study report (CSR).

The number and percentage of patients having important protocol deviation(s) will be summarized within category and subcategory of deviations by treatment group for the ITT Population for the Double-Blind Treatment Period (Period 2).

A by-patient listing of important protocol deviations will be provided.

 Table RHCD.6.12.
 Identification and Action of Important Protocol Deviations

| | | Source to<br>Identify | |
|---|---|---|---|
| Important Protocol Deviation | Action for PPS | Protocol | |
| Category/Subcategory/Study Specific | Analysis | <b>Deviation</b> <sup>a</sup> | Statistical Programming Guidance for Clinical Study Report |
| Category: Eligibility | | | |
| Subcategory: Inclusion/Exclusion | | | |
| [1] No confirmed diagnosis of moderate-to- | Excluded from | Monitor and | Either from monitor's list, or, if date of diagnosis of Ps is missing or |
| severe plaque-type Ps for at least 6 months prior to Visit 2 | PPS | Stats | less than 6 months prior to Visit 2. |
| [2] PASI score <12 or sPGA <3 or BSA | Excluded from | Monitor and | Either from monitor's list, or, If PASI score <12 or sPGA <3 or |
| involvement <10% at Visit 1 or Visit 2 | PPS | Stats | BSA involvement <10% or any missing at Visit 1 or Visit 2. |
| [3] Not a candidate for phototherapy or systemic therapy | Excluded from PPS | Monitor | From monitor's list. |
| [4] Age <6 years or ≥18 years | Excluded from PPS | Monitor | From monitor's list. |
| [5] Improper informed consent | Do not exclude from PPS | Monitor and<br>Stats | Either from monitor's list, or, if patient informed consent date is after Visit 1 date. |
| [6] Immunizations are not up to date in agreement with current immunization guidelines | Excluded from PPS | Monitor | From monitor's list. |
| [7] Have pustular, erythrodermic, and/or guttate forms of Ps | Excluded from PPS | Monitor | From monitor's list. |
| [8] With drug-induced Ps | Excluded from PPS | Monitor | From monitor's list. |
| [9] Have clinical and/or laboratory evidence of untreated latent or active TB | Excluded from PPS | Monitor and<br>Stats | From monitor's list, or If a PPD skin test response of ≥5 mm in duration, or a "positive" for the QuantiFERON-TB® Gold test or T-SPOT.TB test. |

| Important Protocol Deviation Category/Subcategory/Study Specific | Action for PPS<br>Analysis | Source to Identify Protocol Deviation <sup>a</sup> | Statistical Programming Guidance for Clinical Study Report |
|---|---|---|---|
| [10] Have evidence of or test positive for hepatitis B virus (HBV) | Do not exclude<br>from PPS | Monitor and<br>Stats | Either from monitor's list, or, if test positive for HBV at Visit 1 by testing: 1) positive for hepatitis B surface antigen (HBsAg+); or 2) positive for anti-hepatitis B core antibody (HBcAb+) and are HBV deoxyribonucleic acid (DNA) positive. Note: Subjects who are HBcAb+ and HBV DNA negative may be enrolled in the study. Subjects who meet these criteria at screening will be identified by the central laboratory and monitored during the study. |
| [11] Have evidence of or test positive for hepatitis C virus (HCV) | Do not exclude from PPS | Monitor and<br>Stats | Either from monitor's list, or, if test positive for HCV at Visit 1 by testing: 1) positive for hepatitis C antibody (anti-HCVAb); and 2) positive via a confirmatory test for HCV. |
| [13] Have any varicella-zoster virus infection within 12 weeks of Visit 2 | Do not exclude from PPS | Monitor | From monitor's list. |
| [22] Presence of significant uncontrolled neuropsychiatric disorder, or have had a recent past history of a suicide attempt, or marked a yes to C-SSRS question 4 or 5 on ideation or yes to suicide behaviors | Do not exclude from PPS | Monitor | From monitor's list |
| [24] Have not had any immunizations, or are not up to date on immunizations recommended by country specific Pediatric guidance | Do not exclude from PPS | Monitor | From monitor's list. |
| [29] At Visit 1, have a neutrophil count <1500 cells/ $\mu$ L (<1.50×10 <sup>9</sup> / $\mu$ L or <1.50 GI/L), a lymphocyte count <800 cells/ $\mu$ L (<0.80×10 <sup>9</sup> / $\mu$ L or <0.80 GI/L), a platelet count <100,000 cells/ $\mu$ L (<100×10 <sup>9</sup> / $\mu$ L or <100 GI/L) | Do not exclude from PPS | Monitor and<br>Stats | Either from monitor's list, or, If have a neutrophil count <1500 cells/ $\mu$ L (<1.50x10 <sup>9</sup> / $\mu$ L or <1.50 GI/L, a lymphocyte count <800 cells/ $\mu$ L (<0.80x10 <sup>9</sup> / $\mu$ L or <0.80 GI/L), a platelet count <100,000 cells/ $\mu$ L (<100x10 <sup>9</sup> / $\mu$ L or <100 GI/L) or missing at Visit 1. |
| [32] Previously treated with etanercept | Excluded from PPS | Monitor and<br>Stats | Either from monitor's list, or, If have etanercept in the CRFs "Prior Therapy: Psoriasis". |

| Important Protocol Deviation Category/Subcategory/Study Specific | Action for PPS<br>Analysis | Source to Identify Protocol Deviation <sup>a</sup> | Statistical Programming Guidance for Clinical Study Report |
|---|---|---|---|
| [33] Have used any therapeutic agent targeted at reducing interleukin-17 (IL-17) | Excluded from PPS | Monitor | From monitor's list. |
| [35] Had a live vaccination within 12 weeks prior to Visit 2, or intend to have a live vaccination during the course of the study or within 12 weeks of completing treatment in this study, or have participated in a vaccine clinical study within 12 weeks prior to Visit 2 | Do not exclude from PPS | Monitor | From monitor's list. |
| Category: Study Procedures | | | |
| Subcategory: Violation of Discontinuation ( | Criteria | | |
| [D1] ALT or AST >8× ULN | Do not exclude from PPS | Monitor and<br>Stats | Either from monitor's list, or, if a patient still receives study treatment after 10 days with confirmed ALT or AST >8× ULN (defined as a test of 8× ULN and a retest within 10 days still >8 × ULN; if not retest, use the test as the confirmed). |
| [D2] ALT or AST >5× ULN for more than 2 weeks | Do not exclude from PPS | Monitor and<br>Stats | Either from monitor's list, or, if a patient still receives study treatment after 24 days with confirmed ALT or AST >5× ULN (defined as a test of 5× ULN and a retest within 14 days still >5× ULN; if not retest, use the test as the confirmed). |
| [D3] ALT or AST >3× ULN and TBL >2 × ULN or prothrombin time >1.5 time ULN | Do not exclude<br>from PPS | Monitor and<br>Stats | Either from monitor's list, or, if a patient still receives study treatment after 10 days with confirmed ALT or AST >3× ULN and TBL >2× ULN or prothrombin time >1.5× ULN (defined as a test of 3× ULN and 2× ULN or 1.5× ULN and a retest within 10 days still >3× ULN and 2× ULN or 1.5× ULN; if not retest, use the test as the confirmed). |
| [D4] ALT or AST >3× ULN with the appearance of fatigue, nausea, vomiting, right upper-quadrant pain or tenderness, fever, rash, and/or eosinophilia (>5%) | Do not exclude<br>from PPS | Monitor and<br>Stats | Either from monitor's list, or, If a patient still receives study treatment after 10 days with confirmed ALT or AST >3× ULN with the appearance of fatigue, nausea, vomiting, right upper-quadrant pain or tenderness, fever, rash, and/or eosinophilia (>5%) (defined as a test of 3× ULN and a retest within 10 days still >3× ULN; if not retest, use the test as the confirmed). |

| Important Protocol Deviation Category/Subcategory/Study Specific | Action for PPS Analysis | Source to Identify Protocol Deviation <sup>a</sup> | Statistical Programming Guidance for Clinical Study Report |
|---|---|---|---|
| [D5] ALP >3× ULN | Do not exclude from PPS | Monitor and<br>Stats | Either from monitor's list, or, If a patient still receives study treatment after 10 days with confirmed ALP >3× ULN (defined as a test of 3× ULN and a retest within 10 days still >3× ULN; if not retest, use the test as the confirmed). |
| [D6] ALP >2.5× ULN and TBL >2× ULN | Do not exclude from PPS | Monitor and<br>Stats | Either from monitor's list, or, If a patient still receives study treatment after 10 days with confirmed ALP >2.5× ULN and TBL >2× ULN (defined as a test of 3× ULN and 2× ULN and a retest within 10 days still >3× ULN and 2× ULN; if not retest, use the test as the confirmed). |
| [D7] ALP >2.5× ULN with the appearance of fatigue, nausea, vomiting, right upper-quadrant pain or tenderness, fever, rash, and/or eosinophilia (>5%) | Do not exclude<br>from PPS | Monitor and<br>Stats | Either from monitor's list, or, If a patient still receives study treatment after 10 days with confirmed ALP >2.5× ULN with the appearance of fatigue, nausea, vomiting, right upper-quadrant pain or tenderness, fever, rash, and/or eosinophilia (>5%) (defined as a test of 2.5× ULN and a retest within 10 days still >2.5× ULN; if not retest, use the test as the confirmed). |
| [D8] Neutrophil counts <500 cells/ $\mu$ L, or $\geq$ 500 and <1000 cells/ $\mu$ L based on 2 test results, or $\geq$ 1000 and <1500 cells/ $\mu$ L based on 3 test results and a concurrent infection | Do not exclude<br>from PPS | Monitor and<br>Stats | Either from monitor's list, or, If a patient still receives study treatment after 10 days with confirmed segmented neutrophil counts <500 cells/μL (defined as a test of <500 cells/μL and a retest within 10 days still <500 cells/μL; if no retest, use the test as the confirmed). |
| [D9] Total WBC count <2000 cells/μL | Do not exclude from PPS | Monitor and<br>Stats | Either from monitor's list, or, If a patient still receives study treatment after 10 days with confirmed total WBC count <2000 cells/ $\mu$ L (defined as a test of <2000 cells/ $\mu$ L and a retest within 10 days still <2000 cells/ $\mu$ L; if no retest, use the test as the confirmed) |
| [D10] Lymphocyte count <200 cells/μL | Do not exclude<br>from PPS | Monitor and<br>Stats | Either from monitor's list, or, If a patient still receives study treatment after 10 days with confirmed lymphocyte count <200 cells/μL (defined as a test of <200 cells/μL and a retest within 10 days still <200 cells/μL; if no retest, use the test as the confirmed). |

| Important Protocol Deviation | Action for PPS | Source to Identify Protocol | |
|---|---|---|---|
| Category/Subcategory/Study Specific | Analysis | <b>Deviation</b> <sup>a</sup> | Statistical Programming Guidance for Clinical Study Report |
| [D11] Platelet count <50,000 cells/μL | Do not exclude from PPS | Monitor and<br>Stats | Either from monitor's list, or, If a patient still receives study treatment after 10 days with confirmed platelet count $<\!50,\!000$ cells/ $\mu$ L (defined as a test of $<\!50,\!000$ cells/ $\mu$ L and a retest within 10 days still $<\!50,\!000$ cells/ $\mu$ L; if no retest, use the test as the confirmed). |
| [D12] Subject BP readings are greater than 95 <sup>th</sup> percentile at 3 consecutive study visits | Do not exclude from PPS | Monitor | From monitor's list. |
| [D13] A severe AE or an SAE, or a clinically significant change in a laboratory value | Do not exclude from PPS | Monitor and<br>Stats | Either from monitor's list, or, If patient still receives study treatment on the same day or after the date with an AE or SAE. |
| [D14] Clinically significant systemic<br>hypersensitivity reaction that does not<br>respond to treatment | Do not exclude from PPS | Monitor | From monitor's list. |
| [D15] Patient became pregnant | Do not exclude from PPS | Monitor | From monitor's list. |
| [D16] Patient developed a malignancy (more than 2 nonmelanoma skin cancers) | Do not exclude from PPS | Monitor | From monitor's list. |
| [D17] Patient has a positive TB test using PPD or QuantiFERON®-TB Gold | Do not exclude from PPS | Monitor | From monitor's list. |
| [D18] Change in disease phenotype | Excluded from PPS | Monitor | From monitor's list. |
| [D19] Patient requires treatment with another therapeutic agent that has been demonstrated to be effective for the treatment of Ps | Excluded from PPS | Monitor | From monitor's list. |
| [D20] Enrollment in any other clinical trial involving an investigational product or enrollment in any other type of medical research judged not to be scientifically or medically compatible with this study | Excluded from PPS | Monitor | From monitor's list. |
| [D21] The investigator or attending physician decides that the patient should be withdrawn from the study treatment | Do not exclude from PPS | Monitor | From monitor's list. |

| Important Protocol Deviation Category/Subcategory/Study Specific | Action for PPS<br>Analysis | Source to Identify Protocol Deviation <sup>a</sup> | Statistical Programming Guidance for Clinical Study Report |
|---|---|---|---|
| [D22] The patient (or guardian) requests to be withdrawn from the study treatment | Do not exclude from PPS | Monitor | From monitor's list. |
| [D23] The patient, at any time during the study, scores ≥5 for Item 13 on the CDRS-R. Or | Do not exclude from PPS | Monitor and<br>Stats | Either from monitor's list, or, score ≥5 to Item 13 (Suicidal Ideation) of CDRS-R. |
| [D24] Develops active suicidal ideation with some intent to act with or without a specific plan | Do not exclude from PPS | Monitor and<br>Stats | Either from monitor's list, or, yes to question 4 or 5 on the "Suicidal Ideation" Portion of C-SSRS. |
| [D25] Develops suicide-related behaviors as recorded on C-SSRS | Do not exclude from PPS | Monitor and<br>Stats | Either from monitor's list, or, yes to question "suicidal behavior" on the "Suicidal Behavior" Portion of C-SSRS. |
| [D26] It is recommended that the subject be assessed by an appropriately trained professional to assist in deciding whether the subject is to be discontinued from the study | Do not exclude from PPS | Monitor | From monitor's list. |
| [D27] Investigator or Lilly stopped the patient participation | Do not exclude from PPS | Monitor | From monitor's list. |
| Category: Study Procedures | | | |
| Subcategory: Excluded Con-meds | Excluded from PPS | Monitor and<br>Stats | Either from monitor's list, or If patient takes prohibited concomitant medication. Note: Prohibited concomitant medication will be provided by medical in a separate file. |
| Subcategory: Other | | | |
| Missing CDRS-R total score: missing baseline or any scheduled visit prior to discontinuation visit | Do not exclude from PPS | Stats | If missing CDRS-R total score baseline or any scheduled visit prior to discontinuation visit. |
| Missing C-SSRS: missing baseline or any scheduled visit prior to discontinuation visit | Do not exclude from PPS | Stats | If missing C-SSRS baseline or any scheduled visit prior to discontinuation visit. C-SSRS is missing if the whole questionnaire is missing. |

| Important Protocol Deviation Category/Subcategory/Study Specific Missing sPGA: not having Work 12 | Action for PPS Analysis Do not exclude | Source to Identify Protocol Deviationa | Statistical Programming Guidance for Clinical Study Report If not having Week 12 sPGA measurement for patient who have |
|---|---|---|---|
| Missing sPGA: not having Week 12 measurement for patients who have completed Week 12 | from PPS. Note:<br>such patients will<br>be treated as<br>nonresponders at<br>Week 12 | Suis | completed week 12. |
| Missing PASI: not having Week 12 measurement for patients who have completed Week 12 | Do not exclude<br>from PPS. Note:<br>such patients will<br>be treated as<br>nonresponders at<br>Week 12 | Stats | If not having Week 12 PASI measurement for patient who have completed week 12. |
| Had unqualified site personnel perform clinical safety and/or efficacy assessments | Do not exclude from PPS | Monitor | From monitor's list. |
| Missing parents/other adult to respond CDRS-R scale at any visit | Do not exclude from PPS | Monitor | From monitor's list. |
| Missing or Unqualified blinded assessor | Do not exclude from PPS | Monitor | From monitor's list. |
| Category: Investigational Product | | | |
| Subcategory: Treatment Assignment/Rando | | G | ICHWIDG 4 1 1 1 1 1 1 4 4 1 1 1 1 1 1 1 |
| Took incorrect study medication | Do not exclude<br>from PPS.<br>Analyze "As<br>randomized" or<br>"As assigned." | Stats | If IWRS study drug dispense data not match with the treatment label identifier on the Exposure as Collected eCRF page. |
| Moderate-to-severe patients from etanercept approved countries randomized as severe | Do not exclude from PPS | Monitor and<br>Stats | Either from monitor's list, or If patient with PASI <20 and sPGA <4 at baseline received etanercept in P2. |

| Important Protocol Deviation Category/Subcategory/Study Specific | Action for PPS<br>Analysis | Source to<br>Identify<br>Protocol<br>Deviation <sup>a</sup> | Statistical Programming Guidance for Clinical Study Report |
|---|---|---|---|
| Subcategory: Compliance | Excluded from PPS | Stats | If non-compliant with study medication regimen or over-dose during the treatment period. Note: Non-compliance with therapy is defined to be missing more than 20% of expected doses and missing 2 or more consecutive doses; over-dose is defined as to take more injections at the same time point than specified in the protocol. |
| Subcategory: Patient took medication not fit for use | Do not excluded from PPS | Monitor | From monitor's list. |
| Subcategory: Other | I | l | |
| Randomized but did not take any study medication | Excluded from PPS | Stats | If a patient is randomized but does not take any study medication. |
| Overdose/ Underdose in terms of actual volume of IP | Excluded from PPS | Monitor | From monitor's list. |
| Category: Safety | | | |
| Subcategory: SAEs | | | |
| Failure to report within 24 hours of the PI aware | Do not Excluded from PPS | Monitor | From monitor's list. |
| Category: Informed Consent | | | |
| Subcategory: Informed Consent not<br>Obtained/Missing/Late | Excluded from PPS | Monitor and Stats | Either from monitor's list, or, if patient informed consent date is after Visit 1 date or missing informed consent. |
| Subcategory: Improper Informed Consent | Do not Excluded from PPS | Monitor | From monitor's list. |
| Category: Administrative/Oversight | | | |
| Subcategory: Reg/Ethic Approvals | Excluded from PPS | Monitor | From monitor's list. |
| Subcategory: Other | | | |
| Enrolled in a site with significant GCP noncompliance issue | Excluded from PPS | Monitor | From monitor's list. |

Abbreviations: AE = adverse event; BCG = Bacille de Calmette et Guérin; BSA = body surface area; CDRS-R = Children's Depression Rating Scale—Revised; Con-Meds = concomitant medications; C-SSRS = Columbia—Suicide Severity Rating Scale; DV = protocol deviations; eCRF = electronic case report form; GCP = good clinical practice; IgG = immunoglobulin G; IL = interleukin; ITT = intent-to-treat; IV = intravenous; IWRS = interactive web-response system; PASI = Psoriasis Area and Severity Index; PPD = purified protein derivative; PPS = per protocol set; Ps = psoriasis; PsA = psoriatic arthritis; Reg = regulatory; SAE = serious adverse event; sPGA = static Physician Global Assessment; stats = statistics; TB = tuberculosis; TBL = total bilirubin.

- The term "Monitor" indicates the protocol deviation will be identified by site monitors and entered into monitor's list using a spreadsheet. The spreadsheet will be exported as Study Data Tabulation Model (SDTM) DV domain.
  - The term "Stats" indicates the protocol deviation will be programmed based on data in clinical database by statistical programmers with the statistical programming guidance provided as the last column. The detailed programming specification will be documented in Analysis Data Model (ADaM) specification.

The terms "Monitor and Stats" indicates the protocol deviation will be a combination of monitor's list (SDTM.DV domain) and statistical programming from clinical database, the deviation will show if either source identifies.

## 6.17. Interim Analyses and Data Monitoring

Two planned interim analyses will be conducted with an conditional third dependent upon enrollment.

A staggered approach to enrollment by weight group will be used so that a minimum of 15 subjects >12 years and >50 kg will be enrolled and safety evaluated for the initial 12 weeks of dosing before opening enrollment in the middle weight group (25 to 50 kg).

When approximately 15 subjects have enrolled in the middle weight group and completed up to Week 12, an analysis of all available PK data will be conducted to confirm that exposures are within the range expected. All safety data from these subjects will also be analyzed at this time in addition to select efficacy data. Doses for the remaining subjects in the study will be confirmed, based on these analyses. Once confirmed, all weight groups will be open for enrollment of the remaining subjects needed to complete the study.

The first interim analysis will be conducted after approximately 15 subjects in the 25- to 50-kg weight group have completed to Week 12. Pharmacokinetic, safety, and efficacy data on all subjects will be evaluated during this interim. The analysis will include all data available at this time – that is, it will include data from subjects in both weight groups who have enrolled at the time of the interim. The analysis of the data will be conducted by statisticians and PK/PD scientists external to the study team (statistical assessment center). The statistical assessment center will provide the analyses to a data monitoring committee (DMC) consisting of members external to Lilly. The DMC will recommend whether changes to weight-based dosing are necessary, based on the analysis. This committee will consist of 2 physicians external to Lilly, a pediatrician and a dermatologist, a statistician external to Lilly, and an nonvoting PK/PD member internal to Lilly, but external to the study team. No member of the DMC may have contact with study sites. Only the DMC is authorized to evaluate unblinded interim efficacy and safety analyses. Study sites will receive information about interim results ONLY if they need to know for the safety of their subjects.

Study sites will receive information about interim results ONLY if they need to know for the safety of their subjects.

The second interim database lock and unblinding will occur and the analysis will be performed at the time (that is, a cutoff date) the last subject completes Study Period 2 (Week 12) or ETV. This interim database lock will include all data collected by the cutoff date including follow-up data from subjects that have begun Periods 3, 4, or 5. Because the study will still be ongoing at the time of this database lock, the analysis will be referred to as an interim analysis. This interim analysis includes the final analysis for the Double-Blind Treatment Period (Period 2) of the study; therefore, there is no alpha adjustment due to this interim analysis. The DMC is not needed for this interim analysis.

Additional analyses and snapshots of study data may be performed during and/or after completion of Period 3 and/or Period 4 to fulfill the need for regulatory interactions or publication purposes.

Enrollment of each geographic region will be closely monitored. If 120 subjects from the United States and Canada complete the 12-week Double-Blind Randomized Period, and if other regions are behind in reaching their enrollment goal, an additional interim analysis may be conducted to include only the subjects from the United States and Canada to meet the US submission timeline. The DMC is not needed for this interim analysis. The analysis specified in this SAP for Period 2 will be conducted using the ITT Population and Safety Population subsetting on subjects from the United States and Canada and removing the term "region" from the analysis models. There will be no alpha adjustment applied as this will be considered the primary analysis for some regulatory agencies. The details will be documented in the unblinding plan.

A final database lock will occur after the Post-Treatment Follow-Up Period is completed.

## **6.18. Planned Exploratory Analyses**

The following analyses will be conducted for exploratory purposes and are not intended to be included in the CSR.

## 6.18.1. Psychometric Analyses of the Itch NRS

Following the examination of the distributional characteristics of measures, the following psychometric properties of the instruments will be evaluated: test-retest reliability; convergent validity; known-groups validity; and sensitivity to change (responsiveness) using anchor- and distribution-based methods.

## 6.18.1.1. Descriptive Statistics

Descriptive statistics (sample size, mean, standard deviation [SD], minimum, median, maximum, and % missing) will be calculated for the Itch NRS, including scores from Baseline to Week 12. The frequency distributions for Itch NRS responses will be calculated at Baseline and Week 12. Floor and ceiling effects will be evaluated at Baseline. A cut-off of >25% will be used to indicate floor/ceiling effects (McHorney et al. 1994).

#### 6.18.1.2. Test-Retest Reliability

Test-retest reliability has been emphasized by the Food and Drug Administration (FDA) as an important aspect of reliability in the FDA Patient-Reported outcome (PRO) Guidance (FDA 2009). Test-retest reliability reflects the ability of the instrument to give reproducible results when the clinical state is stable and indicates the degree to which a measure produces consistent results over several administrations. Test-retest reliability will be assessed using intra-class correlations coefficients (ICCs) and paired sample t-tests among stable patients only. The ICC will be used to assess the association between Itch NRS at Week 0 and Week 1 in the subsample of placebo arm patients with the same rating on the sPGA at Week 0 and Week 1.

Intra-class correlations coefficients range from 0 to 1.0, with higher scores indicating a more stable instrument. The hypothesis is that there will be no significant differences in scale scores when there is no change in disease status. An ICC of  $\geq$ 0.70 will be considered substantial agreement (Nunnally and Bernstein 1994).

## 6.18.1.3. Construct Validity

## 6.18.1.3.1. Convergent and Discriminant Validity

Construct validity is the degree to which a measure is related to other measures or constructed in a manner that is consistent with theory. *Convergent validity* involves demonstrating that different measures of the same concept substantially correlate, while *discriminant validity* demonstrates that concepts that are supposed to be unrelated are, in fact, unrelated.

Convergent validity will be assessed by Pearson correlations and Spearman rank-based correlation coefficient at baseline and at Week 12 between scores of the Itch NRS and other assessments, including PASI, sPGA, PatGA, DLQI (assessed in patients aged >16 years), and CDLQI (assessed in patients aged 6-16 years).

Cohen's conventions will be used to interpret the absolute value of the correlation results, where a correlation >0.5 is large, 0.3 to  $\le 0.5$  is moderate, 0.1 to < 0.3 is small, and < 0.1 is insubstantial (Cohen 1988). It is hypothesized that small-to-moderate correlations at baseline and moderate-to-large ( $\ge 0.30$ ) correlations at Week 12 are expected between the Itch NRS and PASI, sPGA, PatGA, and DLQI / CDLQI total scores.

Additionally, convergent and discriminant validity will be assessed by Pearson correlation and Spearman rank-based correlation at baseline and at Week 12 between scores of the Itch NRS and the DLQI / CDLQI 6 domains: Symptoms and Feelings, Daily Activities, Leisure, Work and School, Personal Relationships, and Treatment (note the CDLQI domains are Symptoms and Feelings, Sleep, Leisure, School or Holidays, Personal Relationships, and Treatment). It is hypothesized that the Itch NRS will correlate higher with the DLQI / CDLQI Symptoms and Feelings domain than with the other 5 DLQI domains.

## 6.18.1.3.2. Known-Groups Validity

Known-group validity is the extent to which scores from an instrument are different for groups of participants that differ on a relevant clinical or other indicator. Determining known-group validity involves evaluating an instrument in relation to clinical measures of disease status (Stewart et al. 1992; Hays and Revicki 2005). Known-groups validity of the Itch NRS will be evaluated using analysis of covariance to distinguish the Itch NRS scores between subgroups defined on the basis of sPGA score at baseline: sPGA score of 3; or combined 4 and 5. Patients with more severe plaques are hypothesized to report significantly greater itching severity.

## 6.18.1.4. Responsiveness

Responsiveness will be evaluated by correlating calculated changes from baseline in scores on the Itch NRS with changes in PASI, sPGA, and PatGA scores at 12 weeks. Moderate-to-large correlations are hypothesized based on Cohen's conventions. Additionally, responsiveness will be evaluated using 1-way ANCOVA, adjusted for Itch NRS baseline score, for overall and independent-sample t-tests for paired comparisons with Scheffe's correction-based post-hoc tests in distinguishing between subgroups, defined on the basis of the following:

1) PASI scores at Week 12: (1) PASI improved ≥75%; (2) PASI improved ≥50% to <75%; and (3) PASI got worse or improved <50%

- 2) sPGA scores at Week 12: sPGA score of 0 or 1 to those subjects with sPGA score >1
- 3) PatGA scores at Week 12: PatGA no change, improved, or worsened

It is hypothesized that an overall statistically significant difference will be observed (p<.05) with at least 1 statistically significant subgroup comparison (for example, PASI improved  $\geq$ 75% vs. PASI got worse or improved  $\leq$ 50%).

The above responsiveness analysis will be repeated using an ANOVA model (without Itch NRS baseline score) as a sensitivity analysis.

## 6.18.1.5. Clinical Significance (Minimal Within-Patient Change)

To aid in the interpretation of the Itch NRS results we will propose a range of thresholds that will contain minimal within-patient change (MWPC) in scores in the target patient population for FDA review. FDA is interested in what constitutes a meaningful within-patient change in scores from the *patient perspective*, i.e. individual patient level (FDA 2018). A number of analytic methods will be used to assess the MWPC of the Itch NRS. The results of these analyses can be used to guide score interpretation. Both anchor-based methods and distribution-based methods will be used for evaluating MWPC. However, anchor-based methods are preferred by the FDA for interpretation of PRO scores (FDA 2009), and will be considered the primary analysis. Distribution-based methods will be considered supportive and secondary (Revicki et al. 2008).

#### 6.18.1.5.1. Anchor-Based Method

The following analyses will be conducted to confirm the a priori defined Itch NRS ≥4-point reduction from baseline response criterion. The MWPC threshold for Itch NRS improvement will be derived by using the primary anchor variable of sPGA status at Week 12. As a secondary anchor, the PatGA will be used. The mean and median Itch NRS score improvement will be derived for patients meeting the anchor definitions for meaningful improvement.

The anchor-based analyses are as follows:

- 1) Determining the associations between sPGA and Itch NRS; and PatGA and Itch NRS. This will be assessed by Pearson and Spearman correlations at baseline and change from baseline to Week 12. Note these associations will be assessed in previously described convergent validity and responsiveness analyses.
- 2) Categorizing the primary anchor variable, the sPGA change (baseline to Week 12) as:
  - $\geq$ 2 point improvement and sPGA = 0,1
  - >2 point improvement and sPGA = 2.3
  - 1 point improvement
  - no change
  - ≥1 point worsening of sPGA
- 3) Categorizing the secondary anchor variable, the PatGA (baseline to Week 12) as:
  - ≥2 point improvement
  - 1 point improvement
  - no change
  - 1 point worsening

• ≥2 point worsening

If sample size in any above category <10 then it will be combined with adjacent category

#### 6.18.1.5.2. Distribution-Based Methods

Distribution-based methods will provide supportive evidence for the MWPC, secondary to the anchor-based methods..

#### 6.18.1.5.2.1. Standard Error of Measurement

Standard error of measurement has been proposed as a useful distribution-based statistic for evaluating clinically meaningful change in health-related quality of life (HRQL) measures (Wyrwich et al. 1999a; Wyrwich et al. 1999b). The SEM describes the error associated with the measure, and is estimated by the Baseline SD of the measure multiplied by the square root of 1 minus its reliability coefficient (ICC from the test-retest assessment). Previous research suggests that 1 SEM is roughly associated with a clinically important difference for PRO measures (Wyrwich et al. 1999a, Guyatt et al. 2002). Other research suggests changes (or differences) of 0.20 to 0.30 effect size may be indicative of a minimal important difference (Osoba and King 2005; Revicki et al. 2008).

An alternative distribution-based approach consists of calculating a 0.5 SD of the scales of interest at Baseline. It has been suggested that one-half of an SD of a measure represents a clinically meaningful change, while a change corresponding to 0.2 of an SD of measure is a small effect (Norman and Streiner 2003). The 0.5 SD estimate can be considered to provide an upper boundary for what would constitute a meaningful change, while 0.2 provides a lower boundary (Revicki et al. 2008). Given that a clinically important change is of interest, a 0.5 SD will be used, with a 0.2 SD calculated to provide reference for range.

The number and percentage of patients meeting the various RDs derived from anchor- and distribution-based methods for each measure will also be calculated.

Using the results from both the anchor- and distribution-based approaches, triangulation across possible thresholds indicating a minimal, but meaningful change will be considered.

#### 6.18.1.5.2.2. Empirical Cumulative Distribution Functions

As a complement to the confirmation of the MWPC, empirical cumulative distribution function (eCDF) curves will be calculated for the Itch NRS. The eCDF is a continuous (both positive and negative) presentation of the Itch NRS change from basline score at Week 12 on the X-axis and a cumulative proportion of patients with that level of score change on the Y-axis. The eCDF curve will be plotted for each anchor category. The meaningful-within patient threshold of the itch NRS should be considered by the eCDF of the anchor category where patients have experienced a meaningful improvement by definition of the anchor measure.

#### 6.18.1.5.2.3. Probability Density Functions

To aid in the interpretation of the eCDF analyses, probability density function (PDF) curves will be estimated using kernel density estimation of change in the Itch NRS to Week 12 by change in

anchor category. The PDF will present the same data as the eCDF but with probability density on the Y axis.

## 6.19. Clinical Trial Registry Analyses

Additional analyses will be performed for the purpose of fulfilling the Clinical Trial Registry (CTR) requirements.

Analyses provided for the CTR requirements include the following:

Summary of AEs, provided as a dataset which will be converted to an XML file. Both SAEs and "other" AEs are summarized by treatment group and by MedDRA PT.

- An AE is considered "serious" whether or not it is a TEAE.
- An AE is considered in the "other" category if it is both a TEAE and is not serious.
   For each SAE and "other" AE, for each term and treatment group, the following are provided:
  - o the number of participants at risk of an event
  - o the number of participants who experienced each event term
  - o the number of events experienced
- Consistent with www.ClinicalTrials.gov requirements, "other" AEs that occur in fewer than 5% of patients/subjects in every treatment group may not be included if a 5% threshold is chosen (5% is the minimum threshold).
- AE reporting is consistent with other document disclosures for example, the CSR, manuscripts, and so forth.

# 7. Unblinding Plan

Refer to a separate blinding and unblinding plan.

## 8. References

- Basra MK, Fenech R, Gatt RM, Salek MS, Finlay AY. The Dermatology Life Quality Index 1994-2007: a comprehensive review of validation data and clinical results. *Br J Dermatol*. 2008;159(5):997-1035.
- [CDC] Centers for Disease Control and Prevention resources page. National Center for Health Statistics. Data table of weight-for-age charts. Available at: http://www.cdc.gov/growthcharts/html\_charts/wtage.htm. Accessed October 20, 2016.
- Cohen, J. Statistical power analysis for the behavioral sciences (2nd ed.) Hillsdale, NJ: Erlbaum; 1988.
- Columbia University Medical Center. Columbia-Suicide Severity Rating Scale (C-SSRS) web site. Available at: http://www.cssrs.columbia.edu. Accessed January 13, 2016.
- DeVellis RF. Scale Development: Theory and Applications. Newbury Park, CA, USA: Sage, 1991.
- Diggle PJ, Liang KY, Zeger SL. Analysis of longitudinal data. Oxford: Clarendon Press; 1994.
- [EMA] European Medicines Agency. Committee for Medicinal Products for Human Use (CHMP). Guideline on clinical investigation of medicinal products indicated for the treatment of psoriasis. November 18, 2004; CHMP/EWP/2454/02 corr. Available at: http://www.ema.europa.eu/docs/en\_GB/document\_library/Scientific\_guideline/2009/09/WC50 0003329.pdf. Accessed October 19, 2016.
- [FDA] Food and Drug Administration. Guidance for industry patient-reported outcome measures: use in medical product development to support labeling claims. *Fed Regist*. 2009;74(235):65132-65133.
- [FDA] Food and Drug Administration. PATIENT-FOCUSED DRUG DEVELOPMENT GUIDANCE PUBLIC WORKSHOP: Methods to Identify What is Important to Patients & Select, Develop or Modify Fit-for-Purpose Clinical Outcomes Assessments. Workshop date: October 15-16 2018.
- Finlay AY, Khan GK. Dermatology Life Quality Index (DLQI)--a simple practical measure for routine clinical use. *Clin Exp Dermatol*. 1994;19(3):210-216.
- Fredriksson T, Pettersson U. Severe psoriasis--oral therapy with a new retinoid. *Dermatologica*. 1978;157(4):238-244.
- Gordon KB, Blauvelt A, Papp KA, Langley RG, Luger T, Ohtsuki M, Reich K, Amato D, Ball SG, Braun DK, Cameron GS, Erickson J, Konrad RJ, Muram TM, Nickoloff BJ, Osuntokun OO, Secrest RJ, Zhao F, Mallbris L, Leonardi CL; UNCOVER-1 Study Group; UNCOVER-2 Study Group; UNCOVER-3 Study Group. Phase 3 trials of ixekizumab in moderate-to-severe plaque psoriasis. *N Engl J Med.* 2016;375(4):345-356.
- Griffiths CE, Reich K, Lebwohl M, van de Kerkhof P, Paul C, Menter A, Cameron GS, Erickson J, Zhang L, Secrest RJ, Ball S, Braun DK, Osuntokun OO, Heffernan MP, Nickoloff BJ, Papp K; UNCOVER-2 and UNCOVER-3 investigators. Comparison of ixekizumab with etanercept or placebo in moderate-to-severe psoriasis (UNCOVER-2 and UNCOVER-3): results from two phase 3 randomised trials. *Lancet*. 2015;386(9993):541-551.

- Guyatt GH, Osoba D, Wu AW, et al. Methods to explain the clinical significance of health status measures. Paper presented at: Mayo Clinic Proceedings; 2002.
- Hays RD, Revicki D. Reliability and validity (including responsiveness). In: Fayers P, Hays RD, eds. Assessing Quality of Life in Clinical Trials: Methods and Practice. 2nd ed. New York, NY: Oxford University Press; 2005:25-39.
- Hongbo Y, Thomas CL, Harrison MA, Salek MS, Finlay AY. Translating the science of quality of life into practice: What do dermatology life quality index scores mean? *J Invest Dermatol*. 2005;125(4):659-664.
- Khilji FA, Gonzalez M, Finlay AY. Clinical meaning of change in Dermatology Life Quality Index scores. *Br J Dermatol*. 2002;147(suppl 62):50.
- Leonardi CL, Kimball AB, Papp KA, Yeilding N, Guzzo C, Wang Y, Li S, Dooley LT, Gordon KB; PHOENIX 1 study investigators. Efficacy and safety of ustekinumab, a human interleukin- 12/23 monoclonal antibody, in patients with psoriasis: 76-week results from a randomised, double-blind, placebo-controlled trial (PHOENIX 1). *Lancet*. 2008;371(9625):1665-1674. [Erratum appears in Lancet. 2008;371(9627):1838].
- Lewis-Jones MS, Finlay AY. The Children's Dermatology Life Quality Index (CDLQI): initial validation and practical use. *Br J Dermatol.* 1995;132(6):942-949.
- Mayes TL, Bernstein IH, Haley CL, Kennard BD, Emslie GJ. Psychometric properties of the Children's Depression Rating Scale-Revised in adolescents. *J Child Adolesc Psychopharmacol*. 2010;20(6):513-516.
- McHorney CA, Ware JE, Jr., Lu JF, Sherbourne CD. The MOS 36-item Short-Form Health Survey (SF-36): III. Tests of data quality, scaling assumptions, and reliability across diverse patient groups. *Medical care*. Jan 1994;32(1):40-66.
- [NIH] National Institutes of Health. The Fourth Report on The Diagnosis, Evaluation, and Treatment of High Blood Pressure in Children and Adolescents. Revised May 2005. Available at: https://www.nhlbi.nih.gov/files/docs/resources/heart/hbp\_ped.pdf. Accessed Mar 20, 2017.
- Norman GR, Streiner DL. *PDQ statistics*. Vol 1: PMPH-USA; 2003.
- Nunnally JC, Bernstein I. Psychometric theory. 3 ed. New York,: McGraw-Hill; 1994.
- Osoba D, King M. Meaningful differences. *Assessing quality of life in clinical trials*. 2005;2:243-257.
- Papp KA, Langley RG, Lebwohl M, Krueger GG, Szapary P, Yeilding N, Guzzo C, Hsu M-C, Wang Y, Li S, Dooley LT, Reich K. Efficacy and safety of ustekinumab, a human interleukin-12/23 monoclonal antibody, in patients with psoriasis: 52-week results from a randomised, double-blind, placebo-controlled trial (PHOENIX 2). *Lancet*. 2008;371(9625):1675-1684
- Poznanski EO, Mokros HB. Children's depression rating scale, revised (CDRS-R). Los Angeles: Western Psychological Services; 1996.
- Rasmussen AR, Wohlfahrt-Veje C, Tefre de Renzy-Martin K, Hagen CP, Tinggaard J, Mouritsen A, Mieritz MG, Main KM. Validity of self-assessment of pubertal maturation. *Pediatrics*. 2015;135(1):86-93.

- Revicki D, Hays RD, Cella D, Sloan J. Recommended methods for determining responsiveness and minimally important differences for patient-reported outcomes. *J. Clin. Epidemiol.* 2008;61(2):102-109.
- Salek MS, Jung S, Brincat-Ruffini LA, MacFarlane L, Lewis-Jones MS, Basra MK, Finlay AY. Clinical experience and psychometric properties of the Children's Dermatology Life Quality Index (CDLQI), 1995-2012. *Br J Dermatol*. 2013;169(4):734-759.
- Sampson HA, Munoz-Furlong A, Campbell RL, Adkinson NF Jr, Bock SA, Branum A, Brown SG, Camargo CA Jr, Cydulka R, Galli SJ, Gidudu J, Gruchalla RS, Harlor AD Jr, Hepner DL, Lewis LM, Lieberman PL, Metcalfe DD, O'Connor R, Muraro A, Rudman A, Schmitt C, Scherrer D, Simons FE, Thomas S, Wood JP, Decker WW. Second symposium on the definition and management of anaphylaxis: Summary report-Second National Institute of Allergy and Infectious Disease/Food Allergy and Anaphylaxis Network symposium. J Allergy Clin Immunol. 2006;117(2):391–397.
- Schisterman EF, Perkins NJ, Liu A, Bondell H. Optimal cut-point and its corresponding Youden Index to discriminate individuals using pooled blood samples. *Epidemiology*. 2005;16(1):73-81.
- Stewart A, Hays R, Ware J. Methods of validating MOS health measures. In: Stewart A, Ware J, eds. Measuring Functioning and Well-being: The Medical Outcomes Study Approach. Durham, NC: Duke University Press; 1992:25-39.
- Van Voorhees A, Feldman SR, Koo JYM, Lebwohl MG, Menter A. The psoriasis and psoriatic arthritis pocket guide. National Psoriasis Foundation. 2009. Available at: https://www.psoriasis.org/sites/default/files/accessing-health-care/FY10 Pocket Guide WEB.pdf. Accessed November 18, 2016.
- Waters A, Sandhu D, Beattie P, Ezughah F, Lewis-Jones S. Severity stratification of Children's Dermatology Life Quality Index (CDLQI) scores [abstract]. *Br J Dermatol*. 2010;163(Suppl 1):121.
- Wyrwich KW, Nienaber NA, Tierney WM, Wolinksy FD. Linking clinical relevance and statistical significance in evaluating intra-individual changes in health-related quality of life. *Med Care.* 1999a;37(5):469-478.
- Wyrwich KW, Tierney WM, Wolinsky FD. Further evidence supporting an SEM-based criterion for identifying meaningful intra-individual changes in health-related quality of life. *J Clin Epidemiol*. 1999b;52(9):861-873.

# 9. Appendices

# **Appendix 1. Concomitant Topical Therapy Definition**

This appendix provides the instruction to derive flags for patients who took concomitant topical therapy or concomitant topical steroid therapy for ixekizumab psoriasis and psoriatic arthritis studies.

- **Concomitant Topical Therapy** defined as patients who took concomitant medications which met all the following conditions:
  - 1) Route = topical
  - 2) Indication for use = primary study condition
  - 3) ATC codes (defined in the table below):
    D07-- (level 2, include all sub-levels), A11CC, D05AC, D05BB, L04AD, D02AF, D05AA,
    D02A- (Level 3, include all sub-levels), D05AX, V90
    - 20211 (20 voi 3, moidad an suo io vois), 202111, 170
- **Concomitant Topical Steroid Therapy** defined as patients who took concomitant medications which met all the following conditions:
  - 1) Route = topical
  - 2) Indication for use = primary study condition
  - 3) ATC code: D07-- (level 2, include all sub-levels)

Reference Table: List of Topical Treatments that are Prescribed/Administered for Psoriasis or Psoriatic Arthritis Patients with Appropriate ATC Code

| Topical Treatments | ATC Code |
|---|---|
| <b>Topical corticosteroids:</b> These powerful anti-inflammatory drugs are the most frequently prescribed | D07 |
| medications for treating mild-to-moderate psoriasis. They slow cell turnover by suppressing the | (Level 2) |
| immune system, which reduces inflammation and relieves associated itching. Topical corticosteroids | |
| range in strength from mild to very strong. Low-potency corticosteroid ointments are usually | |
| recommended for sensitive areas, such as your face or skinfolds, and for treating widespread patches | |
| of damaged skin. Your doctor may prescribe stronger corticosteroid ointment for small areas of your | |
| skin, for persistent plaques on your hands or feet, or when other treatments have failed. Medicated | |
| foams and scalp solutions are available to treat psoriasis patches on the scalp. Long-term use or | |
| overuse of strong corticosteroids can cause thinning of the skin and resistance to the treatment's | |
| benefits. To minimize side effects and to increase effectiveness, topical corticosteroids are generally | |
| used on active outbreaks until they are under control. | |
| Vitamin D analogs: These synthetic forms of vitamin D slow down the growth of skin cells. | A11CC |
| Calcipotriene (Dovonex) is a prescription cream or solution containing a vitamin D analog that may | |
| be used alone to treat mild-to-moderate psoriasis or in combination with other topical medications or | |
| phototherapy. This treatment can irritate the skin. Calcitriol (Rocaltrol) is expensive, but may be | |
| equally effective and possibly less irritating than calcipotriene. | |
| Anthralin: This medication is believed to normalize DNA activity in skin cells. Anthralin (Dritho- | D05AC |
| Scalp) can also remove scale, making the skin smoother. However, anthralin can irritate skin, and it | |
| stains virtually anything it touches, including skin, clothing, countertops, and bedding. For that | |
| reason, doctors often recommend short-contact treatment – allowing the cream to stay on your skin for | |
| a brief time before washing it off. Anthralin is sometimes used in combination with ultraviolet light. | |
| <b>Topical retinoids:</b> These are commonly used to treat acne and sun-damaged skin, but tazarotene | D05BB |
| (Tazorac, Avage) was developed specifically for the treatment of psoriasis. Like other vitamin A | Boobb |
| derivatives, it normalizes DNA activity in skin cells and may decrease inflammation. The most | |
| common side effect is skin irritation. It may also increase sensitivity to sunlight, so sunscreen should | |
| be applied while using the medication. Although the risk of birth defects is far lower for topical | |
| retinoids than for oral retinoids, your doctor needs to know if you are pregnant or intend to become | |
| pregnant if you are using tazarotene. | |
| Calcineurin inhibitors: Currently, calcineurin inhibitors – tacrolimus (Prograf) and pimecrolimus | L04AD |
| (Elidel) – are approved only for the treatment of atopic dermatitis, but studies have shown them to be | E o m E |
| effective, at times, in the treatment of psoriasis. Calcineurin inhibitors are thought to disrupt the | |
| activation of T cells, which in turn reduces inflammation and plaque buildup. The most common side | |
| effect is skin irritation. Calcineurin inhibitors are not recommended for long-term or continuous use | |
| because of a potential increased risk of skin cancer and lymphoma. Calcineurin inhibitors are used | |
| only with your doctor's input and approval. They may be especially helpful in areas of thin skin, such | |
| as around the eyes, where steroid creams or retinoids are too irritating or may cause harmful effects. | |
| Salicylic acid: Available over-the-counter (nonprescription) and by prescription, salicylic acid | D02AF |
| promotes sloughing of dead skin cells, and reduces scaling. Sometimes it is combined with other | DOZAI |
| medications, such as topical corticosteroids or coal tar, to increase its effectiveness. Salicylic acid is | |
| available in medicated shampoos and scalp solutions to treat scalp psoriasis. | |
| Coal tar: A thick, black byproduct of the manufacture of petroleum products and coal, coal tar is | D05AA |
| probably the oldest treatment for psoriasis. It reduces scaling, itching, and inflammation. Exactly | DUJAA |
| how it works is not known. Coal tar has few known side effects, but it is messy, stains clothing and | |
| bedding, and has a strong odor. Coal tar is available in over-the-counter shampoos, creams, and oils. | |
| It is also available in higher concentrations by prescription. | |
| it is also available in higher concentrations by prescription. | ] |

| Topical Treatments | ATC Code |
|---|---|
| <b>Moisturizers:</b> By themselves, moisturizing creams will not heal psoriasis, but they can reduce itching and scaling and can help combat the dryness that results from other therapies. Moisturizers in an ointment base are usually more effective than are lighter creams and lotions. | D02A-<br>(Level 3) |
| Calcipotriene | D05AX |
| Tazarotene | D05AX |
| Herbal and traditional preparations | V90 |

Note: ATC = WHOCC Anatomical Therapeutic Chemical classification system; WHOCC = World Health Organization Collaborating Centre for Drug Statistics Methodology.
## Appendix 2. Anti-infective Treatments and Anatomical Therapeutic Chemical (ATC) Code List

| ATC | ATC | |
|---|---|---|
| Code | Level | ATC Description (Based on ATC Dictionary 18JAN2016) |
| A01AB | 4 | ANTIINFECTIVES AND ANTISEPTICS FOR LOCAL ORAL TREA |
| A02BD | 4 | COMBINATIONS FOR ERADICATION OF HELICOBACTER PYLOR |
| A07A | 3 | INTESTINAL ANTIINFECTIVES |
| A07AA | 4 | ANTIBIOTICS |
| A07AB | 4 | SULFONAMIDES |
| A07AC | 4 | IMIDAZOLE DERIVATIVES |
| A07AX | 4 | OTHER INTESTINAL ANTIINFECTIVES |
| B05CA | 4 | ANTIINFECTIVES |
| C05AB | 4 | ANTIBIOTICS |
| D01 | 2 | ANTIFUNGALS FOR DERMATOLOGICAL USE |
| D01A | 3 | ANTIFUNGALS FOR TOPICAL USE |
| D01AA | 4 | ANTIBIOTICS |
| D01AC | 4 | IMIDAZOLE AND TRIAZOLE DERIVATIVES |
| D01AE | 4 | OTHER ANTIFUNGALS FOR TOPICAL USE |
| D01B | 3 | ANTIFUNGALS FOR SYSTEMIC USE |
| D01BA | 4 | ANTIFUNGALS FOR SYSTEMIC USE |
| D06 | 2 | ANTIBIOTICS AND CHEMOTHERAPEUTICS FOR DERMATOLOGIC |
| D06A | 3 | ANTIBIOTICS FOR TOPICAL USE |
| D06AA | 4 | TETRACYCLINE AND DERIVATIVES |
| D06AX | 4 | OTHER ANTIBIOTICS FOR TOPICAL USE |
| D06B | 3 | CHEMOTHERAPEUTICS FOR TOPICAL USE |
| D06BA | 4 | SULFONAMIDES |
| D06BB | 4 | ANTIVIRALS |
| D06BX | 4 | OTHER CHEMOTHERAPEUTICS |
| D06C | 3 | ANTIBIOTICS AND CHEMOTHERAPEUTICS, COMBINATIONS |
| D07C | 3 | CORTICOSTEROIDS, COMBINATIONS WITH ANTIBIOTICS |
| D07CA | 4 | CORTICOSTEROIDS, WEAK, COMBINATIONS WITH ANTIBIOTICS |
| | | CORTICOSTEROIDS, MODERATELY POTENT, COMBINATIONS WITH |
| D07CB | 4 | ANTIBIOTICS |
| D07CC | 4 | CORTICOSTEROIDS, POTENT, COMBINATIONS WITH ANTIBIOTICS |
| D07CD | 4 | CORTICOSTEROIDS, VERY POTENT, COMBINATIONS WITH ANTIBIOTICS |
| D09AA | 4 | MEDICATED DRESSINGS WITH ANTIINFECTIVES |
| D10AF | 4 | ANTIINFECTIVES FOR TREATMENT OF ACNE |
| G01AA | 4 | ANTIBIOTICS |
| G01AC | 4 | QUINOLINE DERIVATIVES |
| G01AE | 4 | SULFONAMIDES |
| G01AF | 4 | IMIDAZOLE DERIVATIVES |
| G01AG | 4 | TRIAZOLE DERIVATIVES |
| G01AX | 4 | OTHER ANTIINFECTIVES AND ANTISEPTICS |
| G01BA | 4 | ANTIBIOTICS AND CORTICOSTEROIDS |

| ATC<br>Code | ATC<br>Level | ATC Description (Based on ATC Dictionary 18JAN2016) |
|---|---|---|
| G01BC | 4 | QUINOLINE DERIVATIVES AND CORTICOSTEROIDS |
| G01BE | 4 | SULFONAMIDES AND CORTICOSTEROIDS |
| G01BF | 4 | IMIDAZOLE DERIVATIVES AND CORTICOSTEROIDS |
| G04AB | 4 | QUINOLONE DERIVATIVES (EXCL. J01M) |
| G04AC | 4 | NITROFURAN DERIVATIVES |
| G04AG | 4 | OTHER URINARY ANTISEPTICS AND ANTIINFECT |
| G04AH | 4 | SULFONAMIDES IN COMBINATION WITH OTHER DRUGS |
| G04AK | 4 | URINARY ANTISEPT&ANTIINF, COMB EXCL SULFONAMIDES |
| J01 | 2 | ANTIBACTERIALS FOR SYSTEMIC USE |
| J01A | 3 | TETRACYCLINES |
| J01AA | 4 | TETRACYCLINES |
| J01B | 3 | AMPHENICOLS |
| J01BA | 4 | AMPHENICOLS |
| J01C | 3 | BETA-LACTAM ANTIBACTERIALS, PENICILLINS |
| J01CA | 4 | PENICILLINS WITH EXTENDED SPECTRUM |
| J01CE | 4 | BETA-LACTAMASE SENSITIVE PENICILLINS |
| J01CF | 4 | BETA-LACTAMASE RESISTANT PENICILLINS |
| J01CG | 4 | BETA-LACTAMASE INHIBITORS |
| J01CR | 4 | COMBINATIONS OF PENICILLINS, INCL. BETA-LACTAMASE |
| J01D | 3 | OTHER BETA-LACTAM ANTIBACTERIALS |
| J01DA | 4 | CEPHALOSPORINS AND RELATED SUBSTANCES |
| J01DB | 4 | FIRST-GENERATION CEPHALOSPORINS |
| J01DC | 4 | SECOND-GENERATION CEPHALOSPORINS |
| J01DD | 4 | THIRD-GENERATION CEPHALOSPORINS |
| J01DE | 4 | FOURTH-GENERATION CEPHALOSPORINS |
| J01DF | 4 | MONOBACTAMS |
| J01DH | 4 | CARBAPENEMS |
| J01DI | 4 | OTHER CEPHALOSPORINS |
| J01E | 3 | SULFONAMIDES AND TRIMETHOPRIM |
| J01EA | 4 | TRIMETHOPRIM AND DERIVATIVES |
| J01EB | 4 | SHORT-ACTING SULFONAMIDES |
| J01EC | 4 | INTERMEDIATE-ACTING SULFONAMIDES |
| J01ED | 4 | LONG-ACTING SULFONAMIDES |
| J01EE | 4 | COMBINATIONS OF SULFONAMIDES AND TRIMETHOPRIM, INC |
| J01F | 3 | MACROLIDES, LINCOSAMIDES AND STREPTOGRAMINS |
| J01FA | 4 | MACROLIDES |
| J01FF | 4 | LINCOSAMIDES |
| J01FG | 4 | STREPTOGRAMINS |
| J01G | 3 | AMINOGLYCOSIDE ANTIBACTERIALS |
| J01GA | 4 | STREPTOMYCINS |
| J01GB | 4 | OTHER AMINOGLYCOSIDES |
| J01M | 3 | QUINOLONE ANTIBACTERIALS |
| J01MA | 4 | FLUOROQUINOLONES |
| J01MB | 4 | OTHER QUINOLONES |
| J01R | 3 | COMBINATIONS OF ANTIBACTERIALS |
| J01RA | 4 | COMBINATIONS OF ANTIBACTERIALS |

| ATC<br>Code | ATC<br>Level | ATC Description (Based on ATC Dictionary 18JAN2016) |
|---|---|---|
| J01WA | 4 | HERBAL ANTIBACTERIALS FOR SYSTEMIC USE |
| J01WB | 4 | HERBAL URINARY ANTISEPTICS AND ANTIINFECTIVES |
| J01X | 3 | OTHER ANTIBACTERIALS |
| J01XA | 4 | GLYCOPEPTIDE ANTIBACTERIALS |
| J01XB | 4 | POLYMYXINS |
| J01XC | 4 | STEROID ANTIBACTERIALS |
| J01XD | 4 | IMIDAZOLE DERIVATIVES |
| J01XE | 4 | NITROFURAN DERIVATIVES |
| J01XX | 4 | OTHER ANTIBACTERIALS |
| J02 | 2 | ANTIMYCOTICS FOR SYSTEMIC USE |
| J02A | 3 | ANTIMYCOTICS FOR SYSTEMIC USE |
| J02AA | 4 | ANTIBIOTICS |
| J02AB | 4 | IMIDAZOLE DERIVATIVES |
| J02AC | 4 | TRIAZOLE DERIVATIVES |
| J02AX | 4 | OTHER ANTIMYCOTICS FOR SYSTEMIC USE |
| J04AA | 4 | AMINOSALICYLIC ACID AND DERIVATIVES |
| J04AB | 4 | ANTIBIOTICS |
| J04AC | 4 | HYDRAZIDES |
| J04AK | 4 | OTHER DRUGS FOR TREATMENT OF TUBERCULOSIS |
| J04AM | 4 | COMBINATIONS OF DRUGS FOR TREATMENT OF TUBERCULOSI |
| J04B | 3 | DRUGS FOR TREATMENT OF LEPRA |
| J04BA | 4 | DRUGS FOR TREATMENT OF LEPRA |
| J05 | 2 | ANTIVIRALS FOR SYSTEMIC USE |
| J05A | 3 | DIRECT ACTING ANTIVIRALS |
| J05AA | 4 | THIOSEMICARBAZONES |
| J05AB | 4 | NUCLEOSIDES AND NUCLEOTIDES EXCL. REVERSE TRANSCRI |
| J05AC | 4 | CYCLIC AMINES |
| J05AD | 4 | PHOSPHONIC ACID DERIVATIVES |
| J05AE | 4 | PROTEASE INHIBITORS |
| J05AF | 4 | NUCLEOSIDE AND NUCLEOTIDE REVERSE TRANSCRIPTASE IN |
| J05AG | 4 | NON-NUCLEOSIDE REVERSE TRANSCRIPTASE INHIBITORS |
| J05AH | 4 | NEURAMINIDASE INHIBITORS |
| J05AR | 4 | ANTIVIRALS FOR TREATMENT OF HIV INFECTIONS, COMBIN |
| J05AX | 4 | OTHER ANTIVIRALS |
| P01A | 3 | AGENTS AGAINST AMOEBIASIS AND OTHER PROTOZOAL DISE |
| P01AA | 4 | HYDROXYQUINOLINE DERIVATIVES |
| P01AB | 4 | NITROIMIDAZOLE DERIVATIVES |
| P01AC | 4 | DICHLOROACETAMIDE DERIVATIVES |
| P01AR | 4 | ARSENIC COMPOUNDS |
| P01AX | 4 | OTHER AGENTS AGAINST AMOEBIASIS AND OTHER PROTOZOA |
| P01BA | 4 | AMINOQUINOLINES |
| P01BC | 4 | METHANOLQUINOLINES |
| P01BD | 4 | DIAMINOPYRIMIDINES |
| P01BE | 4 | ARTEMISININ AND DERIVATIVES, PLAIN |
| P01BF | 4 | ARTEMISININ AND DERIVATIVES, COMBINATIONS |
| P01BX | 4 | OTHER ANTIMALARIALS |

| ATC<br>Code | ATC<br>Level | ATC Description (Based on ATC Dictionary 18JAN2016) |
|---|---|---|
| P01C | 3 | AGENTS AGAINST LEISHMANIASIS AND TRYPANOSOMIASIS |
| P01CA | 4 | NITROIMIDAZOLE DERIVATIVES |
| P01CB | 4 | ANTIMONY COMPOUNDS |
| P01CC | 4 | NITROFURAN DERIVATIVES |
| P01CD | 4 | ARSENIC COMPOUNDS |
| P01CX | 4 | OTHER AGENTS AGAINST LEISHMANIASIS AND TRYPANOSOMI |
| P02 | 2 | ANTHELMINTICS |
| P02B | 3 | ANTITREMATODALS |
| P02BA | 4 | QUINOLINE DERIVATIVES AND RELATED SUBSTANCES |
| P02BB | 4 | ORGANOPHOSPHOROUS COMPOUNDS |
| P02BX | 4 | OTHER ANTITREMATODAL AGENTS |
| P02C | 3 | ANTINEMATODAL AGENTS |
| P02CA | 4 | BENZIMIDAZOLE DERIVATIVES |
| P02CB | 4 | PIPERAZINE AND DERIVATIVES |
| P02CC | 4 | TETRAHYDROPYRIMIDINE DERIVATIVES |
| P02CE | 4 | IMIDAZOTHIAZOLE DERIVATIVES |
| P02CF | 4 | AVERMECTINES |
| P02CX | 4 | OTHER ANTINEMATODALS |
| P02D | 3 | ANTICESTODALS |
| P02DA | 4 | SALICYLIC ACID DERIVATIVES |
| P02DW | 4 | HERBAL ANTICESTODALS |
| P02DX | 4 | OTHER ANTICESTODALS |
| P02WA | 4 | HERBAL ANTHELMINTICS |
| P03A | 3 | CTOPARASITICIDES, INCL. SCABICIDES |
| P03AA | 4 | SULFUR CONTAINING PRODUCTS |
| P03AB | 4 | CHLORINE CONTAINING PRODUCTS |
| P03AC | 4 | PYRETHRINES, INCL. SYNTHETIC COMPOUNDS |
| P03AX | 4 | OTHER ECTOPARASITICIDES, INCL. SCABICIDES |
| P03BA | 4 | PYRETHRINES |
| R02AB | 4 | ANTIBIOTICS |
| S01A | 3 | ANTIINFECTIVES |
| S01AA | 4 | ANTIBIOTICS |
| S01AB | 4 | SULFONAMIDES |
| S01AD | 4 | ANTIVIRALS |
| S01AE | 4 | FLUOROQUINOLONES |
| S01AX | 4 | OTHER ANTIINFECTIVES |
| S01C | 3 | ANTIINFLAMMATORY AGENTS AND ANTIINFECTIVES IN COMB |
| S01CA | 4 | CORTICOSTEROIDS AND ANTIINFECTIVES IN COMBINATION |
| S01CB | 4 | CORTICOSTEROIDS/ANTIINFECTIVES/MYDRIATICS IN COMBI |
| S01CB<br>S01CC | 4 | ANTIINFLAMMATORY AGENTS, NON-STEROIDS AND ANTIINFECTIVES |
| S02A | 3 | ANTIINFEAMMATORY AGENTS, NON-STEROIDS AND ANTIINFECTIVES ANTIINFECTIVES |
| S02A<br>S02AA | 4 | ANTIINFECTIVES ANTIINFECTIVES |
| | 3 | |
| S02C | | CORTICOSTEROIDS AND ANTIINFECTIVES IN COMBINATION |
| S02CA | 3 | CORTICOSTEROIDS AND ANTIINFECTIVES IN COMBINATION |
| S03A | | ANTIINFECTIVES |
| S03AA | 4 | ANTIINFECTIVES |

| ATC | ATC | |
|-------|-------|-----------------------------------------------------|
| Code | Level | ATC Description (Based on ATC Dictionary 18JAN2016) |
| S03C | 3 | CORTICOSTEROIDS AND ANTIINFECTIVES IN COMBINATION |
| S03CA | 4 | CORTICOSTEROIDS AND ANTIINFECTIVES IN COMBINATION |

Abbreviation: ATC = WHOCC Anatomical Therapeutic Chemical classification system; INCL. = including; WHOCC = World Health Organization Collaborating Centre for Drug Statistics Methodology.

# Appendix 3. Lilly-Defined MedDRA V21.0 Preferred Terms for Opportunistic Infections (OIs)

| Opportunistic Infection | Preferred Term<br>(MedDRA Version 21.0) | Lilly Defined<br>Classification |
|---|---|---|
| Pneumocystis jirovecii (II) | Pneumocystis jirovecii infection | Narrow |
| 1 neumocystis fil ovecti (11) | Pneumocystis jirovecii pneumonia | Tullow |
| | Blood beta-D-glucan | Broad |
| | Blood beta-D-glucan abnormal | 21044 |
| | Blood beta-D-glucan increased | |
| | Gomori methenamine silver stain | |
| | Carbon monoxide diffusing capacity | |
| | decreased | |
| | Carbon monoxide diffusing capacity | |
| | Pneumocystis test positive | |
| Human Polyomavirus Infection | BK virus infection | Narrow |
| including BK virus disease and | Human polyomavirus infection | |
| PVAN (V), and Progressive | JC virus granule cell neuronopathy | |
| Multifocal Leukoencephalopathy | JC virus infection | |
| (IV) | Polyomavirus-associated nephropathy | |
| | Progressive multifocal leukoencephalopathy | |
| | Anti-JC virus antibody index | Broad |
| | JC polyomavirus test | |
| | JC virus test | |
| | JC virus test positive | |
| | Polyomavirus test | |
| | Polyomavirus test positive | |
| Cytomegalovirus disease (V) | Cytomegalovirus chorioretinitis | Narrow |
| | Cytomegalovirus colitis | |
| | Cytomegalovirus duodenitis | |
| | Cytomegalovirus enteritis | |
| | Cytomegalovirus enterocolitis | |
| | Cytomegalovirus gastritis | |
| | Cytomegalovirus gastroenteritis | |
| | Cytomegalovirus gastrointestinal infection | |
| | Cytomegalovirus gastrointestinal ulcer | |
| | Cytomegalovirus hepatitis | |
| | Cytomegalovirus infection | |
| | Cytomegalovirus mononucleosis | |
| | Cytomegalovirus mucocutaneous ulcer | |
| | Cytomegalovirus myelomeningoradiculitis | |
| | Cytomegalovirus acceptagitis | |
| | Cytomegalovirus penersetitis | |
| | Cytomegalovirus parceatitis | |
| | Cytomegalovirus pericarditis | |

| Opportunistic Infection | Preferred Term (MedDRA Version 21.0) | Lilly Defined<br>Classification |
|---|---|---|
| | Cytomegalovirus syndrome | |
| | Cytomegalovirus urinary tract infection | |
| | Cytomegalovirus viraemia | |
| | Disseminated cytomegaloviral infection | |
| | Encephalitis cytomegalovirus | |
| | Pneumonia cytomegaloviral | |
| | Cytomegalovirus test | Broad |
| | Cytomegalovirus test positive | |
| Post-transplant lymphoproliferative | Epstein-Barr virus associated lymphoma | Narrow |
| disorder (EBV) (V) | Epstein-Barr virus associated | |
| | lymphoproliferative disorder | |
| | Epstein Barr virus positive mucocutaneous | |
| | ulcer | |
| | Post transplant lymphoproliferative disorder | |
| | Epstein-Barr viraemia | Broad |
| | Epstein-Barr virus infection | |
| | Lymphoproliferative disorder | |
| | Lymphoproliferative disorder in remission | |
| | Oral hairy leukoplakia | |
| Bartonellosis (disseminated disease | Bacillary angiomatosis | Narrow |
| only) (V) | Peliosis hepatis | 1 (4110 )) |
| | Splenic peliosis | |
| | Systemic bartonellosis | |
| | Trench fever | |
| | Bartonella test | Broad |
| | Bartonella test positive | Dioau |
| | Bartonellosis | |
| | Cat scratch disease | |
| Dit(IV) | | N |
| Blastomycosis (IV) | Blastomycosis | Narrow |
| | Epididymitis blastomyces | |
| | Osteomyelitis blastomyces | |
| | Pneumonia blastomyces | D 1 |
| | NA | Broad |
| Toxoplasmosis (myocarditis, | Cerebral toxoplasmosis | Narrow |
| pneumonitis, or characteristic | Eye infection toxoplasmal | |
| retinochoroiditis only) (IV) | Hepatitis toxoplasmal | |
| | Meningitis toxoplasmal | |
| | Myocarditis toxoplasmal | |
| | Pneumonia toxoplasmal | |
| | Toxoplasma serology | Broad |
| | Toxoplasma serology positive | |
| | Toxoplasmosis | |
| Coccidioidomycosis (II) | Coccidioides encephalitis | Narrow |
| J ( -) | Coccidioidomycosis | |
| | Cutaneous coccidioidomycosis | |
| | Camillous coccidioidoiliycosis | <u> </u> |

| Opportunistic Infection | Preferred Term<br>(MedDRA Version 21.0) | Lilly Defined<br>Classification |
|---|---|---|
| | Meningitis coccidioides | |
| | NA | Broad |
| Histoplasmosis (II) | Acute pulmonary histoplasmosis | Narrow |
| 1 ( ) | Chronic pulmonary histoplasmosis | |
| | Endocarditis histoplasma | |
| | Histoplasmosis | |
| | Histoplasmosis cutaneous | |
| | Histoplasmosis disseminated | |
| | Meningitis histoplasma | |
| | Pericarditis histoplasma | |
| | Retinitis histoplasma | |
| | Presumed ocular histoplasmosis syndrome | Broad |
| Aspergillosis (invasive disease only) | Aspergillosis oral | Narrow |
| (II) | Cerebral aspergillosis | |
| | Meningitis aspergillus | |
| | Oro-pharyngeal aspergillosis | |
| | Aspergillus infection | Broad |
| | Aspergillus test | |
| | Aspergillus test positive | |
| | Bronchopulmonary aspergillosis | |
| | Sinusitis aspergillus | |
| Candidiasis (invasive disease or | Candida endophthalmitis | Narrow |
| oral) (II) | Candida osteomyelitis | |
| | Candida pneumonia | |
| | Candida retinitis | |
| | Candida sepsis | |
| | Cerebral candidiasis | |
| | Endocarditis candida | |
| | Fungal oesophagitis | |
| | Gastrointestinal candidiasis | |
| | Hepatic candidiasis | |
| | Hepatosplenic candidiasis | |
| | Meningitis candida | |
| | Oesophageal candidiasis | |
| | Oropharyngeal candidiasis | |
| | Peritoneal candidiasis | |
| | Splenic candidiasis | |
| | Systemic candida | D 1 |
| | Bladder candidiasis | Broad |
| | Candida infection | |
| | Candida test | |
| | Candida test positive | |
| | Mucocutaneous candidiasis Oral candidiasis | |
| | Oral fungal infection | |
| | Respiratory moniliasis | |

| | Preferred Term | Lilly Defined |
|---|---|---|
| Opportunistic Infection | (MedDRA Version 21.0) | Classification |
| Cryptococcosis (II) | Cryptococcal cutaneous infection | Narrow |
| - JF ( ) | Cryptococcal fungaemia | |
| | Cryptococcosis | |
| | Disseminated cryptococcosis | |
| | Gastroenteritis cryptococcal | |
| | Meningitis cryptococcal | |
| | Neurocryptococcosis | |
| | Osseous cryptococcosis | |
| | Pneumonia cryptococcal | |
| | Cryptococcus test | Broad |
| | Cryptococcus test positive | |
| Other invasive fungi: Mucormycosis | Allescheriosis | Narrow |
| (zygomycosis), Rhizopus, Mucor, | Fusarium infection | |
| and Lichtheimia, Scedosporum/ | Mucormycosis | |
| Pseudallescheria boydii, Fusarium | Scedosporium infection | |
| (II) | Phaeohyphomycosis | |
| | Phaeohyphomycotic brain abscess | |
| | Pseudallescheria infection | |
| | Pseudallescheria sepsis | |
| | See "Non-specific terms" below | Broad |
| Legionellosis (II) | Legionella infection Pneumonia legionella | Narrow |
| | Pontiac fever | |
| | Legionella test | Broad |
| | Legionella test positive | |
| Listeria monocytogenes (invasive | Listeria encephalitis | Narrow |
| disease only) (II) | Listeria sepsis | |
| 3, ( ) | Meningitis listeria | |
| | Listeria test | Broad |
| | Listeria test positive | |
| | Listeraemia | |
| | Listeriosis | |
| Tuberculosis (I) | Adrenal gland tuberculosis | Narrow |
| | Bone tuberculosis | |
| | Choroid tubercles | |
| | Conjunctivitis tuberculous | |
| | Cutaneous tuberculosis | |
| | Disseminated Bacillus Calmette-Guerin | |
| | infection | |
| | Disseminated tuberculosis | |
| | Ear tuberculosis | |
| | Epididymitis tuberculous | |

| Opportunistic Infection | Preferred Term<br>(MedDRA Version 21.0) | Lilly Defined<br>Classification |
|---|---|---|
| | Extrapulmonary tuberculosis | |
| | Immune reconstitution inflammatory | |
| | syndrome associated tuberculosis | |
| | Intestinal tuberculosis | |
| | Joint tuberculosis | |
| | Lymph node tuberculosis | |
| | Male genital tract tuberculosis | |
| | Meningitis tuberculous | |
| | Oesophageal tuberculosis | |
| | Oral tuberculosis | |
| | Pericarditis tuberculous | |
| | Peritoneal tuberculosis | |
| | Prostatitis tuberculous | |
| | Pulmonary tuberculoma | |
| | Pulmonary tuberculosis | |
| | Renal tuberculosis | |
| | Salpingitis tuberculous | |
| | Silico tuberculosis | |
| | Spleen tuberculosis | |
| | Thyroid tuberculosis | |
| | Tuberculid | |
| | Tuberculoma of central nervous system | |
| | Tuberculosis | |
| | Tuberculosis bladder | |
| | Tuberculosis gastrointestinal | |
| | Tuberculosis liver | |
| | Tuberculosis of central nervous system | |
| | Tuberculosis of eye | |
| | Tuberculosis of genitourinary system | |
| | Tuberculosis of intrathoracic lymph nodes | |
| | Tuberculosis of peripheral lymph nodes | |
| | Tuberculosis or peripheral lymph hodes Tuberculosis ureter | |
| | Tuberculous abscess central nervous system | |
| | Tuberculous endometritis | |
| | Tuberculous laryngitis | |
| | Tuberculous pleurisy | |
| | <del>-</del> _ <del>-</del> | |
| | Tuberculous tenosynovitis | Drand |
| | Interferon gamma release assay | Broad |
| | Interferon gamma release assay positive | |
| | Mycobacterium tuberculosis complex test | |
| | Mycobacterium tuberculosis complex test | |
| | positive | |
| | Tuberculin test | |
| | Tuberculin test false negative | |
| | Tuberculin test positive | |
| Nocardiosis (II) | Cutaneous nocardiosis | Narrow |

| | Preferred Term | Lilly Defined |
|---|---|---|
| Opportunistic Infection | (MedDRA Version 21.0) | Lilly Defined<br>Classification |
| Opportunistic infection | Nocardia sepsis | Classification |
| | Nocardiosis | |
| | Pulmonary nocardiosis | |
| | Nocardia test positive | Broad |
| Nontuberculous Mycobacterium | Atypical mycobacterial infection | Narrow |
| disease (II) | Atypical mycobacterial infection Atypical mycobacterial lower respiratory tract | Ivaliow |
| disease (11) | infection | |
| | Atypical mycobacterial lymphadenitis | |
| | Atypical mycobacterial pneumonia | |
| | Atypical mycobacterium pericarditis | |
| | Borderline leprosy | |
| | Bovine tuberculosis | |
| | Indeterminate leprosy | |
| | Leprosy | |
| | Leprosy Lepromatous leprosy | |
| | Mycobacterial infection | |
| | Mycobacterial infection Mycobacterial peritonitis | |
| | Mycobacterium abscessus infection | |
| | Mycobacterium avium complex immune | |
| | restoration disease | |
| | Mycobacterium avium complex infection | |
| | Mycobacterium avium complex infection | |
| | Mycobacterium fortuitum infection | |
| | Mycobacterium kansasii infection | |
| | Mycobacterium marinum infection | |
| | Mycobacterium ulcerans infection | |
| | Superinfection mycobacterial | |
| | Tuberculoid leprosy | |
| | Type 1 lepra reaction | |
| | ** | |
| | Type 2 lepra reaction | Droad |
| | Atypical mycobacterium test positive | Broad |
| | Mycobacterial disease carrier | |
| | Mycobacterium leprae test positive | |
| | Mycobacterium test | |
| Salmonallagia (invasiva disessa | Mycobacterium test positive Aortitis salmonella | Norrow |
| Salmonellosis (invasive disease | Arthritis salmonella | Narrow |
| only) (II) | | |
| | Meningitis salmonella | |
| | Osteomyelitis salmonella | |
| | Paratyphoid fever Pneumonia salmonella | |
| | Salmonella bacteraemia | |
| | Salmonella sepsis | |
| | Typhoid fever | Donal |
| | Salmonella test positive | Broad |
| | Salmonellosis | 1 |

| Opportunistic Infection | Preferred Term<br>(MedDRA Version 21.0) | Lilly Defined<br>Classification |
|---|---|---|
| HBV reactivation (IV) | Hepatitis B reactivation | Narrow |
| | Asymptomatic viral hepatitis | Broad |
| | Chronic hepatitis B | |
| | HBV-DNA polymerase increased | |
| | Hepatitis B | |
| | Hepatitis B antigen | |
| | Hepatitis B antigen positive | |
| | Hepatitis B core antigen | |
| | Hepatitis B core antigen positive | |
| | Hepatitis B DNA assay | |
| | Hepatitis B DNA assay positive | |
| | Hepatitis B DNA increased | |
| | Hepatitis B e antigen | |
| | Hepatitis B e antigen positive | |
| | Hepatitis B surface antigen | |
| | Hepatitis B surface antigen positive | |
| | Hepatitis B virus test | |
| | Hepatitis B virus test positive | |
| | Hepatitis infectious | |
| | Hepatitis post transfusion | |
| | Hepatitis viral | |
| | Withdrawal hepatitis | |
| Herpes simplex (invasive disease | Colitis herpes | Narrow |
| only) (IV) | Gastritis herpes | |
| - 5/( - / | Herpes oesophagitis | |
| | Herpes sepsis | |
| | Herpes simplex colitis | |
| | Herpes simplex encephalitis | |
| | Herpes simplex gastritis | |
| | Herpes simplex hepatitis | |
| | Herpes simplex meningitis | |
| | Herpes simplex meningoencephalitis | |
| | Herpes simplex meningomyelitis | |
| | Herpes simplex necrotising retinopathy | |
| | Herpes simplex oesophagitis | |
| | Herpes simplex preumonia | |
| | Herpes simplex sepsis | |
| | Herpes simplex viraemia | |
| | Herpes simplex visceral | |
| | Meningitis herpes | |
| | Meningoencephalitis herpetic | |
| | Meningoeneephantis herpete Meningomyelitis herpes | |
| | Pneumonia herpes viral | |
| | Eczema herpeticum | Broad |
| | Herpes ophthalmic | Divau |
| | Herpes simplex | |

| Opportunistic Infection | Preferred Term (MedDRA Version 21.0) | Lilly Defined<br>Classification |
|---|---|---|
| Opportunistic infection | Herpes simplex DNA test positive | Classification |
| | Herpes virus infection | |
| | Herpes virus test abnormal | |
| | Herpes simplex virus test positive | |
| | Ophthalmic herpes simplex | |
| Herpes zoster (any form) (II) | Disseminated varicella zoster vaccine virus | Narrow |
| Therpes zoster (any form) (ii) | infection | Ivanow |
| | Encephalitis post varicella | |
| | Genital herpes zoster | |
| | Herpes zoster | |
| | Herpes zoster cutaneous disseminated | |
| | Herpes zoster disseminated Herpes zoster disseminated | |
| | Herpes zoster infection neurological | |
| | Herpes zoster meningitis | |
| | Herpes zoster meningoencephalitis | |
| | Herpes zoster meningomyelitis | |
| | Herpes zoster meningomyenus Herpes zoster necrotising retinopathy | |
| | Herpes zoster necrousing retinopathy Herpes zoster oticus | |
| | * | |
| | Herpes zoster pharyngitis Necrotising herpetic retinopathy | |
| | Ophthalmic herpes zoster | |
| | Varicella zoster virus infection | Dungal |
| | Varicella virus test | Broad |
| Comment of the Comment of the comment | Varicella virus test positive | N |
| Stronglyoides (hyperinfection | Strongyloidiasis | Narrow |
| syndrome and disseminated forms only) (IV) | NA | Broad |
| Paracoccidioides infections (V) | Paracoccidioides infection | Narrow |
| | Pulmonary paracoccidioidomycosis | |
| | NA | Broad |
| Penicillium marneffei (V) | Penicilliosis | Narrow |
| - | Penicillium test positive | Broad |
| Sporothrix schenckii (V) | Cutaneous sporotrichosis | Narrow |
| | Pulmonary sporotrichosis | |
| | Sporotrichosis | |
| | NA | Broad |
| Cryptosporidium species (chronic | Biliary tract infection cryptosporidial | Narrow |
| disease only) (IV) | Cryptosporidiosis infection | Broad |
| , , , | Gastroenteritis cryptosporidial | |
| Microsporidiosis (IV) | Microsporidia infection | Narrow |
| 1 | NA | Broad |
| Leishmaniasis (Visceral only) (IV) | Visceral leishmaniasis | Narrow |
| (iv) | Leishmaniasis | Broad |
| Trypanosoma cruzi infection | Chagas' cardiomyopathy | Narrow |
| (Chagas' Disease) (progression of | Meningitis trypanosomal | TAITOW |
| chronic and disseminated disease | American trypanosomiasis | Broad |
| chi onic and dissentificated disease | American u ypanosomiasis | Divau |

| | Preferred Term | Lilly Defined |
|---|---|---|
| Opportunistic Infection | (MedDRA Version 21.0) | Classification |
| only) (V) | Trypanosomiasis | |
| | Trypanosoma serology positive | 27 |
| Campylobacteriosis (invasive disease only) (V) | Campylobacter sepsis | Narrow |
| | Campylobacter infection | Broad |
| | Campylobacter test positive | |
| Shigellosis (invasive disease only) | Shigella sepsis | Narrow |
| (V) | Shigella infection | Broad |
| | Shigella test positive | |
| Vibriosis (invasive disease due to $V$ . | NA | Narrow |
| vulfnificus) (V) | Vibrio test positive | Broad |
| | Vibrio vulnificus infection | |
| HCV progression (V) | NA | Narrow |
| | Chronic hepatitis C | Broad |
| | Hepatitis C | |
| | Hepatitis C RNA | |
| | Hepatitis C RNA increased | |
| | Hepatitis C RNA fluctuation | |
| | Hepatitis C RNA positive | |
| | Hepatitis C virus test | |
| | Hepatitis C virus test positive | |
| Non-specific terms | NA | Narrow |
| Tion specific terms | Abscess fungal | Broad |
| | Alternaria infection | Broud |
| | Arthritis fungal | |
| | Biliary tract infection fungal | |
| | Central nervous system fungal infection | |
| | Cerebral fungal infection | |
| | Encephalitis fungal | |
| | Erythema induratum | |
| | Eye infection fungal | |
| | Fungaemia | |
| | Fungal abscess central nervous system | |
| | Fungal endocarditis | |
| | Fungal labyrinthitis | |
| | Fungal peritonitis | |
| | Fungal pharyngitis | |
| | Fungal retinitis | |
| | Fungal sepsis | |
| | Hepatic infection fungal | |
| | Meningitis fungal | |
| | Mycotic endophthalmitis | |
| | Myocarditis mycotic | |
| | Oropharyngitis fungal | |
| | Osteomyelitis fungal | |
| | Otitis media fungal | |
| | _ | |
| | Pancreatitis fungal | |

| Opportunistic Infection | Preferred Term<br>(MedDRA Version 21.0) | Lilly Defined<br>Classification |
|---|---|---|
| | Parasitic lung infection | |
| | Parasitic pneumonia | |
| | Pericarditis fungal | |
| | Phaehyphomycosis | |
| | Pneumonia fungal | |
| | Pulmonary mycosis | |
| | Pulmonary trichosporonosis | |
| | Sinusitis fungal | |
| | Splenic infection fungal | |
| | Systemic mycosis | |

Abbreviations: EBV = Epstein-Barr virus; HBV = hepatitis B virus; HCV = hepatitis C virus; NA = not applicable; PVAN = polyomavirus-associated nephropathy.

# Appendix 4. MedDRA Preferred Terms for each Category Associated with Criterion 2 for Anaphylactic Allergic Reactions/Hypersensitivity Events

| Preferred Terms (MedDRA Version 21.0) | |
|---|---|
| Category A: Involvement of the Skin/Mucosal Tissue | , |
| Administration site hypersensitivity | Localised oedema |
| Administration site rash | Mouth swelling |
| Administration site urticarial | Nasal obstruction |
| Allergic oedema | Nodular rash |
| Allergic otitis externa | Ocular hyperaemia |
| Angioedema | Oedema |
| Circumoral oedema | Oedema mouth |
| Drug eruption | Oedema mucosal |
| Erythema | Orbital oedema |
| Eye allergy | Palatal oedema |
| Eye oedema | Palatal swelling |
| Eye pruritus | Perineal rash |
| Eye swelling | Periorbital oedema |
| Eyelid oedema | Pruritus |
| Face oedema | Pruritus allergic |
| Flushing | Pruritus generalised |
| Generalised erythema | Rash |
| Gingival oedema | Rash erythematous |
| Gingival swelling | Rash generalised |
| Idiopathic urticaria | Rash pruritic |
| Injection site dermatitis | Skin oedema |
| Injection site hypersensitivity | Skin swelling |
| Injection site rash | Swelling |
| Injection site urticaria | Swelling face |
| Injection site vasculitis | Swollen tongue |
| Lip oedema | Tongue oedema |
| Lip swelling | Urticaria |
| | Urticaria papular |
| Category B: Respiratory Compromise | |
| Acute respiratory failure | Laryngotracheal oedema |
| Allergic cough | Oropharyngeal spasm |
| Allergic pharyngitis | Oropharyngeal swelling |
| Asthma | Pharyngeal oedema |
| Asthmatic crisis | Respiratory arrest |
| Bronchial hyperreactivity | Respiratory distress |
| Bronchial oedema | Respiratory failure |
| Bronchospasm | Respiratory tract oedema |
| Cardio-respiratory distress | Reversible airways obstruction |
| Chest discomfort | Sensation of foreign body |
| Choking | Sneezing |

| Preferred Terms (MedDRA Version 21.0) | |
|---|---|
| Choking sensation | Spasmodic dysphonia |
| Cough | Status asthmaticus |
| Cyanosis | Stridor |
| Dyspnoea | Tachypnea |
| Epiglottic oedema | Throat tightness |
| Hyperventilation | Tracheal obstruction |
| Нурохіа | Tracheal oedema |
| Laryngeal dyspnoea | Upper airway obstruction |
| Laryngeal obstruction | Wheezing |
| Laryngeal oedema | |
| Laryngitis allergic | |
| Laryngospasm | |
| Category C: Reduced Blood Pressure or Associated Symptoms | |
| Blood pressure decreased | Hypoperfusion |
| Blood pressure diastolic decreased | Hypotension |
| Blood pressure systolic decreased | Hypovolaemic shock |
| Cardiac arrest | Incontinence |
| Cardiopulmonary failure | Mean arterial pressure decreased |
| Cardio-respiratory arrest | Peripheral circulatory failure |
| Cardiovascular insufficiency | Presyncope |
| Circulatory collapse | Shock |
| Diastolic hypotension | Shock symptom |
| Distributive shock | Syncope |
| Dizziness | Urinary Incontinence |
| Category D: Persistent Gastrointestinal Symptoms | |
| Abdominal discomfort | Gastrointestinal pain |
| Abdominal pain | Intestinal angioedema |
| Abdominal pain lower | Nausea |
| Abdominal pain upper | Retching |
| Diarrhoea | Visceral pain |
| Epigastric discomfort | Vomiting |
| Gastrointestinal oedema | |

Abbreviations: MedDRA = Medical Dictionary for Regulatory Activities.

### Appendix 5. Allergic Reactions/Hypersensitivity MedDRA Preferred Term List

Allergic reactions/hypersensitivities will be defined using the following MedDRA Preferred Terms as defined in MedDRA:

- Broad and narrow terms in the Anaphylactic reaction SMQ (20000021)
- Broad and narrow terms in the Angioedema SMQ (20000024)
- Broad and narrow terms in the Severe cutaneous adverse reactions SMQ (20000020)
- Broad and narrow terms in the Hypersensitivity SMQ (20000214), excluding the preferred terms as noted below.

| Preferred Terms (MedDRA v.21.0) from Hypersensitivity SMQ Excluded from Analysis | |
|---|---|
| Administration site dermatitis | Injection site rash |
| Administration site eczema | Injection site recall reaction |
| Administration site rash | Injection site urticaria |
| Administration site recall reaction | Injection site vasculitis |
| Allergic otitis externa | Instillation site hypersensitivity |
| Allergic otitis media | Instillation site rash |
| Allergic sinusitis | Instillation site urticaria |
| Allergic transfusion reaction | Iodine allergy |
| Allergy alert test positive | Mast cell degranulation present |
| Allergy test positive | Medical device site dermatitis |
| Allergy to surgical sutures | Medical device site eczema |
| Allergy to vaccine | Medical device site hypersensitivity |
| Anaphylactic transfusion reaction | Medical device site rash |
| Antiallergic therapy | Medical device site recall reaction |
| Application site dermatitis | Medical device site urticaria |
| Application site eczema | Nodular rash |
| Application site hypersensitivity | Pathergy reaction |
| Application site rash | Radioallergosorbent test positive |
| Application site recall reaction | Reaction to azo-dyes |
| Application site urticaria | Reaction to colouring |
| Application site vasculitis | Shock |
| Arthritis allergic | Shock symptom |
| Aspirin-exacerbated respiratory disease | Skin test positive |
| Asthma-chronic obstructive pulmonary disease | Solvent sensitivity |
| overlap syndrome | Stoma site hypersensitivity |
| Blepharitis allergic | Stoma site rash |
| Blood immunoglobulin E abnormal | Urticaria contact |
| Blood immunoglobulin E increased | Urticarial vasculitis |
| Bromoderma | Vaccination site dermatitis |
| Catheter site dermatitis | Vaccination site exfoliation |
| Catheter site eczema | Vaccination site eczema |
| Catheter site hypersensitivity | Vaccination site hypersensitivity |
| Catheter site rash | Vaccination site rash |

#### Preferred Terms (MedDRA v.21.0) from Hypersensitivity SMQ Excluded from Analysis

Catheter site urticaria Catheter site vasculitis

Chronic eosinophilic rhinosinusitis

Chronic hyperplastic eosinophilic sinusitis

Circulatory collapse Conjunctivitis allergic Contact stomatitis

Complement factor decreased Complement factor increased Complement factor C1 decreased Complement factor C1 increased Complement factor C2 decreased

Complement factor C2 decreased Complement factor C3 decreased Complement factor C3 increased Complement factor C4 decreased Complement factor C4 increased Complement fixation abnormal Complement fixation test positive

Contrast media allergy
Contrast media reaction
Dennie-Morgan fold
Dermatitis acneiform
Dermatitis contact
Dermatitis herpetiformis
Dermatitis infected
Device allergy

Dialysis membrane reaction

Distributive shock
Drug cross-reactivity
Drug provocation test
Eczema infantile
Eczema vaccinatum
First use syndrome
Fixed drug eruption

Giant papillary conjunctivitis

Heparin-induced thrombocytopenia

Hereditary angioedema Implant site dermatitis Implant site hypersensitivity

Implant site rash
Implant site urticaria

Immune-mediated adverse reaction

Incision site dermatitis Incision site rash Infusion site dermatitis Infusion site eczema

Infusion site hypersensitivity

Vaccination site recall reaction

Vaccination site urticaria Vaccination site vasculitis Vaccination site vesicles

Vessel puncture site rash Vessel puncture site vesicles

Vulvovaginal rash Acute respiratory failure Allergy to chemicals

Allergy to fermented products Anti-insulin antibody increased Anti-insulin antibody positive

Anti-insulin receptor antibody increased Anti-insulin receptor antibody positive Blood immunoglobulin A abnormal Blood immunoglobulin A increased Blood immunoglobulin D increased Blood immunoglobulin G abnormal Blood immunoglobulin G increased Blood immunoglobulin G increased Blood immunoglobulin M abnormal Blood immunoglobulin M increased Immune complex level increased Immunoglobulins abnormal Immunoglobulins increased Immunoglobulins increased Immunology test abnormal

Haemolytic transfusion reaction

Infantile asthma Fixed eruption Rhinitis perennial Seasonal allergy

| Preferred Terms (MedDRA v.21.0) from Hypersensitivity SMQ Excluded from Analysis |
|---|
| Infusion site rash |
| Infusion site recall reaction |
| Infusion site urticaria |
| Infusion site vasculitis |
| Injection site dermatitis |
| Injection site eczema |
| Injection site hypersensitivity |

# Appendix 6. Lilly-Defined MedDRA V21.0 Preferred Terms for Inflammatory Bowel Disease (IBD)

| | | Lilly-Defined |
|---|---|---|
| Condition | Preferred Term (MedDRA version 21.0) | Classification |
| Inflammatory bowel disease | Inflammatory bowel disease | Narrow |
| Crohn's disease | Crohn's disease | Narrow |
| Ulcerative colitis | Acute haemorrhagic ulcerative colitis | Narrow |
| | Colitis ulcerative | Narrow |
| | Proctitis ulcerative | Narrow |
| Non-specific terms | Abscess intestinal | Broad |
| | Anal abscess | Broad |
| | Anal fistula | Broad |
| | Anal fistula excision | Broad |
| | Anal fistula infection | Broad |
| | Anovulvar fistula | Broad |
| | Aorto-duodenal fistula | Broad |
| | Colitis | Broad |
| | Colon fistula repair | Broad |
| | Colonic fistula | Broad |
| | Diverticular fistula | Broad |
| | Duodenal fistula | Broad |
| | Enterocolitis haemorrhagic | Broad |
| | Enterocolonic fistula | Broad |
| | Enterocutaneous fistula | Broad |
| | Enterovesical fistula | Broad |
| | Gastrointestinal fistula | Broad |
| | Gastrointestinal fistula repair | Broad |
| | Fistula of small intestine | Broad |
| | Intestinal fistula | Broad |
| | Intestinal fistula infection | Broad |
| | Intestinal fistula repair | Broad |
| | Jejunal fistula | Broad |
| | Large intestinal ulcer perforation | Broad |
| | Rectal fistula repair | Broad |
| | Faecal calprotectin abnormal | Broad |
| | Faecal calprotectin increased | Broad |
| | Proctitis haemorrhagic | Broad |
| | Pseudopolyposis | Broad |
| | Rectoprostatic fistula | Broad |
| | Rectourethral fistula | Broad |

Leo Document ID = 49b21032-dd6b-42de-b571-d08947d59dd4

Approver: PPD

Approval Date & Time: 26-Jun-2019 15:54:01 GMT Signature meaning: Approved